An Open-label, Baseline-controlled, Multicenter, Phase 3 Dosetitration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents From 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)

Open-label Phase 3 Study with Mirabegron in Children From 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (Crocodile Study)

ISN/Protocol 178-CL-206A

ClinicalTrials.gov Identifier: NCT02751931

Date of Protocol v2: 02 Nov 2016

Sponsor: Astellas Pharma Europe B.V. (APEB)

Sylviusweg 62 2333 BE Leiden, the Netherlands **Sponsor: APEB** EudraCT number 2015-002876-25


An Open-label, Baseline-controlled, Multicenter, Phase 3 Dose-titration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents From 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)

Open-label Phase 3 Study with Mirabegron in Children from 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (Crocodile Study)

# ISN/Protocol 178-CL-206A

# Version 2.0

# Incorporating Substantial Amendment 1 [See Attachment 1] 02 November 2016



EudraCT 2015-002876-25

# Sponsor:

# Astellas Pharma Europe B.V. (APEB)

Sylviusweg 62 2333 BE Leiden, the Netherlands

Protocol History: Version 1.0 [09 Dec 2015]

**Investigator**: Investigator information is on file at Astellas

\_\_\_\_\_

This confidential document is the property of the Sponsor. No unpublished information contained in this document may be disclosed without prior written approval of the Sponsor.

# **Table of Contents**

| I. | | S | SIGNATURES ·····8 | |
|---|---|---|---|---|
| II. | | ( | CONTACT DETAILS OF KEY SPONSOR'S PERSONNEL·····10 | |
| III. | | L | LIST OF ABBREVIATIONS AND DEFINITION OF KEY TERMS11 | |
| IV. | | S | SYNOPS | 6IS ·······15 |
| V. | | F | LOW ( | CHART AND SCHEDULE OF ASSESSMENTS ······25 |
| 1 | | Ι | | OUCTION28 |
| | 1.1 | | Bacl | kground ······28 |
| | 1.2 | 2 | Non | clinical and Clinical Data · · · · · 29 |
| | | 1.2 | 2.1 | Nonclinical Data —————————————————————————————————— |
| | | 1.2 | 2.2 | Clinical Data · · · · · 31 |
| | 1.3 | ; | Sum | mary of Key Safety Information for Study Drugs ······34 |
| | 1.4 | | Risk | -Benefit Assessment · · · · · 34 |
| 2 | | S | TUDY | OBJECTIVE(S), DESIGN, AND ENDPOINTS ······37 |
| | 2.1 | | Stud | y Objectives |
| | | 2.1 | 1 | Primary Objectives: |
| | | 2.1 | 2 | Secondary Objectives: 37 |
| | 2.2 | 2 | Stud | y Design and Dose Rationale · · · · · · 37 |
| | | 2.2 | 2.1 | Study Design · · · · · 37 |
| | | | 2.2.1.1 | Pretreatment Period······37 |
| | | | 2.2.1.2 | Efficacy Treatment Period · · · · · 38 |
| | | | 2.2.1.3 | Long-term Safety Period · · · · · 39 |
| | | 2.2 | 2.2 | Dose Rationale 39 |
| | 2.3 | ; | End | points 40 |
| | | 2.3 | 3.1 | Primary Efficacy Endpoint · · · · · 40 |
| | | 2.3 | 3.2 | Secondary Efficacy Endpoints · · · · · 40 |
| | | | 2.3.2.1 | Urodynamic Measures ·····40 |
| | | | 2.3.2.2 | Bladder Volume and Leakage Measures ······40 |
| | | | 2.3.2.3 | Patient- or Clinician-reported Questionnaire Endpoints · · · · · 41 |
| | | 2.3 | 3.3 | Safety Endpoints 41 |
| | | 2.3 | 3.4 | Pharmacokinetics 41 |
| | | 2.3 | 3.5 | Exploratory Endpoints · · · · 42 |
| | | | 2.3.5.1 | Exploratory Efficacy Endpoints42 |

| | | 2. | 3.5.2 Exploratory Safety Endpoints · · · · · 42 |
|---|---|---|---|
| 3 | | STU | UDY POPULATION 42 |
| | 3.1 | | Selection of Study Population · · · · · 42 |
| | 3.2 | | Inclusion Criteria · · · · · 42 |
| | 3.3 | | Exclusion Criteria · · · · · 44 |
| 4 | | TR | EATMENTS45 |
| | 4.1 | | Identification of Investigational Products · · · · · · 45 |
| | | 4.1.1 | Test Drug45 |
| | | 4.1.2 | Comparative Drug(s)······46 |
| | 4.2 | | Packaging and Labeling · · · · · · 46 |
| | 4.3 | | Study Drug Handling ·····46 |
| | 4.4 | | Blinding ······47 |
| | 4.5 | | Assignment and Allocation |
| | | 4.5.1 | Subject Numbering · · · · · · 47 |
| | [ | 4.5.2 | Subject Replacement · · · · · · 47 |
| 5 | | TR | EATMENTS AND EVALUATION······47 |
| | 5.1 | | Dosing and Administration of Study Drug · · · · · 47 |
| | | 5.1.1 | Dose/Dose Regimen and Administration Period · · · · · · · 47 |
| | | 5.1.2 | Increase or Reduction in Dose of the Study Drug(s) · · · · · · 48 |
| | | 5.1.3 | Previous and Concomitant Treatment (Medication and Nonmedication |
| | | | Therapy)49 |
| | | 5.1.4 | Treatment Compliance 49 |
| | | 5.1.5 | Restrictions for Foods and Drinks During the Study49 |
| | 5.2 | | Demographics and Baseline Characteristics |
| | | 5.2.1 | Demographics·····49 |
| | | 5.2.2 | Medical History·····49 |
| | | 5.2.3 | Diagnosis of the Target Disease, Severity, and Duration of Disease50 |
| 5.3 Efficacy and Pharmacokinetics Assessment ····· | | Efficacy and Pharmacokinetics Assessment50 | |
| | | 5.3.1 | Urodynamic Assessments · · · · · 50 |
| | | 5.3.2 | Bladder Diary ·····51 |
| | | 5.3.3 | Questionnaires · · · · 52 |
| | | 5.3.4 | Pharmacokinetics |
| | 5.4 | | Safety Assessments · · · · · 54 |

| | | 5.4.1 | Vital Signs·····54 |
|---|---|---|---|
| | | 5.4.1.1 | Clinic Measurement of Vital Signs · · · · 54 |
| | | 5.4.1.2 | Self-measurement of Vital Signs · · · · 54 |
| | | 5.4.2 | Adverse Events · · · · 55 |
| | | 5.4.2.1 | Adverse Events of Possible Hepatic Origin · · · · 55 |
| | | 5.4.3 | Laboratory Assessments · · · · 55 |
| | | 5.4.4 | Physical Examination |
| | | 5.4.5 | Electrocardiograms |
| | | 5.4.6 | Self-measurement of Intravesical Pressure |
| | | 5.4.7 | Estimated Glomerular Filtration Rate and Upper Urinary Tract Ultrasound ····· 58 |
| | 5.5 | 5 Adv | erse Events and Other Safety Aspects59 |
| | | 5.5.1 | Definition of Adverse Events · · · · 59 |
| | | 5.5.2 | Definition of Serious Adverse Events · · · · 59 |
| | | 5.5.3 | Criteria for Causal Relationship to the Study Drug ······60 |
| | | 5.5.4 | Criteria for Defining the Severity of an Adverse Event ······61 |
| | | 5.5.5 | Reporting of Serious Adverse Events · · · · 61 |
| | | 5.5.6 | Follow-up of Adverse Events · · · · 62 |
| | | 5.5.7 | Monitoring of Common Serious Adverse Events · · · · 62 |
| | | 5.5.8 | Procedure in Case of Pregnancy 62 |
| | | 5.5.9 | Emergency Procedures and Management of Overdose · · · · · 63 |
| | | 5.5.10 | Supply of New Information Affecting the Conduct of the Study63 |
| | 5.6 | Test | Drug Concentration · · · · 63 |
| | 5.7 | ' Oth | er Measurements, Assessments or Methods ······63 |
| | 5.8 | 3 Tota | al Amount of Blood ······64 |
| 6 | | DISCO | NTINUATION······64 |
| | 6.1 | Disc | continuation of Individual Subject(s) |
| | 6.2 | . Disc | continuation of the Site65 |
| | 6.3 | Disc | continuation of the Study65 |
| 7 | | STATIS | TICAL METHODOLOGY ······65 |
| | 7.1 | Sam | pple Size·····65 |
| | 7.2 | . Ana | lysis Set66 |
| | | 7.2.1 | Full Analysis Set66 |
| | | 7.2.2 | Per Protocol Set·····66 |
| | | 7.2.3 | Safety Analysis Set ····· 67 |

| 7.2.4 Pharmacokinetics Analysis Set ·······67 |
|---|
| 7.3 Demographics and Other Baseline Characteristics 67 |
| 7.4 Analysis of Efficacy6 |
| 7.4.1 Analyses of Primary Endpoint · |
| 7.4.1.1 Primary Analysis 67 |
| 7.4.1.2 Secondary Analyses · · · · · 68 |
| 7.4.1.3 Subgroup and Sensitivity Analyses of Primary Endpoint |
| 7.4.2 Analysis of Secondary Endpoints |
| 7.4.3 Analysis of Exploratory Endpoints 69 |
| 7.5 Analysis of Safety 69 |
| 7.5.1 Vital Signs |
| 7.5.2 Adverse Events · · · · · 69 |
| 7.5.3 Laboratory Assessments 69 |
| 7.5.4 Physical Examination 70 |
| 7.5.5 Electrocardiograms 70 |
| 7.5.6 Estimated Glomerular Filtration Rate and Upper Urinary Tract Ultrasound70 |
| 7.5.7 Analysis of Exploratory Endpoints |
| 7.6 Analysis of Pharmacokinetics · |
| 7.6.1 Estimation of Pharmacokinetic Parameters71 |
| 7.7 Protocol Deviations and Other Analyses · · · · · 71 |
| 7.8 Interim Analysis (and Early Discontinuation of the Clinical Study)71 |
| 7.9 Handling of Missing Data, Outliers, Visit Windows, and Other Information · · · · · · · 71 |
| 8 OPERATIONAL AND ADMINISTRATIVE CONSIDERATIONS ······72 |
| 8.1 Procedure for Clinical Study Quality Control · |
| 8.1.1 Data Collection · |
| 8.1.1.1 Electronic Patient Reported Outcomes · |
| 8.1.2 Specification of Source Documents |
| 8 1 3 Clinical Study Monitoring |
| 8.1.4 Direct Access to Source Data/Documents |
| 8.1.5 Data Management ·······74 |
| 8.1.6 Protocol Deviations |
| 8.1.7 End of Trial in All Participating Countries |
| 8.2 Ethics and Protection of Subject Confidentiality |
| 8.2.1 Independent Ethics Committee/Competent Authorities |

| | 0.2.2 | | |
|---|---|---|---|
| | 8.2.2 | Ethical Conduct of the Study 76 | |
| | 8.2.3 | Informed Consent of Subjects ······76 | |
| 8.2.3.1 Subject Information and Consent ···································· | | | |
| | 8 | 2.3.2 Supply of New and Important Information Influencing the Subject's | _ |
| | | Consent and Revision of the Written Information ······77 | |
| | 8.2.4 | Subject Confidentiality · · · · · · · 78 | |
| | 8.3 | Administrative Matters ······78 | |
| | 8.3.1 | Arrangement for Use of Information and Publication of the Clinical Study ·····78 | |
| | 8.3.2 | Documents and Records Related to the Clinical Study ······78 | |
| | 8.3.3 | Protocol Amendment and/or Revision ······79 | |
| | 8.3.4 | Insurance of Subjects and Others ·······79 | |
| | 8.3.5 | Signatory Investigator for Clinical Study Report ·······79 | |
| 9 | QU | ALITY ASSURANCE·····80 | |
| 10 | STU | UDY ORGANIZATION·····80 | |
| | 10.1 | Independent Data-Monitoring Committee Data and Safety Monitoring Board | |
| | | Monitoring Committee Other Evaluation Committee(s) | |
| | 10.2 | Other Study Organization · · · · 80 | |
| 11 | RE | FERENCES81 | |
| 12 | AP | PENDICES 83 | |
| | 12.1 | List of Excluded Concomitant Medications · · · · · 83 | |
| | 12.2 | Liver Safety Monitoring and Assessment ······84 | |
| | 12.3 | Laboratory Assessments · · · · · · 87 | |
| | 12.4 | Pediatric Incontinence Questionnaire | |
| | 12.5 | Patient Global Impression of Severity Scale | |
| | 12.6 | Acceptability Questionnaire for Tablets 90 | |
| | 12.7 | Acceptability Questionnaire for Oral Suspension91 | |
| | 12.8 | Clinical Global Impression of Change Scale · · · · 93 | |
| | 12.9 | Centiles of heart rate for normal children from birth to 18 years of age [Fleming | |
| | | et al, 2011] · · · · · · 94 | |
| | 12.10 | CDC Data Table of Stature-for-age Chart for Males · · · · 95 | |
| | 12.11 | CDC Data Table of Stature-for-age Chart for Females · · · · 102 | |
| | 12.12 | Blood Pressure Levels for Boys by Age and Height Percentile [NIH 2005] · · · · · 109 | |
| | 12.13 | Blood Pressure Levels for Girls by Age and Height Percentile [NIH 2005] 111 | |

EudraCT number 2015-002876-25


| 13 | ATTACHMENT 1: SUBSTANTIAL AMENDMENT 1 |
|----|---------------------------------------|
| 14 | SPONSOR'S SIGNATURES |

# **List of Tables**

| Table 1 | Schedule of Assessments 26 |
|---|---|
| Table 2 | Overview of Current Supporting Mirabegron Studies in the Pediatric Clinical |
| | Development Program for NDO and OAB ······31 |
| Table 3 | 178-CL-208 Draft Results: Relative Bioavailability of the Mirabegron 8 mg/mL |
| | Oral Suspension Formulation versus 2 mg/mL Oral suspension Formulation |
| | (Pharmacokinetics Analysis Set) ·······33 |
| Table 4 | Weight-based Doses for Tablets or Suspension ·······48 |
| Table 5 | Total Amount of Blood Volume per Subject During the Study Period · 64 |

**Sponsor: APEB** 

EudraCT number 2015-002876-25


# I. SIGNATURES

# 1. SPONSOR'S SIGNATURE

Required signatures (e.g., Protocol authors, Sponsor's reviewers and contributors, etc.) are located in Section 4 Sponsor's Signatures; e-Signatures (when applicable) are located at the end of this document.

Sponsor: APEB ISN/Protocol 178-CL-206A

EudraCT number 2015-002876-25


## 2. INVESTIGATOR'S SIGNATURE

An Open-label, Baseline-controlled, Multicenter, Phase 3 Dose-titration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents From 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)

ISN/Protocol 178-CL-206A

**Version 2.0 Incorporating Substantial Amendment 1** 

# **02 November 2016**

I have read all pages of this clinical study protocol for which Astellas is the Sponsor. I agree to conduct the study as outlined in the protocol and to comply with all the terms and conditions set out therein. I confirm that I will conduct the study in accordance with ICH GCP guidelines and applicable local regulations. I will also ensure that sub-investigator(s) and other relevant members of my staff have access to copies of this protocol and the ICH GCP guidelines to enable them to work in accordance with the provisions of these documents.

| Principal Investigator: | |
|---|---|
| Signature: <insert and="" investigator="" name="" of="" qualifications="" the=""></insert> | |
| <insert and="" investigator="" name="" of="" qualifications="" the=""></insert> | Date (DD Mmm YYYY) |
| Printed Name: | |
| Address: | |

# II. CONTACT DETAILS OF KEY SPONSOR'S PERSONNEL



Sponsor: APEB

EudraCT number 2015-002876-25


# III. LIST OF ABBREVIATIONS AND DEFINITION OF KEY TERMS

# **List of Abbreviations**

| List of Abbreviations | |
|---|---|
| Abbreviation | Description |
| APEB | Astellas Pharma Europe B.V. |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AST | aspartate aminotransferase |
| AUC <sub>24</sub> | Area under the plasma concentration-time curve from time zero to 24 h |
| CIC | clean intermittent catheterization |
| CGI-C | Clinician Global Impression of Change |
| CL/F | apparent total clearance of the drug from plasma after oral administration |
| $C_{max}$ | maximum (peak) plasma drug concentration |
| CRO | contract research organization |
| CSR | clinical study report |
| $C_{\text{trough}}$ | trough plasma concentration (measured concentration at the end of a dosing |
| | interval at steady state) |
| CYP | cytochrome P450 |
| DSD | detrusor sphincter dyssynergia |
| DSMB | Data and Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | electronic case report form |
| e-diary | electronic diary |
| eGFR | estimated glomerular filtration rate |
| EOS | end of study |
| EOT | end of treatment |
| FAS | full analysis set |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| IB | Investigator's Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IMPD | Investigational Medicinal Product Dossier |
| INR | international normalized ratio |
| ISN | international study number |
| IUD | intrauterine device |
| IUS | intrauterine system |
| LA-CRF | liver abnormality case report form |
| LC-MS/MS | liquid chromatography-mass spectrometry and tandem mass spectrometry |
| LOCF | last observation carried forward |
| LFT | liver function test |
| LQTS | long QT syndrome |
| MCC | maximum cystometric capacity |
| NDO | neurogenic detrusor overactivity |
| OAB | overactive bladder |
| PED | pediatric equivalent dose |

EudraCT number 2015-002876-25

| Abbreviation | Description |
|---|---|
| PGI-S | Patient Global Impression of Severity Scale |
| P-gp | P-glycoprotein P-glycoprotein |
| PIN-Q | Pediatric Incontinence Questionnaire |
| PKAS | pharmacokinetics analysis set |
| PND | postnatal day |
| popPK | population pharmacokinetics |
| PPS | per protocol set |
| QTcB | QT interval corrected by Bazett's formula |
| QTcF | QT interval corrected by Fridericia's formula |
| SAE | serious adverse event |
| SAF | safety analysis set |
| SAP | statistical analysis plan |
| SBPM | self blood pressure measurement |
| SMIP | self-measurement of intravesical pressure |
| SOP | standard operating procedure |
| TEAE | treatment-emergent adverse event |
| TBL | total bilirubin |
| TLF | tables, listings and figures |
| $t_{max}$ | time to reach maximum (peak) plasma concentration following drug |
| | administration |
| ULN | upper limit of normal |
| UTI | urinary tract infection |
| V <sub>z</sub> /F | apparent volume of distribution after nonintravenous administration |

# **Definition of Key Study Terms**

| Terms | Definition of terms |
|---|---|
| Baseline | Observed values/findings which are considered to be the starting point for comparison. |
| Discontinuation | The act of concluding participation in a trial by an enrolled subject, prior to completion of all protocol required elements. |
| | Note: subject discontinuation does not necessarily imply exclusion of subject data from analysis that was collected prior to discontinuation. |
| Enroll | To register or enter into a clinical trial, i.e., signing the informed consent form (ICF). Once a subject has been enrolled, the clinical trial protocol applies to the subject. |
| Investigational period | Period of time where major interests of protocol objectives are observed, and where the study drug is given to a subject. This period continues until the last assessment after completing the last dose of the study drug. |
| Pediatric equivalent dose (PEDx) | Weight-range based doses predicted to achieve plasma concentrations equivalent to steady state exposures expected with "x" mg mirabegron administered once daily in adults. |
| Postinvestigational period | Period of time after the last assessment of the protocol. Follow-up observations for sustained adverse events and/or survival are done in this period. |
| Screening | A process of active consideration of potential subjects for a trial. |
| Screening period | Period of time before entering the investigational period, usually from the time the subject signed informed consent until just before the first dose of the study drug is given to a subject. |
| Screening failure | Screened subject who did not fulfill protocol inclusion and/or exclusion criteria, or decided not to participate anymore (withdrew consent) prior to first dose of study drug. |
| Source data | All information in original records or certified copies of original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Source data are contained in source documents (original records, certified copies). |
| Source documents | Original documents, data, and records including source data. |
| Steady state | When the amount of drug intake is equilibrium with the rate of drug elimination. |
| | Note: for mirabegron steady state is considered to be reached after 10 days of daily dosing. |
| Study completion | Status of subject who completed the last protocol-defined assessment. |
| Study period | Period of time from the first site initiation date to the last site completing the study. |
| Subject | An individual in the population of interest who participates in a clinical trial as recipient of the investigational product. |

**Sponsor: APEB** 

EudraCT number 2015-002876-25

| Terms | Definition of terms |
|---|---|
| Treatment emergent adverse event | An adverse event observed after starting administration of the study drug. |
| Trough sample | Pharmacokinetic sample taken just prior to the next dose of study drug. |

Sponsor: APEB

EudraCT number 2015-002876-25


# IV. SYNOPSIS

| Date and Version # of Protocol Synopsis: | 02 November 2016, Version 2.0 |
|---|---|
| Sponsor: | Protocol Number: |
| Astellas Pharma Europe BV (APEB) | 178-CL-206A |
| Name of Study Drug: | Phase of Development: |
| Mirabegron | Phase 3 |

#### Title of Study:

An Open-label, Baseline-controlled, Multicenter, Phase 3 Dose-titration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents from 3 to less than 18 Years of Age with Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)

#### **Planned Study Period:**

From 2Q2016 to 3Q2019.

#### **Study Objectives:**

#### Primary objective:

• To evaluate the efficacy of mirabegron after multiple-dose administration in the pediatric population.

#### Secondary objectives:

- To evaluate the safety and tolerability of mirabegron after multiple-dose administration in the pediatric population.
- To evaluate the pharmacokinetics of mirabegron after multiple-dose administration in the pediatric population.

#### Planned Total Number of Study Centers and Location(s):

Approximately 50 enrolling study centers in Europe, Latin America, Africa, Middle East and Asia-Pacific.

#### **Study Population:**

Male and female pediatric child and adolescent subjects aged 3 to less than 18 years of age with neurogenic detrusor overactivity (NDO) on clean intermittent catheterization (CIC).

#### Number of Subjects to be Enrolled/Randomized:

At least 44 evaluable subjects (estimate 63 enrolled), with at least 10 subjects from each age group (children aged 3 to less than 12 years of age; adolescents aged 12 to less than 18 years of age) are planned. A subject is considered being evaluable if the subject has a valid (as by the central reviewer's assessment) nonmissing maximum cystometric capacity (MCC) measurement at baseline and at a postbaseline visit.

## **Study Design Overview:**

This is a phase 3, open-label, baseline-controlled, multicenter study. The study will consist of 3 periods:

- Pretreatment period: for a maximum of 28 days before baseline, including screening, washout (if applicable) and baseline
- Efficacy treatment period: beginning the day after baseline and continuing to visit 8/week 24
- Long-term safety period: beginning after visit 8/week 24 and continuing to visit 10/week 52 (end of study [EOS]), or to the end of treatment (EOT)

ISN/Protocol 178-CL-206A

Sponsor: APEB
EudraCT number 2015-002876-25


#### Pretreatment Period

After informed consent and visit 1/screening, subjects are grouped according to their current NDO therapy and/or other medication:

- Group A: Subjects who are currently not receiving any prohibited medication including any oral drug treatment to manage their NDO, or when botulinum toxin is no longer considered effective.
- Group B: Subjects who currently are receiving oral drug treatment to manage their NDO or receive any other prohibited medication.

After the screening visit a 2-day weekend e-diary has to be completed by the subjects to get acquainted with the electronic diary (e-diary) and the home assessments:

- Group A: Following successful completion of the first 2-day weekend e-diary, confirmed at visit 2, the subjects will start to complete the 7-day baseline e-diary followed by visit 3/baseline.
- Group B: Following successful completion of the first 2-day weekend e-diary, confirmed at visit 2, the subjects will start their 2-week washout period. In the second week of their washout period, they will complete the 7-day baseline e-diary followed by visit 3/baseline.

If a subject is suffering from a symptomatic urinary tract infection (UTI) at visit 1/screening or is diagnosed with one between visit 1/screening and visit 3/baseline, the UTI should be treated successfully (clinical recovery) prior to baseline. If a symptomatic UTI is present at baseline, all baseline assessments should be postponed for a maximum of 7 days until the UTI is successfully treated (clinical recovery).

The 7-day baseline e-diary does not have to be repeated if at least the 2-day weekend e-diary and 1 day of the weekday e-diary were completed while the subject did not suffer from a symptomatic UTI.

Subjects will enter the efficacy treatment period if they meet the eligibility criteria and satisfactorily complete the pretreatment period (ability to complete bladder diary, catheterized volumes and questionnaires).

In case the subject or the subject's parent(s)/caregiver(s) are not able or willing to perform the SMIP, the measuring device is not available at the site, or there is a technical problem, the SMIP may be omitted.

#### **Efficacy Treatment Period**

Daily study drug administration will begin the day after the baseline visit. The initial dose of mirabegron will be based on the subject's weight, and is predicted to achieve plasma concentrations equivalent to the steady state exposures expected with 25 mg mirabegron administered once daily in adults (pediatric equivalent dose [PED25]).

At visit 4/week 2, visit 5/week 4 or visit 6/week 8, subjects must be up-titrated to the pediatric equivalent dose of 50 mg in adults (PED50) based on the given dose titration criteria.

At visit 8/week 24, the primary efficacy endpoint will be assessed, which is the change from baseline in MCC.

If a subject is suffering from a symptomatic UTI in the week prior to any (un)scheduled urodynamic investigation (e.g., visit 5/week 4, visit 8/week 24), the UTI should be treated successfully first (until clinical recovery). To allow for treatment of the UTI, these visits may be postponed with an additional maximum of 7 days on top of the already existing visit window.

The 7-day e-diary does not have to be repeated if at least the 2-day weekend e-diary and 1 day of the weekday e-diary were completed while the subject did not suffer from a symptomatic UTI.

If a subject suffers from a symptomatic UTI in the week prior to any other study visit, these visits do not need to be postponed and the 7-day e-diary does not have to be repeated.

Sponsor: APEB ISN/Protocol 178-CL-206A

EudraCT number 2015-002876-25


#### Long-term Safety Period

For long-term safety evaluation, following visit 8/week 24, subjects will stay on their individual dose level until visit 10/week 52 (EOS or EOT).

#### **Dose Titration**

The aim is to obtain a safe low-pressure bladder, to inhibit overactive detrusor contractions and to reach continence.

Dose up-titration to PED50 must be performed at visit 4/week 2, visit 5/week 4 or visit 6/week 8, unless:

- 1. The investigator considers the subject to be effectively treated with PED25, based on urodynamics and the e-diary;
- 2. There are safety or tolerability issues with PED25.

Dose down-titration to PED25 can be performed at any time if there is a safety issue.

If an insufficient control of the NDO is observed at the highest tolerated mirabegron dose due to insufficient effect (based on, for example, ultrasound showing upper tract dilation; the appearance of a high grade reflux; high intravesical pressures; high detrusor pressures or high amplitude overactive contractions), the investigator should reconsider the subject's further participation in the study and consider an alternative treatment.

#### Inclusion/Exclusion Criteria:

Inclusion:

Subject is eligible for the study if all of the following apply:

- 1. Independent Ethics Committee (IEC)/Institutional Review Board (IRB)-approved written Informed Consent and privacy language as per national regulations must be obtained from the subject and/or from the subject's parent(s) or legal guardian(s) prior to any study-related procedures (including discontinuation of prohibited medication, if applicable); assent by the subject is given as required by local law.
- 2. Subject is male or female from 3 to less than 18 years of age.
- 3. Subject has a body weight of  $\geq 11$  kg.
- 4. Subject suffers from NDO confirmed by urodynamic investigation at baseline. The diagnosis of NDO must be confirmed by the presence of at least 1 involuntary detrusor contraction > 15 cm H<sub>2</sub>O from baseline detrusor pressure, and/or a decrease in compliance leading to an increase in baseline detrusor pressure of > 20 cm H<sub>2</sub>O.
- 5. Subject has been using CIC for at least 4 weeks prior to visit 1/screening.
- 6. Subject has a current indication for drug therapy to manage NDO.
- 7. Subject is able to take the study drugs in accordance with the protocol.
- 8. Female subject must either:
  - Be of nonchildbearing potential:
    - o Clearly premenarchal or in the judgment of the investigator is premenarchal,
    - o Documented surgically sterile,
  - Or, if of childbearing potential:
    - Agree not to try to become pregnant during the study and for 28 days after the final study drug administration,
    - And have a negative pregnancy test at visit 1/screening and at visit 3/baseline,
    - And, if sexually active must agree to use a highly effective method of birth control, which includes established use of oral, injected or implanted hormonal methods of contraception, OR placement of an intrauterine device (IUD) or intrauterine system (IUS). Birth control must be practiced from visit 1/screening and continuing throughout the study period, and for 28 days after the final study drug administration.

- 9. Male subject and their female spouse/partner who are of childbearing potential must be using a highly effective method of birth control, which includes established use of oral, injected or implanted hormonal methods of contraception, placement of an IUD or IUS. Birth control must be practiced from visit 1/screening and continuing throughout the study period, and for 28 days after the final study drug administration.
- 10. Female subject must not be breastfeeding from visit 1/screening until 28 days after last study drug administration.
- 11. Subject and subject's parent(s)/legal guardian(s) agree that the subject will not participate in another interventional study while participating in the study.
- 12. Subject and subject's parent(s)/legal guardian(s) are willing and able to comply with the study requirements and with the concomitant medication restrictions.

Waivers to the inclusion criteria will NOT be allowed.

#### Exclusion:

Subject will be excluded from participation if any of the following apply:

- 1. Subject has a known genitourinary condition (other than NDO) that may cause overactive contractions or incontinence (e.g., bladder extrophy, urinary tract obstruction, urethral diverticulum or fistula) or kidney/bladder stones or another persistent local pathology that may cause urinary symptoms.
- 2. Subject has one of following gastrointestinal problems: partial or complete obstruction, decreased motility such as paralytic ileus, subject at risk of gastric retention.
- 3. Subject has a urinary indwelling catheter within 4 weeks prior to visit 1/screening
- 4. Subject has a surgically treated underactive urethral sphincter
- 5. Subject has vesico-ureteral reflux grade 3 to 5.
- 6. Subject has undergone bladder augmentation surgery.
- 7. Subject receives electrostimulation therapy, if started within 30 days before visit 1/screening or is expected to start during the study period. Subjects who are on an established regimen may remain on this for the duration of the study.
- 8. Subject suffers from a symptomatic urinary tract infection (UTI) at baseline (symptomatic is defined as pain, fever, hematuria, new onset foul-smelling urine). If present at visit 1/screening or diagnosed between visit 1/screening and visit 3/baseline, the UTI should be treated successfully (clinical recovery) prior to baseline. If a symptomatic UTI is present at baseline, all baseline assessments should be postponed for a maximum of 7 days until the UTI is successfully treated (clinical recovery).
- 9. Subject has a (mean) resting pulse rate > 99<sup>th</sup> percentile [Fleming et al. 2011].
- 10. Subject has an established hypertension and a systolic or diastolic blood pressure greater than the 99th percentile of the normal range determined by sex, age and height, plus 5 mmHg [NIH 2005].
- 11. Subject has a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS]; or family history of LQTS, exercise-induced syncope).
- 12. Subject has severe renal impairment (estimated glomerular filtration rate [eGFR] according to Larsson equation < 30 mL/min).
- 13. Subject's aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is greater than or equal to 2 times the upper limit of normal (ULN) or total bilirubin greater than or equal to 1.5 times the ULN according to age and sex.

**Sponsor: APEB** EudraCT number 2015-002876-25


- 14. Subject has a history or presence of any malignancy prior to visit 1/screening.
- 15. Subject has known or suspected hypersensitivity to mirabegron, any of the excipients used in the current formulations or previous severe hypersensitivity to any drug.
- 16. Subject has participated in another clinical trial (and/or has taken an investigational drug) within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1/screening.
- 17. Subject uses any of the following prohibited medications (after start of washout):
  - Any medication, other than the study drug, used for the management of NDO;
  - Any drugs that are sensitive cytochrome (CYP) 2D6 substrates with a narrow therapeutic index or sensitive P-glycoprotein (P-gp) substrates
  - Any strong cytochrome P450 (CYP) 3A4 inhibitors if the subject has a mild to moderate renal impairment (eGFR 30 89 mL/min).
- 18. Subject has been administered intravesical botulinum toxin; except if given > 4 months prior to visit 1/screening and the subject experiences symptoms comparable to those existing prior to the botulinum toxin injections.
- 19. Subject has any other condition, which in the opinion of the Investigator, precludes the subject's participation in the study.
- 20. Subject's parent/legal guardian is an employee of the Astellas Group, the Contract Research Organization (CRO) involved, or the investigator site executing the study.

Waivers to the exclusion criteria will NOT be allowed.

## **Investigational Products:**

Mirabegron prolonged-release tablets, strengths 25 mg and 50 mg

Mirabegron oral suspension, strength 8 mg/mL

#### **Doses:**

#### Selection of the formulation:

Subjects with a body weight < 35 kg: mirabegron oral suspension.

Subjects with a body weight  $\geq$  35 kg: mirabegron tablets.

## Selection of the dose:

Doses are calculated weight-based. The bodyweight at visit 3/baseline determines the weight range for the starting dose (PED25) and the up-titration dose (PED50) to be used in the table below:

#### Weight-based Doses for Tablets or Suspension

| | Weight Range | Suspension Volume † | <b>Tablet Dose</b> |
|-------|--------------|---------------------|--------------------|
| | 11 - < 22 kg | 3 mL | - |
| PED25 | 22 - < 35 kg | 4 mL | - |
| | ≥ 35 kg | 6 mL | 25 mg |
| PED50 | 11 - < 22 kg | 6 mL | - |
| | 22 - < 35 kg | 8 mL | - |
| | ≥ 35 kg | 11 mL | 50 mg |

PED25: Pediatric equivalent dose 25 mg; PED50: Pediatric equivalent dose 50 mg † Suspension strength: 8 mg/mL

Sponsor: APEB ISN/Protocol 178-CL-206A

EudraCT number 2015-002876-25


#### Further dosing information:

- For subjects with a body weight ≥ 35 kg who do not want to or are unable to take tablets, the oral suspension can be supplied.
- At visit 8/week 24 subjects on mirabegron oral suspension may switch to tablets if the body weight turns to be ≥ 35 kg.
- Subjects receiving mirabegron tablets can switch to mirabegron oral suspension (and vice versa) for acceptability reasons after Sponsor's prior approval and on a case-by-case basis.

#### **Mode of Administration:**

Study drug will be taken orally, once a day in the morning around the same time of day and around time of food intake (i.e., within 1 hour before or after breakfast).

Mirabegron tablets will be taken with a sip of water (tablet should be taken as a whole and should not be chewed, divided or crushed).

Mirabegron oral suspension will be administered via an oral syringe with a sip of water afterwards. On visit days where a pharmacokinetic sample is planned in the clinic, completion of breakfast and study drug dosing should occur in the clinic.

# **Comparative Drug(s):**

Not applicable

# Dose(s):

Not applicable

#### **Mode of Administration:**

Not applicable

#### **Concomitant Medication Restrictions or Requirements:**

During the study, starting from visit 2 until visit 10/week 52 (EOT/EOS), subjects are not allowed to use treatment with any of the following prohibited medications:

- Any medication, other than the study drug, used for the management of NDO.
- Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index or sensitive P-gp substrates
- Any strong CYP 3A4 inhibitors if the subject has a mild to moderate renal impairment (eGFR 30 89 mL/min).

#### **Duration of Treatment:**

Once a day for 52 weeks

#### **Formal Stopping Rules:**

Criteria for treatment discontinuation for individual subjects:

- If, within 7 days of the first dose of mirabegron:
  - o The centrally read urodynamic trace reveals no evidence of NDO
  - The centrally read electrocardiogram (ECG) has an average QT interval corrected by Bazett's formula (QTcB) greater than 450 ms, based on the QTcB mean from the visit 1/screening and visit 3/baseline ECG triplicates
- If signs or symptoms of hypersensitivity to mirabegron are observed (e.g., anaphylactic reaction, erytheme multiforme or exfoliative dermatitis).

Discontinuation of treatment should be considered if:

- $\circ$  ALT or AST  $> 8 \times ULN$
- o ALT or AST  $> 5 \times ULN$  for more than 2 weeks
- o ALT or AST > 3  $\times$  ULN and TBL > 2  $\times$  ULN or INR > 1.5) (If INR testing is applicable/evaluated)

EudraCT number 2015-002876-25


- o ALT or AST > 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%).
- o In addition, if close monitoring for a subject with moderate or severe hepatic laboratory tests is not possible, the drug should be discontinued.

#### **Endpoints for Evaluation:**

#### **Primary:**

**Efficacy** 

Change from baseline in MCC after 24 weeks of treatment (based on filling urodynamics)

#### **Secondary:**

**Efficacy** 

### Based on filling urodynamics:

Change from baseline at visit 5/week 4 and visit 8/week 24 in:

- MCC (only visit 5/week 4)
- Bladder compliance  $(\Delta V/\Delta P)$
- Number of overactive detrusor contractions (> 15 cm H<sub>2</sub>0) until end of filling
- Detrusor pressure at end of filling
- Filling volume until first overactive detrusor contraction (> 15 cm  $H_20$ )

#### Based on e-diary:

Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) in:

- Average catheterized volume per catheterization
- Maximum catheterized volume
- Maximum catheterized daytime volume
- Average morning catheterized volume (based on first catheterization after subject woke up)
- Mean number of leakage episodes per day (day and night time)
- Number of dry (leakage-free) days/7 days (day and night time)

# Based on questionnaires:

- Change from baseline at visit 8/week 24 and visit 10/week 52 (EOT/EOS) in Pediatric Incontinence Questionnaire (PIN-Q)
- Change from baseline at visit 8/week 24 and visit 10/week 52 (EOT/EOS) in Patient Global Impression of Severity Scale (PGI-S)
- Acceptability questionnaire at visit 5/week 4, visit 8/week 24 and visit 10/week 52 (EOT/EOS)
- Clinician Global Impression of Change (CGI-C) at visit 8/week 24 and visit 10/week 52 (EOT/EOS)

#### Safety

- Incidence and severity of treatment-emergent adverse events (TEAEs)
- Change from baseline in vital signs (clinic measurements): systolic blood pressure, diastolic blood pressure, pulse rate and temperature at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS)
- Change from baseline in vital signs (self blood pressure measurement [SBPM]): systolic blood pressure, diastolic blood pressure, pulse rate at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) and on 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50 (visit 4/week 2, visit 5/week 4 or visit 6/week 8), if not already covered by the scheduled visit 4/week 2 and/or visit 5/week 4 SBPM.

- Change from baseline in hematology and biochemistry tests at visit 7/week 12 and visit 10/week 52 (EOT/EOS) and urinalysis tests at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS)
- Change from baseline in ECG parameters at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS)
- Change from baseline to visit 10/week 52 (EOT/EOS) in upper urinary tract ultrasound assessment
- Change from baseline in eGFR at visit 7/week 12 and visit 10/week 52 (EOT/EOS)

#### Pharmacokinetics of mirabegron

- C<sub>max</sub>, t<sub>max</sub>, AUC<sub>24</sub>, C<sub>trough</sub>, CL/F and V<sub>z</sub>/F.
- Additional pharmacokinetic parameters may be calculated based on the model used.

#### **Exploratory:**

Efficacy:

# Based on filling urodynamics:

Change from baseline at visit 5/week 4 and visit 8/week 24 in:

• Filling volume at 20 cm, 30 cm and at 40 cm H<sub>2</sub>O detrusor pressure, given that the pressures are reached during the examination.

#### Based on e-diary:

Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) in:

- Mean grade of leakage
- Total catheterized volume per day
- Change from baseline in SMIP-derived bladder compliance
- Number of CICs/day
- Responder in respect to leakage (complete, partial, no response)

Safety:

# <u>Intravesical pressure (SMIP):</u>

• Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS).

## Body weight and height:

• Change from baseline at visit 8/week 24 and visit 10/week 52 (EOT/EOS).

#### **Assessments:**

Urodynamic Assessments:

Subjects will undergo urodynamic assessment at baseline, visit 5/week 4 and visit 8/week 24. Additional urodynamic assessments can be performed at visit 10/week 52 (EOT/EOS), or at any other time point when deemed necessary by the investigator.

#### Patient-reported Outcome Data:

The following information will be collected and entered by the subject or the subject's parent(s)/caregiver(s) at home in the e-diary during the week preceding the visits as indicated in the Schedule of Assessments.

- Bladder diary:
  - o Each day for 7 days: time of CICs
  - o Each day for 7 days: presence of leakage between CICs

**Sponsor: APEB** EudraCT number 2015-002876-25


- o Each day for 7 days: sleep time and wake-up time
- On the 2 weekend days: catheterized volume
- On the 2 weekend days: SMIP (if applicable)
- o On the 2 weekend days: grade and number of leakages between CICs
- On the 2 weekend days (visit 3/baseline and visit 8/week 24): weight of diaper/pad
- SBPM (blood pressure and pulse rate):
  - o On the 2 weekend days: triplicate measurements in the morning and evening
  - o On 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM.
- Questionnaires: on 1 weekend day at selected visits
  - o PIN-Q
  - o PGI-S
  - Acceptability
- Confirmation of study drug intake: daily

The Investigator must guide the subject and subject's parent(s)/caregiver(s) to ensure that on the evening before and during the two weekend days of collection of catheterized volume and SMIP (if applicable), the subject's fluid intake should be regulated to an appropriate level taking e.g. age, sex and subject's condition into account. The intake must remain as consistent as possible on these volume collecting days throughout the entire study.

At the screening visit, detailed on-site training of the e-diary and the assessments and a booklet with operating instructions in local language will be provided to the subject and the subject's parent(s)/caregiver(s).

#### Pharmacokinetics:

When the subject reached steady state of her/his optimal dose, a total of 4 pharmacokinetic samples will be collected divided over 2 sampling days:

- Sampling day 1: 1 sample prior to dosing (i.e., trough sample).
- Sampling day 2: 1 trough and 2 postdose samples between 2h and 5h postdose, with at least 1 hour in between the samples.

On visit days where a pharmacokinetic sample is planned in the clinic, completion of breakfast and study drug dosing should occur in the clinic. Dosing must occur within 1 hour after completion of breakfast. Dosing time on the sampling day and dosing time of the previous day will be collected. In addition to the dosing time, the time of completion of breakfast, and type of breakfast will be collected in the eCRF on the sampling day with postdose sampling.

#### Safety:

During the study collection of adverse events (AEs), vital signs, body temperature, laboratory tests, ECG parameters, renal function, and height and weight will take place.

#### **Statistical Methods:**

# Sample size justification:

In order to allow the detection of a statistically significant change from baseline in MCC in the overall NDO with CIC study population with 90% power, 44 evaluable subjects for the assessment of the endpoint need to be enrolled, i.e., subjects with a valid (as by the central reviewer's assessment) nonmissing MCC measurement at baseline and at a postbaseline visit. The power calculation is based upon a paired t-test with a 2-sided significance level of 0.05, an expected change from baseline of at least 52 mL and a SD of not larger than 103 mL. Assuming 30% of enrolled subjects will not be evaluable, a total of approximately 63 subjects may need to be enrolled.

Four analysis populations will be defined: the safety analysis set (SAF), full analysis set (FAS), per protocol set (PPS), and pharmacokinetics analysis set (PKAS) for pharmacokinetic population analysis.

Sponsor: APEB ISN/Protocol 178-CL-206A

EudraCT number 2015-002876-25


## Efficacy:

The primary analysis will be a paired t-test for the change from baseline to visit 8/week 24 for subjects included in the FAS to test the hypothesis that the change from baseline in MCC is not equal to zero with a 2-sided alpha level of 0.05. A 95% CI will be calculated for mean change from baseline and it will be assessed whether the estimated lower bound of the interval is greater than zero. Additionally 95% CIs per age group will be presented.

Continuous secondary efficacy variables will be analyzed in the same way as the primary efficacy variable. Discrete secondary efficacy variables will be analyzed descriptively.

#### Pharmacokinetics:

Pharmacokinetic parameters will be summarized for the PKAS using descriptive statistics.

#### Pharmacodynamics:

Not applicable.

# Safety:

Safety endpoints will be summarized for the SAF using descriptive statistics. Safety parameters such as vital signs, height and weight will also be summarized with respect to age- and sex-specific percentiles.

#### Other Analyses:

Descriptive statistics will be used to explore whether there is an association between certain subject characteristics (such as medical history) and the final titrated mirabegron doses. Collected data on study drug compliance rates and maintenance of treatment will be analyzed using descriptive statistics

#### Interim analyses:

Not applicable.

Sponsor: APEB ISN/Protocol 178-CL-206A

EudraCT number 2015-002876-25


# V. FLOW CHART AND SCHEDULE OF ASSESSMENTS

#### Flow Chart

| | Study Period<br>(56 weeks) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Pretreatment Period<br>(4 weeks) | | | Efficacy Treatment Period † (24 weeks) | | | | | Long-term Safety Period ‡ (28 weeks) | |
| Visit 1 | Visit 2/TC 1 | Visit 3 | Visit 4/TC 2<br>Week 2 | Visit 5<br>Week 4 | Visit 6/TC 3<br>Week 8 | Visit 7<br>Week 12 | Visit 8<br>Week 24 | Visit 9/TC 4<br>Week 36 | Visit 10/EOS<br>Week 52 |
| Screening | Group A & B §: Review of 2-day e-diary Group B: Start washout on day -15 | Baseline | 1 <sup>st</sup> up-titration<br>possibility | 2 <sup>nd</sup> up-titration<br>possibility | 3 <sup>rd</sup> up-titration<br>possibility | Fixed dose | Fixed dose | Fixed dose | End of Study |

TC: telephone contact; EOS: end of study

- † The efficacy treatment period begins with the first dose, the day after baseline measurements on visit 3/baseline.
- † The long-term safety period begins immediately after visit 8/week 24.
- § Group A: Subjects who are currently not receiving any prohibited medication including any oral drug treatment to manage their NDO, or when botulinum toxin is no longer considered effective. Group B: Subjects who currently are receiving oral drug treatment to manage their NDO or receive any other prohibited medication.

Sponsor: APEB
ISN/Protocol 178-CL-206A

EudraCT number 2015-002876-25


 Table 1
 Schedule of Assessments

| | Visit 1 | Visit 2 /TC 1 <sup>†</sup> | Visit 3 | Visit 4<br>/TC 2 <sup>†</sup> | Visit 5 | Visit 6<br>/TC 3 <sup>†</sup> | Visit 7 | Visit 8 | Visit 9<br>/TC 4 <sup>†</sup> | Visit 10<br>/EOS <sup>‡</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Screening | Start of<br>Washout ††† | Baseline | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | Week 36 | Week 52 |
| | Day -28 to<br>Day -15 | Day -15 to<br>Day -8 | Day -1 | Day 14<br>(+3 days) | Day 28<br>(+3 days) | Day 56<br>(±7 days) | Day 84<br>(±7 days) | Day 168<br>(±7 days) | Day 252<br>(±14 days) | Day 364<br>(±14 days) |
| Signing informed consent form | X | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | X | | | | | | | |
| Demographics | X | | | | | | | | | |
| Height & weight | X | | X | | | | | X | | X |
| Medical history (including NDO) | X | | | | | | | | | |
| Current NDO medications | X | X | | | | | | | | |
| Vital signs (triplicate) and body temperature (ear) § | X | | x | | X | | x | X | | x |
| Physical examination | X | | | | | | | | | X |
| 12-lead ECG (triplicate) ¶ | X | | X | | X | | X | X | | X |
| Hematology/Biochemistry/eGFR | X | | (X) <sup>††</sup> | | (X) <sup>††</sup> | | X | | | X |
| Urinalysis | X | | X | | X | | X | X | | X |
| Pregnancy test <sup>‡‡</sup> | X | | X | | X | | X | X | | X |
| Pharmacokinetics §§ | | | | | (X) | (X) | (X) | (X) | (X) | (X) |
| Upper urinary tract ultrasound | | | X | | | | | | | X |
| Urodynamic assessments ¶ | | | X | | X | | | X | | |
| Dose-titration assessment | | | | X | X | X | | | | |
| Dispense study drug ††† | | | X | | X | | X | X | (X) | |
| Bladder diary, SMIP and collection of catheterized volume <sup>‡‡‡</sup> | | X | X | X | X | Х | X | Х | X | х |
| SBPM (triplicate) §§§ | | X | X | X | X | X | X | X | X | X |
| PIN-Q, PGI-S | | | X | | | | | X | | X |
| CGI-C | | | | | | | | X | | X |
| Acceptability questionnaire | | | | | X | | | X | | X |
| Adverse events and previous and | | | | | | | | | | |
| concomitant medication | | | | | | | | | | |

ECG: Electrocardiogram; EOS: end of study; CGI-C: Clinician Global Impression of Change scale; DSMB: Data and Safety Monitoring Board; NDO: neurogenic detrusor overactivity; PGI-S: Patient Global Impression of Severity Scale; PIN-Q: Pediatric Incontinence Questionnaire; SBPM: self blood pressure measurement; SMIP: self-measurement of intravesical pressure; TC: telephone contact. Table footnotes continued on next page

Sponsor: APEB
ISN/Protocol 178-CL-206A

EudraCT number 2015-002876-25


† For the visits where a TC is indicated there is no need for the subject to visit the clinic, provided that the e-diary data is reviewed by the investigator prior to the TC and discussed and confirmed with the subject or the subject's parent(s)/caregiver(s) during the TC.

- \$\frac{1}{2}\$ Subjects who withdraw early from the study after having received study drug should complete the EOS visit. If the final dose is reached before the last possibility for up-titration at 8 weeks, the fixed-dose treatment period will be extended to keep the entire treatment period 364 days as a minimum. The maximum is 378 days in order to allow for visit windows.
- § Triplicate vital signs with an interval of approximately 2 minutes in the sitting position (when possible, otherwise supine, but always in the same position). Preferably the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Clinic measurements will be used to assess eligibility. Single measurements for body temperature must be performed with an ear thermometer.
- ¶ Triplicate 12-lead ECG with an interval of about 30 seconds to 5 minutes in the supine position (when possible, but always in the same position). Subject should have been calm and without distress for at least 5 minutes.
- †† Additional hematology/biochemistry taken at baseline only if an AE related to hematology/biochemistry parameters occurred between visit 1/screening and visit 3/baseline. The first group of subjects (minimum of 5, maximum of 10) who reach study visit 5/week 4 will have an additional blood draw for a DSMB-mandated interim safety check at this visit. For sampling, preferably the left arm should be used. Blood sampling should occur after vital signs and ECG measurements.
- ‡‡ Pregnancy test in female subjects of childbearing potential in serum (if blood is drawn) or urine (at other visits).
- §§ If the subject reached steady state of her/his optimal dose, a total of 4 pharmacokinetic samples will be collected, divided over 2 sampling days. Sampling day 1: 1 trough sample; Sampling day 2: 1 trough and 2 postdose samples between 2 h and 5 h postdose, with at least 1 hour in between the samples. These 2 sampling days do not have to be in a specific order and can be selected from the given options. To allow for an early assessment of the dose-response relationship by the DSMB, it is preferred the pharmacokinetic sampling takes place as early in the study as possible. Dosing on a sampling day with postdose samples must occur within 1 hour after completion of breakfast [Section 5.3.4]. On days where a pharmacokinetic visit is planned in the clinic, breakfast and dosing should occur in the clinic. Blood sampling should occur after vital signs and ECG measurements.
- ¶¶ Additional urodynamic assessments may be performed if deemed necessary by the investigator.
- ††† Daily study drug administration will begin on Day 1 (the day after visit 3/baseline). Due to shelf-life limitations, an additional dispensing visit is foreseen at visit 9/week 36 for subjects receiving mirabegron oral suspension. This dispensing visit does not need to be accompanied by the subject.
- After a successful screening visit, all subjects start with the completion of a 2-day weekend e-diary visit to get acquainted with the e-diary and the assessments. Completion of this diary should start in the weekend prior to visit 2. Completion of subsequent bladder diaries should start approximately 7 days prior to the indicated visit (or TC). If successful completion of the 2-day weekend e-diary is confirmed at visit 2, subjects from group A start with collection of the 7-day baseline e-diary, followed by the baseline visit. Subjects in group B start with a 14-day washout. In the second week of the washout period, collection of their 7-day baseline e-diary starts, followed by the baseline visit.
- §§§ Triplicate SBPM will be performed in the morning and evening during the 2-day weekend e-diary collection period and on 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM. Measurements to be taken with an interval of approximately 2 minutes in the sitting position (when possible, otherwise supine, but always in the same position). Preferably the right arm should be used. Morning measurements should be taken after waking-up, before breakfast and before study drug intake, evening measurements prior to bedtime. Subject should have been calm and without distress for at least 5 minutes.

Sponsor: APEB

EudraCT number 2015-002876-25


# 1 INTRODUCTION

# 1.1 Background

Protocol 178-CL-206A is part of the Sponsor's clinical program to develop mirabegron for neurogenic detrusor overactivity (NDO) and overactive bladder (OAB) in pediatric patients. In the EU the development of mirabegron for the indication of NDO is outlined in the pediatric investigation plan (PIP) for mirabegron and approved by the Pediatric Committee (PDCO).

In the US, the protocol 178-CL-206 is planned to fulfill the Pediatric Research Equity Act (PREA) requirement commitment and the Proposed Pediatric Study Request (PPSR).

Protocol 178-CL-206A will start in the regions as mentioned in the synopsis. Protocol 178-CL-206 will start later in the US after review and approval of further mirabegron data by the FDA. Protocol 178-CL-206A and 178-CL-206 will be kept identical and subject data from both protocols will be pooled and analyzed as outlined in the statistical section of the protocol [see Section 7].

The population for this pediatric clinical efficacy study with mirabegron is children and adolescents with NDO who require clean intermittent catheterization (CIC). NDO is defined by the International Children's Continence Society as detrusor overactivity when there is a relevant neurologic condition. "Detrusor overactivity is the occurrence of involuntary detrusor contractions during filling cystometry. They may be spontaneous or provoked and produce a waveform of variable duration and amplitude. Contractions may be phasic or terminal. Symptoms of urgency and/or urgency incontinence may or may not occur" [Austin et al, 2014].

NDO can develop as a result of a lesion at any level in the nervous system, including the cerebral cortex, spinal cord, or peripheral nervous system. In 85% of the children with NDO, the condition is caused by myelomeningocoele (spina bifida) [Bauer et al, 2012]. In a subset of NDO patients (typically patients who suffer from detrusor sphincter dyssynergia [DSD] or have a surgically repaired underactive sphincter), treatment requires constant and fastidious bladder management from shortly after birth, including performance of CIC [Bauer et al, 2012]. Performance of CIC ensures that bladder volumes are regularly reduced to zero, thereby decreasing end-filling bladder pressure.

In the population of NDO patients requiring CIC, the medical need for treatment is the highest, due to the underlying pathophysiology of the urinary tract. In these patients, the overactive detrusor contracts against a closed or partially closed sphincter instead of a relaxed sphincter, due to DSD and/or sphincter surgery. The consequence is that these children cannot void normally, but instead leak when the pressure in the bladder exceeds the sphincter pressure (incontinence). This is independent of age and bladder training.

If left untreated, NDO leads to deterioration of urinary tract function at early age. Kidney function deteriorates from hydronephrosis due to backpressure caused by high (end-filling) bladder pressure. Further renal damage can occur from ascending urinary tract infections

Sponsor: APEB
EudraCT number 2015-002876-25


(UTIs) resulting from vesico-urethral reflux. Fibrosis of the bladder wall, induced by strong and uninhibited overactive contractions and frequent UTIs, contributes to the development of a noncompliant bladder (loss of expansile capability; high pressures at low volumes). In a noncompliant bladder, the critical level of detrusor pressure is reached at lower filling volumes, further predisposing the patient to kidney damage.

Current drug therapy consists of oral antimuscarinics or botulinum toxin injected into the bladder wall. The drug therapy decreases end-filling pressure, overactive contractions and increases bladder capacity and as such protects against kidney damage and deterioration of bladder wall. Although to date, the vast majority (approximately 90%) of patients can be treated successfully with the gold standard treatment of oxybutynin (oral or intravesical) and CIC [Verpoorten et al, 2008], development of alternative therapy is desirable because of insufficient efficacy and/or the side effects of antimuscarinics; dry mouth, constipation, blurred vision, headache, tiredness (somnolence), impaired school performance, facial flushing, gastrointestinal discomfort, and dry itchy skin [Rawashdeh et al, 2012] and the invasive administration of botulinum toxin, which is bothersome for the patient.

Mirabegron, a beta-3 adrenergic receptor agonist, represents a new class of drugs for treatment of OAB. The use of mirabegron as an alternative therapy to control detrusor overactivity in patients with NDO has not yet been established, although some reports of a positive effect of mirabegron on urodynamic parameters in patients with NDO have been published [Wöllner et al, 2015; Wada et al, 2015; Skobejko 2014].

## 1.2 Nonclinical and Clinical Data

Detailed information on studies conducted with mirabegron can be found in the most recent pediatric mirabegron Investigator's Brochure (IB). Nonclinical and clinical data are also summarized in the package insert for mirabegron (current locally-available product information for mirabegron).

Summaries of findings from nonclinical and clinical studies with mirabegron which have relevance for the current study are presented below.

#### 1.2.1 Nonclinical Data

The primary pharmacology studies showed that mirabegron induced bladder relaxation during the filling phase and inhibited the frequency of nonvoiding activity. Other pharmacological effects, such as the glucogenolytic effects of mirabegron in rodents, did not translate to any effect in adult humans.

The safety pharmacology and toxicological studies showed that the safety profile of mirabegron, when administered to achieve exposures similar to those seen at the maximum recommended human dose, compares favorably with the currently approved antimuscarinic drug therapies indicated for the treatment of OAB.

The 39 toxicology studies that have been conducted with mirabegron in adult mice, rats, rabbits, dogs and cynomolgus monkeys support the safety of mirabegron for the treatment of OAB in adults and adolescents. The ages of the rats and monkeys that were used in the

02 Nov 2016 Astellas 

nonclinical repeated-dose toxicity studies were 8 weeks and 3 to 4 years old, respectively, which corresponds to a human age of 12 to 13 years. In support of clinical trials in children from 6 months of age and older, 2 repeated-dose toxicity studies were conducted in 10-day-old juvenile rats (postnatal day 10 [PND10]): a 14-day oral dose range-finding study (Study 178-TX-054) and a 13-week oral repeated dose toxicity study with a 4-week recovery period (Study 178-TX-055).

Modest elevation of alanine aminotransferase (ALT) was observed in monkeys, but the changes observed were below the level of toxicological significance, and there were no changes in liver histopathology. There were no significant changes in liver enzymes or liver histopathology in dogs. In the toxicology studies in juvenile rats, increased activities in aspartate aminotransferase (AST) and ALT were noted in male rats at doses of 30 mg/kg (22-fold higher than the maximum recommended human dose). Modest (less than 2-fold) increases in plasma alkaline phosphatase (ALP) were observed at high doses (72-fold higher than the maximum recommended human dose), together with reversible changes in hepatocytes. Single and repeated dose toxicology studies in dogs, monkeys and rats demonstrated cardiovascular changes at high doses (please refer to the mirabegron IB).

In rodents, beta 3-agonists have an anti-obesity effect due to an increase in metabolic rate due to the activation of thermogenesis in brown adipocytes and to lipolysis in white adipocytes [Lafontan & Berlan, 1993]. In adult and juvenile rats treated with > 10 mg/kg mirabegron, decreased lipid droplets were observed in the brown adipose tissues and white adipose tissues. In addition, behavioral effects like decreased activity, which could be related to an increased body temperature, were also observed in juvenile rats in males and females in the 10 and 30 mg/kg groups. However, no comparable effect in primates was seen. In clinical studies with mirabegron in adults no effects on weight or body temperature have been observed. In healthy subjects, neither single nor repeat dose administration affected mean blood glucose, C-peptide, triglyceride, insulin levels or oral temperature compared with placebo, suggesting that mirabegron does not affect lipid or glucose metabolism in healthy subjects. In subjects with type 2 diabetes mellitus, mirabegron induced no substantial changes from baseline in body weight or oral temperature. However, since brown adipose tissue is more prevalent in children than in adults, it could be that brown adipose tissue has a greater physiological role in children than in adults. Therefore, it cannot be excluded that administration of mirabegron has an effect on body weight and/or body temperature in young children.

In the toxicology studies, increased activities in aspartate aminotransferase (AST) and ALT were noted in male rats at doses of 30 mg/kg (22-fold higher than the maximum recommended human dose). Modest (less than 2-fold) increases in plasma alkaline phosphatase (ALP) were observed at high doses (72-fold higher than the maximum recommended human dose), together with reversible changes in hepatocytes.

Mirabegron was not found to be genotoxic, carcinogenic, or teratogenic in the battery of in vitro and in vivo studies. The in vitro oxidative metabolism of mirabegron in human liver microsomes is primarily mediated by cytochrome P450 (CYP) 3A4, but a possible role for

**Sponsor: APEB** EudraCT number 2015-002876-25


CYP2D6 could not be excluded. In vitro CYP inhibition studies suggest that mirabegron is a moderate and time-dependent inhibitor of CYP2D6 and a weak inhibitor of CYP3A4.

Exposure levels in juvenile (PND10) rats were 5-fold to 10-fold increased compared to adult rats (PND100). The exposure levels of mirabegron in young (PND21) and adolescent (PND45) rats were 2-fold to 5-fold lower than the exposures observed in the adult rats (PND100). The increased exposure levels of mirabegron on PND10 and decreased exposure levels on PND21 and PND45 are in line with the knowledge on the ontogeny of drug metabolizing (phase I and phase II) enzymes and (efflux) transporters in rats [de Zwart et al, 2008; Saghir et al, 2012]. This could translate into differences in exposures between adults/adolescents and pediatric subjects, in which the phase I (until 2 years of age) and/or phase II (until 11 years of age) enzymes are still maturing.

#### 1.2.2 Clinical Data

The main clinical aspects of mirabegron prolonged-release tablets in adults are described in the current locally-available product information for mirabegron.

To support the doses and formulations (tablets and oral suspension) selected for this study, the pediatric development program for mirabegron includes 4 phase 1 studies [Table 2].

Table 2 Overview of Current Supporting Mirabegron Studies in the Pediatric Clinical Development Program for NDO and OAB

| Study Number | Study Title | Study Progress |
|---|---|---|
| 178-CL-201 | A phase 1, single dose, 4-period crossover study to assess the bioavailability of mirabegron oral suspension relative to the mirabegron prolonged-release tablet and to assess the effect of food on the pharmacokinetics of mirabegron oral suspension in healthy young male and female subjects. | Completed |
| 178-CL-202 | A multicentre, open-label, single ascending dose phase 1 study to evaluate the pharmacokinetics, safety and tolerability of mirabegron OCAS tablets in pediatric subjects from 5 to less than 18 years of age with neurogenic detrusor overactivity (NDO) or overactive bladder (OAB). | Completed |
| 178-CL-203 | A multicentre, open-label, single dose, phase 1 study to evaluate the pharmacokinetics, safety and tolerability of mirabegron oral suspension in pediatric subjects from 3 to less than 12 years of age with neurogenic detrusor overactivity (NDO) or overactive bladder (OAB). | Ongoing |
| 178-CL-208 | A phase 1, single dose, 3-period crossover study to assess the bioavailability of an oral suspension of 8 mg/mL mirabegron relative to the oral suspension of 2 mg/mL mirabegron and to assess the effect of food on the pharmacokinetics of the oral suspension of 8 mg/mL mirabegron in healthy male and female adult subjects | Ongoing |

The results of studies 178-CL-201 and 178-CL-202 are reported in the most recent version of the pediatric IB. The data from these studies were used to support the use of tablets in pediatric subjects with a body weight of  $\geq$  35 kg in this study.

**Sponsor: APEB** EudraCT number 2015-002876-25


For those pediatric subjects that cannot be dosed with tablets because their body weight is 35 kg or less or because they cannot swallow tablets, an oral suspension with a strength of 2 mg/mL was developed. The relative bioavailability was assessed in healthy subjects (178-CL-201) to be 53.44% lower compared to tablets. The results of this study and study 178-CL-202 was used to support the use of the 2 mg/mL in study 178-CL-203.

That study is a single dose phase 1 study with mirabegron oral suspension in pediatric subjects from 3 to less than 12 years of age with NDO and in pediatric subjects from 5 to less than 12 years of age with OAB. This study is currently ongoing with 6 of 9 planned subjects having completed the study. Single doses of mirabegron are administered that are predicted to result in an exposure comparable to that in adults when dosed with 50 mg mirabegron tablets once daily at steady-state (188 ng·h/mL). Subjects received mirabegron oral suspension within 1 hour after a light breakfast. Doses were compensated for the lower bioavailability of suspension versus tablets (see above). This study is ongoing but the preliminary results are provided below.

It became apparent that with a strength of 2 mg/mL the volume of the doses the patients have to take every day would be too high (up to 44 mL). To overcome this issue, an oral suspension of 8 mg/mL was developed.

To support the use of this 8 mg/mL mirabegron oral suspension in pediatric subjects, study 178-CL-208 was conducted. The study follows a single dose, three period cross over design in healthy subjects. Subjects received the following three treatments in random order: 1) 11mL 8 mg/mL oral suspension of mirabegron under fasted conditions, 2) 11mL 8 mg/mL oral suspension of mirabegron under fed conditions and 3) 44 mL 2 mg/mL oral suspension of mirabegron under fasted conditions. This study is ongoing, but a summary of the preliminary results is provided below.

## Exposure:

The single doses of the 2 mg/mL oral suspension for Study 178-CL-203 were predicted using a population pharmacokinetic (popPK) model developed on pharmacokinetic data obtained in Study 178-CL-201, with food, dose, and formulation effects on the bioavailability, and was validated on data from Study 178-CL-202. The observed exposures were in line with the target exposure of 188 ng·h/mL; the median AUC<sub>24</sub> was 207 ng·h/mL (n=6, mean (SD): 226.4 (152.3), range: 39.7-467). These preliminary results suggest that the use of the popPK model is appropriate for dose selection. The model predictions of the PED50 doses at a strength of 2 mg/mL would require large volumes of oral suspension every day (up to 44 mL). Therefore, to reduce the volume, a higher strength oral suspension was developed.

The primary objective of study 178-CL-208 was to assess the relative bioavailability of the 8 mg/mL oral suspension compared to the 2 mg/mL oral suspension under fasted conditions. The results of study 178-CL-208 show that the bioavailability of both strengths is comparable Table 3.

Sponsor: APEB

EudraCT number 2015-002876-25


Table 3 178-CL-208 Draft Results: Relative Bioavailability of the Mirabegron 8 mg/mL Oral Suspension Formulation versus 2 mg/mL Oral suspension Formulation (Pharmacokinetics Analysis Set)

| Parameter (units) | Geometric LS Mean for<br>8 mg/mL Suspension<br>Fasted<br>(n=24) | Geometric LS Mean for<br>2 mg/mL Oral Suspension<br>Fasted<br>(n=23) | Geometric LS<br>Mean Ratio<br>(%)† | 90% CI of<br>Ratio (%)† |
|---|---|---|---|---|
| AUC <sub>inf</sub> (ng•h/mL) | 253 | 251 | 100.6 | (90.9, 111.3) |
| AUC <sub>last</sub> (n•.h/mL) | 234 | 232 | 100.9 | (90.6, 112.4) |
| C <sub>max</sub><br>(ng/mL) | 12.1 | 11.3 | 106.7 | (84.2, 135.2) |

CI: confidence interval; LS: least squares.

The analysis was performed on log-transformed pharmacokinetic parameters using a linear mixed model with treatment and investigational period as fixed effects and accounting for the longitudinal nature of the data by subject using a REPEATED statement. The covariance matrix is structured by period.

The information obtained in studies 178-CL-203 and 178-CL-208 was taken into account when predicting the doses for this study as outlined in Section 2.2.2 of this protocol.

The doses described in Section 2.2.2 suggest tablets for pediatric subjects with a body weight of  $\geq$  35 kg, and the 8 mg/mL oral suspension for children with a body weight between 11 and 35 kg, or for those subjects with a body weight  $\geq$  35 kg who do not want to or are unable to take tablets.

## Safety and tolerability:

In study 178-CL-203 the safety and tolerability of the oral suspension when dosed in children was evaluated and it was concluded that it was safe and well tolerated.

From the 6 subjects who completed the study (3 with NDO and 3 with OAB) 1 treatment emergent adverse event (TEAE) was reported: pyrexia on day 1 in a NDO subject. The intensity was mild and was judged by the investigator not to be related to study drug. No clinically significant electrocardiogram (ECG) abnormalities have been seen throughout the study, there were no QTcF values > 450 ms and no QTc prolongation > 30 ms versus baseline was observed (mean of triplicates).

Increases in vital signs have been observed but these were not considered clinically significant per investigator's assessment.

A 24-hour Holter recording was recorded in all subjects on a reference day and on the dosing day. The main objective of the Holter recording was to evaluate the effect of mirabegron on heart rate in a time-matched manner, taking into account the circadian rhythm. A median increase in 24-hour heart rate of 5.1 bpm has been observed. This was not considered as

<sup>†</sup> The geometric LS mean ratios (and associated 90% CIs) were obtained by back-transforming (antilogging) the LS means of the treatment differences.

**Sponsor: APEB**EudraCT number 2015-002876-25


clinically relevant taken into account the multiple blood draws, the low number of subjects and the absence of a placebo group.

Some changes in laboratory values were observed, but they were not considered as clinically relevant.

For Study 178-CL-208 single doses of 88 mg mirabegron oral suspension to adults were safe and well tolerated. Eleven of 24 subjects reported 22 adverse events (AEs). All except for 2 events (1 headache moderate and 1 dysmenorrhea moderate) were mild. 20 AEs were considered not related; 2 were considered possibly related (dizziness, mild and orthostatic dizziness mild).

# 1.3 Summary of Key Safety Information for Study Drugs

Mirabegron has not been approved or marketed for use in pediatric subjects.

For further information reference is made to the most recent version of the pediatric IB for mirabegron, and current locally-available product information for mirabegron.

Mirabegron has been approved in more than 65 countries worldwide. In adults, the safety of mirabegron treatment has been well characterized in 5863 subjects (95% with overactive bladder) in the phase 2/3 registration studies treated with mirabegron at doses ranging from 25 to 200 mg once daily. Identified risks include increased heart rate and tachycardia, hypersensitivity reactions, increased blood pressure and urinary retention. Potential risks include QT prolongation, UTI, fetal disorders after exposure during pregnancy and events induced by concomitant treatment with CYP2D6 substrates with a narrow therapeutic index. The risks of QT prolongation, increased heart rate or increased blood pressure are greater with increasing exposure at supratherapeutic doses and can be mitigated with optimal dose selection. The maximum therapeutic dose of mirabegron based on the overall benefit-risk is 50 mg once daily in adults.

## 1.4 Risk-Benefit Assessment

Mirabegron tablets have a favorable risk-benefit profile in adults in the indication OAB. Mirabegron oral suspension has been shown to be safe and well tolerated in 2 phase 1 studies in healthy adult subjects (Studies 178-CL-201 and 178-CL-208). In the pediatric phase 1 studies executed thus far, mirabegron tablets and mirabegron oral suspension had an acceptable safety profile and were well tolerated.

Successful management of NDO prevents the occurrence of progressive kidney impairment and decrease in bladder compliance in subjects with NDO. As such, the benefit of successful treatment in this subject population is large, and is expected to be larger than in subjects suffering from OAB, provided that mirabegron is effective and has an acceptable safety profile in this population.

The use of mirabegron as an alternative therapy to control detrusor contraction in subjects with NDO has not yet been established. However some reports have been published showing a positive effect of mirabegron on urodynamic parameters in patients with NDO [Wöllner et

02 Nov 2016 Astellas 

al, 2015; Wada et al, 2015; Skobejko 2014]. Beneficial effects are also expected on gaining continence.

The major risk in this study is periods of uncontrolled high end-filling detrusor pressure. This risk is monitored on a regular basis and can be mitigated by the investigator as follows:

- A washout period is necessary to achieve an adequate baseline. The washout period has been restricted to 2 weeks in order to prevent renal damage and minimize the burden for the subject. At baseline a urodynamic investigation is planned, allowing the investigator to judge the risk to the subject in case mirabegron would not be efficacious. At this stage the risk can be mitigated by increasing the CIC frequency.
- The initial dose of mirabegron will be based on the subject's weight, and predicted to achieve plasma concentrations equivalent to the steady state exposures expected with 25 mg mirabegron administered once daily in adults (pediatric equivalent dose [PED] 25). This low dose is chosen considering possible beta-adrenergic side effects of mirabegron.
- After 2 weeks on PED25 all subjects will be up-titrated to PED50 unless there is a safety
  issue with mirabegron or the investigator considers that with the low mirabegron dose full
  efficacy has been reached. By striving to get an efficacious dose of mirabegron early after
  start of dosing, the risk for bladder and kidney damage is mitigated.
- At 4 weeks of therapy, a second urodynamic investigation allows the investigator to judge and mitigate the risk by increasing the dose in subjects without prior dose increase or, in subjects on the maximum dose, by increasing the CIC frequency or by withdrawal of the subject.
- Additional urodynamic assessments may be performed at any time in the study if deemed necessary by the investigator.

Concerning drug safety, important identified or potential risks in adults and their monitoring in this study are listed below:

- Increased heart rate and tachycardia is monitored in this study by at-home measurement of vital signs and measurement of vital signs at the study visits at the center;
- Hypersensitivity reactions (immediate or nonimmediate and cutaneous or noncutaneous) are monitored in this study by AE monitoring;
- Increased blood pressure is monitored in this study by at-home measurement of vital signs and measurement of vital signs at the study visits at the center;
- Urinary retention does not apply in children on CIC;
- Potential QT prolongation is monitored by ECG at each visit at the center;
- Potential urinary tract infection is monitored by urine analysis at each visit in the center;
- Potential fetal disorders after exposure during pregnancy is mitigated by the inclusion criteria;
- Potential events by concomitant treatment with CYP2D6 substrates with narrow therapeutic index is mitigated by excluding these medications;
- Although not observed in adults, the potential activation of thermogenesis will be monitored by temperature measurement. Weight loss due to activation of thermogenesis in brown fat will be monitored by regular weight measurements.
EudraCT number 2015-002876-25


Regarding the formulations to be administered: for both the tablet and the oral suspension formulation, all excipients are pharmaceutical grade materials and are considered safe for the intended pediatric population. Their concentrations remain below the acceptable daily intake as set by the Joint Food and Agriculture Organization of the United Nations (FAO) and the World Health Organization (WHO) (JECFA) [FAO 2015].

The protocol is designed to minimize the burden to the subject by restricting the number of urodynamic investigations, the number of blood draws (safety and pharmacokinetic sampling) and the number of study visits to a minimum.

The use of popPK for the analysis of the pharmacokinetic profile of mirabegron allows reducing the number of blood draws for pharmacokinetic analysis to 4. Butterfly needles can be used and are allowed to stay in place to reduce the number of punctures.

The blood draws for safety assessment have been reduced by omitting a baseline safety blood draw in subjects where the hematology and biochemistry results obtained at the screening visit did not show significant abnormalities and no AEs occurred after the screening visit that could influence the hematology/biochemistry results.

The assessments to be performed are routine assessments and generally do not pose any particular risk to the subjects. Every effort will be made to reduce the anxiety felt by subjects, e.g., during a blood test, topical anesthetic will be offered at venipuncture to minimize distress of the subject. The investigator should not include any subject for whom it is expected that their condition will not allow protocol compliance.

Subjects may experience AEs associated with the assessments performed during the study, such as local irritations due to ECG recording, and bleeding, hematoma as a result of blood collection, or the experience of transient stinging or burning during emptying or of the passing of a little blood as a result of the urodynamic investigation. There is also a small risk of developing a bladder infection in relation to the urodynamic procedure.

Data and Safety Monitoring Board (DSMB) assessment including review of safety and efficacy (no, or insufficient efficacy is a safety risk) is planned after the first 5 subjects have reached visit 5/week 4 allowing a risk /benefit assessment early after start of the study. In case the DSMB cannot reach a verdict based on the safety samples of these 5 subjects, this group will be increased with 5 more subjects, to obtain a maximum of 10 visit 5/week 4 safety samples for early DSMB assessment. In the DSMB charter detailed information can be found. In view of the above considerations, the risk-benefit ratio for this study is considered to be acceptable for the subjects that will participate in this study.

Sponsor: APEB
EudraCT number 2015-002876-25


### 2 STUDY OBJECTIVE(S), DESIGN, AND ENDPOINTS

## 2.1 Study Objectives

## 2.1.1 Primary Objectives:

• To evaluate the efficacy of mirabegron after multiple-dose administration in the pediatric population.

### 2.1.2 Secondary Objectives:

- To evaluate the safety and tolerability of mirabegron after multiple-dose administration in the pediatric population.
- To evaluate the pharmacokinetics of mirabegron after multiple-dose administration in the pediatric population.

## 2.2 Study Design and Dose Rationale

## 2.2.1 Study Design

This is a phase 3, open-label, baseline-controlled, multicenter study in male and female children and adolescents aged 3 to less than 18 years of age with NDO on CIC. Approximately 50 enrolling study centers in Europe, Latin America, Africa, Middle East and Asia-Pacific are planned.

At least 44 evaluable subjects (estimate of 63 enrolled), with at least 10 subjects from each age group (children aged 3 to less than 12 years of age; adolescents aged 12 to less than 18 years of age) are planned. A subject is considered being evaluable if the subject has a valid (as by the central reviewer's assessment) nonmissing maximum cystometric capacity (MCC) measurement at baseline and at a postbaseline visit. An enrolled subject withdrawing or discontinuing before dosing will be replaced. A subject discontinuing treatment after dosing can be replaced at the discretion of the Sponsor. The study is conducted under the aegis of a DSMB.

The study will consist of 3 periods:

- Pretreatment period: for a maximum of 28 days before baseline, including screening, washout (if applicable) and baseline
- Efficacy treatment period: beginning the day after baseline and continuing to visit 8/week 24
- Long-term safety period: beginning after visit 8/week 24 and continuing to visit 10/week 52 (end of study [EOS]), or to the end of treatment (EOT).

#### 2.2.1.1 Pretreatment Period

After informed consent and visit 1/screening, subjects are grouped according to their current NDO therapy and/or other medication:

Group A: Subjects who are currently not receiving any prohibited medication including
any oral drug treatment to manage their NDO, or when botulinum toxin is no
longer considered effective.

Group B: Subjects who currently are receiving oral drug treatment to manage their NDO
or receive any other prohibited medication.

After the screening visit, a 2-day weekend e-diary has to be completed by the subjects to get acquainted with the e-diary and the home assessments:

- Group A: Following successful completion of the first 2-day weekend e-diary, confirmed at visit 2, the subjects will start to complete the 7-day baseline e-diary followed by the baseline visit (visit 3).
- Group B: Following successful completion of the first 2-day weekend e-diary, confirmed at visit 2, the subjects will start their 2-week washout period. In the second week of their washout period, they will complete the 7-day baseline e-diary followed by the baseline visit (visit 3).

If a subject is suffering from a symptomatic UTI at visit 1/screening or is diagnosed with one between visit 1/screening and visit 3/baseline, the UTI should be treated successfully (clinical recovery) prior to baseline. If a symptomatic UTI is present at or just before visit 3/baseline, all baseline assessments should be postponed with a maximum of 7 days until the UTI is successfully treated (clinical recovery). The 7-day baseline e-diary does not have to be repeated if at least the 2-day weekend e-diary and 1 day of the weekday e-diary were completed while the subject did not suffer from a symptomatic UTI.

Subjects will enter the efficacy treatment period if they meet the eligibility criteria and satisfactorily complete the pretreatment period (ability to complete bladder diary, catheterized volumes and questionnaires).

In case the subject or the subject's parent(s)/caregiver(s) are not able or willing to perform the SMIP, the measuring device is not available at the site, or there is a technical problem, the SMIP may be omitted.

#### 2.2.1.2 Efficacy Treatment Period

Study drug administration will begin on the day after the baseline visit (i.e., on day 1). The initial dose of mirabegron is predicted to achieve plasma concentrations equivalent to the steady state exposures expected with 25 mg mirabegron administered once daily in adults (PED25).

At visit 4/week 2, visit 5/week 4 or visit 6/week 8, subjects must be up-titrated to the pediatric equivalent dose of 50 mg in adults (PED50), based on the given dose titration criteria [see Section 5.1.2].

At visit 8/week 24, the primary efficacy endpoint will assessed, which is the change from baseline in MCC.

If a subject is suffering from a symptomatic UTI in the week prior to any (un)scheduled urodynamic investigation (e.g., visit 5/week 4, visit 8/week 24), the UTI should be treated successfully first (clinical recovery). To allow for treatment of the UTI, these visits may be postponed with an additional maximum of 7 days on top of the already existing visit window.

The 7-day e-diary does not have to be repeated if at least the 2-day weekend e-diary and 1 day of the weekday e-diary were completed while the subject did not suffer from a symptomatic UTI.

If a subject suffers from a symptomatic UTI in the week prior to any other study visit, these visits do not need to be postponed and the 7-day e-diary does not have to be repeated.

#### 2.2.1.3 Long-term Safety Period

For long-term safety evaluation, following visit 8/week 24, subjects will stay on their individual dose level until visit 10/week 52 (EOT/EOS).

#### 2.2.2 Dose Rationale

The target exposures of 69 and 188 ng·h/mL for pediatric equivalent dose 25 mg (PED25) and pediatric equivalent dose 50 mg (PED50) were derived from the adult phase 3 program and are the mean steady state AUC<sub>tau</sub> values following 25 and 50 mg prolonged-release tablets once daily in adults.

A population pharmacokinetic model was used to predict the PED for subjects in the 178-CL-206A study. In brief, this popPK model was developed on adult phase 3 data, and allometric (weight-based) scaling was added to all clearance and volume terms to allow for scaling of the pharmacokinetics to pediatric subjects. The model was validated on pediatric data in Study 178-CL-202 (single ascending-dose study) and was shown to appropriately predict the pharmacokinetics of mirabegron in pediatric subjects.

Simulations were then performed to determine a body weight at which subjects would have steady state exposures comparable to those in adults when dosed with 25 or 50 mg daily; this weight was determined to be  $\geq$  35 kg. Based on prior experience obtained in an ongoing Astellas study in another program in patients with NDO (Study 905-CL-047; IND 58135), the average age at which children reach a body weight of 35 kg is approximately 11 years. The dosing recommendation based on this modeling is in line with the literature [Momper et al, 2013] in which a meta-analysis of compounds submitted to the FDA with a similar indication in adults and adolescents showed that in almost all cases, the adolescents required the same dose as the adults.

Therefore, subjects with a body weight of  $\geq$  35 kg can be dosed with mirabegron tablets. Subjects with a body weight < 35 kg cannot be dosed with the 25 and 50 mg tablets because that would result in higher than target exposures. Subjects with a body weight < 35 kg will therefore be dosed with mirabegron oral suspension.

Mirabegron oral suspension (8 mg/mL) has been developed for use in the pediatric population. The population pharmacokinetic model referred to above includes a formulation factor to account for the different (lower) relative bioavailability of the oral suspension compared to the tablet. This factor has been used in simulations to predict the suspension doses and weight categories that would have a reasonable variance around the target exposures.

EudraCT number 2015-002876-25


For dosing with oral suspension, the weight range to be covered is from 11 kg (the approximate body weight of a 3-year-old child, according to the NHANES database [McDowell et al, 2008]) to 35 kg (above which pediatric subjects could be dosed with the tablet formulation). Subjects with a body weight < 11 kg will not be included in the study. Suspension dosing for body weights  $\geq$  35 kg was also determined for cases in which a pediatric subject in that weight category does not want or would be unable to swallow a tablet. The simulation resulted in the 3 body weight categories that can be found in the dosing schedule (see [Section 5.1.1]).

## 2.3 Endpoints

## 2.3.1 Primary Efficacy Endpoint

The primary efficacy endpoint will be the change from baseline in MCC after 24 weeks of treatment (based on filling urodynamics).

#### 2.3.2 Secondary Efficacy Endpoints

#### 2.3.2.1 Urodynamic Measures

Secondary efficacy endpoints will include the change from baseline in the following urodynamic measures:

- MCC at visit 5/week 4
- Bladder compliance  $(\Delta V/\Delta P)$  at visit 5/week 4 and visit 8/week 24
- Number of overactive detrusor contractions (> 15 cm H<sub>2</sub>0) until end of filling at visit 5/week 4 and visit 8/week 24
- Detrusor pressure at end of filling at visit 5/week 4 and visit 8/week 24
- Filling volume until first overactive detrusor contraction (> 15 cm H<sub>2</sub>0) at visit 5/week 4 and visit 8/week 24

#### 2.3.2.2 Bladder Volume and Leakage Measures

The following endpoints will be obtained from the e-diary and be analyzed as the change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS).

- Average catheterized volume per catheterization
- Maximum catheterized volume
- Maximum catheterized daytime volume
- Average morning catheterized volume (based on first catheterization after subject woke up)
- Mean number of leakage episodes per day (day and night time)
- Number of dry (leakage-free) days/7 days (day and night time)

For this study the first morning catheterization after waking up is regarded as part of the 'night', whilst the last evening catheterization before sleep time is part of the 'day'.

EudraCT number 2015-002876-25


The collected urine volume will be weighed by the subject or subject's parent(s)/caregiver(s) and the results will be entered in the e-diary. The conversion factor used for weight-to-volume is 1g = 1 mL.

## 2.3.2.3 Patient- or Clinician-reported Questionnaire Endpoints

The following endpoints will be obtained from patient- or clinician-reported questionnaires.

- Change from baseline at visit 8/week 24 and visit 10/week 52 (EOT/EOS) in PIN-Q
- Change from baseline at visit 8/week 24 and visit 10/week 52 (EOT/EOS) in PGI-S
- Clinician Global Impression of Change (CGI-C) at visit 8/week 24 and visit 10/week 52 (EOT/EOS)
- Acceptability at visit 5/week 4, visit 8/week 24 and visit 10/week 52 (EOT/EOS)

#### 2.3.3 Safety Endpoints

The following safety endpoints will be assessed:

- Incidence and severity of TEAEs
- Change from baseline in vital signs (clinic measurements): systolic blood pressure, diastolic blood pressure, pulse rate and temperature at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS)
- Change from baseline in vital signs (self blood pressure measurement [SBPM]): systolic blood pressure, diastolic blood pressure, pulse rate at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) and on 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50 (visit 4/week 2, visit 5/week 4 or visit 6/week 8), if not already covered by the scheduled visit 4/week 2 and/or visit 5/week 4 SBPM.
- Change from baseline in hematology and biochemistry tests at visit 7/week 12 and visit 10/week 52 (EOT/EOS) and urinalysis tests at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS)
- Change from baseline in ECG parameters at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS)
- Change from baseline to visit 10/week 52 (EOT/EOS) in upper urinary tract ultrasound assessment
- Change from baseline in eGFR at visit 7/week 12 and visit 10/week 52 (EOT/EOS)

#### 2.3.4 Pharmacokinetics

The following pharmacokinetic parameters will be determined for each individual:

• C<sub>max</sub>, t<sub>max</sub>, AUC<sub>24</sub>, C<sub>trough</sub>, CL/F and V<sub>z</sub>/F

Additional pharmacokinetic parameters may be calculated based on the model used.

**Sponsor: APEB**EudraCT number 2015-002876-25


#### 2.3.5 Exploratory Endpoints

## 2.3.5.1 Exploratory Efficacy Endpoints

The following efficacy endpoints will be examined:

- Change from baseline at visit 5/week 4 and visit 8/week 24 in filling volume at 20 cm, 30 cm and at 40 cm H<sub>2</sub>O detrusor pressure, given that those pressures are reached during the examination
- Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/ week 52 (EOT/EOS), as determined from the e-diary entries in:
  - Mean grade of leakage
  - o Total catheterized volume per day
  - o Change from baseline in SMIP-derived bladder compliance
  - o Number of CICs/day
  - Responder in respect to leakage (complete, partial, no response)

#### 2.3.5.2 Exploratory Safety Endpoints

- Change from baseline in intravesical pressure (SMIP) at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS)
- Change from baseline in body height and weight at visit 8/week 24 and visit 10/week 52 (EOT/EOS)

#### 3 STUDY POPULATION

## 3.1 Selection of Study Population

The study population will be male and female child and adolescent subjects aged 3 to less than 18 years of age with NDO on CIC. The age of the subjects at the date of signing the informed consent or assent form at visit 1/screening will determine the age of the subject for inclusion into the study.

Re-screening is not allowed.

#### 3.2 Inclusion Criteria

Subject is eligible for the study if all of the following apply:

- 1. Independent Ethics Committee (IEC)/Institutional Review Board (IRB)-approved written Informed Consent and privacy language as per national regulations must be obtained from the subject and/or from the subject's parent(s) or legal guardian(s) prior to any study-related procedures (including discontinuation of prohibited medication, if applicable); assent by the subject is given as required by local law.
- 2. Subject is male or female from 3 to less than 18 years of age.
- 3. Subject has a body weight of  $\geq 11$  kg.

02 Nov 2016 Astellas 

- **4.** Subject suffers from NDO confirmed by urodynamic investigation at baseline. The diagnosis of NDO must be confirmed by the presence of at least 1 involuntary detrusor contraction > 15 cm H<sub>2</sub>O from baseline detrusor pressure, and/or a decrease in compliance leading to an increase in baseline detrusor pressure of > 20 cm H<sub>2</sub>O.
- 5. Subject has been using CIC for at least 4 weeks prior to visit 1/screening.
- **6.** Subject has a current indication for drug therapy to manage NDO.
- 7. Subject is able to take the study drug in accordance with the protocol.
- **8.** Female subject must either:
  - Be of nonchildbearing potential:
    - o Clearly premenarchal or in the judgment of the investigator is premenarchal,
    - o Documented surgically sterile,
  - Or, if of childbearing potential:
    - Agree not to try to become pregnant during the study and for 28 days after the final study drug administration,
    - o And have a negative pregnancy test at visit 1/screening and at baseline,
    - And, if sexually active must agree to use a highly effective method of birth control, which includes established use of oral, injected or implanted hormonal methods of contraception, OR placement of an intrauterine device (IUD) or intrauterine system (IUS). Birth control must be practiced from visit 1/screening and continuing throughout the study period, and for 28 days after the final study drug administration.
- 9. Male subject and their female spouse/partner who are of childbearing potential must be using a highly effective method of birth control, which includes established use of oral, injected or implanted hormonal methods of contraception, placement of an IUD or IUS. Birth control must be practiced from visit 1/screening and continuing throughout the study period, and for 28 days after the final study drug administration.
- **10.** Female subject must not be breastfeeding from visit 1/screening until 28 days after last study drug administration.
- 11. Subject and subject's parent(s)/legal guardian(s) agree that the subject will not participate in another interventional study while participating in the study.
- **12.** Subject and subject's parent(s)/legal guardian(s) are willing and able to comply with the study requirements and with the concomitant medication restrictions.

Waivers to the inclusion criteria will NOT be allowed.

#### 3.3 Exclusion Criteria

Subject will be excluded from participation if any of the following apply:

- 1. Subject has a known genitourinary condition (other than NDO) that may cause overactive contractions or incontinence (e.g., bladder extrophy, urinary tract obstruction, urethral diverticulum or fistula) or kidney/bladder stones or another persistent local pathology that may cause urinary symptoms.
- 2. Subject has one of the following gastrointestinal problems: partial or complete obstruction, decreased motility such as paralytic ileus, subjects at risk of gastric retention.
- 3. Subject has a urinary indwelling catheter within 4 weeks prior to visit 1/screening
- 4. Subject has a surgically treated underactive urethral sphincter
- **5.** Subject has vesico-ureteral reflux grade 3 to 5.
- **6.** Subject has undergone bladder augmentation surgery.
- 7. Subject receives electrostimulation therapy, if started within 30 days before visit 1/screening or is expected to start during the study period. Subjects who are on an established regimen may remain on this for the duration of the study.
- **8.** Subject suffers from a symptomatic UTI at baseline (symptomatic is defined as pain, fever, hematuria, new onset foul-smelling urine). If present at visit 1/screening or diagnosed between visit 1/screening and visit 3/baseline, the UTI should be treated successfully (clinical recovery) prior to baseline. If a symptomatic UTI is present at baseline, all baseline assessments should be postponed for a maximum of 7 days until the UTI is successfully treated (clinical recovery).
- 9. Subject has a (mean) resting pulse rate > 99<sup>th</sup> percentile [Fleming et al, 2011].
- **10.** Subject has an established hypertension and a systolic or diastolic blood pressure greater than the 99th percentile of the normal range determined by sex, age and height, plus 5 mmHg [NIH 2005].
- **11.** Subject has a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS]; or family history of LQTS, exercise-induced syncope).
- **12.** Subject has severe renal impairment (eGFR according to Larsson equation < 30 mL/min).
- **13.** Subject's AST or ALT is greater than or equal to 2 times the upper limit of normal (ULN) or total bilirubin (TBL) greater than or equal to 1.5 times the ULN according to age and sex.
- **14.** Subject has a history or presence of any malignancy prior to visit 1/screening.
- **15.** Subject has known or suspected hypersensitivity to mirabegron, any of the excipients used in the current formulations or previous severe hypersensitivity to any drug.

**Sponsor: APEB**EudraCT number 2015-002876-25


- **16.** Subject has participated in another clinical trial (and/or has taken an investigational drug) within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1/screening.
- 17. Subject uses any of the following prohibited medications (after start of washout):
  - Any medication, other than the study drug used, for the management of NDO;
  - Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index or sensitive P-glycoprotein (P-gp) substrates
  - Any strong CYP3A4 inhibitors if the subject has a mild to moderate renal impairment (eGFR 30 – 89 mL/min).
- **18.** Subject has been administered intravesical botulinum toxin; except if given > 4 months prior to visit 1/screening and the subject experiences symptoms comparable to those existing prior to the botulinum toxin injections.
- **19.** Subject has any other condition, which in the opinion of the Investigator, precludes the subject's participation in the study.
- **20.** Subject's parent/legal guardian is an employee of the Astellas Group, the Contract Research Organization (CRO) involved, or the investigator site executing the study.

Waivers to the exclusion criteria will NOT be allowed.

For exclusion criterion 9 please refer to Appendix 12.9 and for exclusion criterion 10 please refer to Appendix 12.10 Appendix 12.11 Appendix 12.12 and Appendix 12.13

#### 4 TREATMENTS

## 4.1 Identification of Investigational Products

#### 4.1.1 Test Drug

Mirabegron prolonged-release (or extended-release) tablets were approved in Japan in 2011, and to date have been approved in more than 65 countries worldwide; trade names include Betanis®, Betmiga® and Myrbetriq®. The approved indication is the treatment of OAB with symptoms of urge urinary incontinence, urgency and urinary frequency in adults.

Mirabegron oral suspension has been developed as an appropriate formulation for weight based dosing in smaller children.

For detailed information on mirabegron prolonged-release tablets and mirabegron granules for oral suspension, please refer to the applicable Investigational Medicinal Product Dossier (IMPD).

Mirabegron tablets are supplied as prolonged-release tablets containing 25 mg or 50 mg of active ingredient.

For the oral suspension, mirabegron prolonged-release granules are supplied and will be reconstituted with water to prepare an oral suspension of 8 mg/mL. Detailed information on the preparation of the mirabegron oral suspension will be provided to the subject and

02 Nov 2016 Astellas 

EudraCT number 2015-002876-25


subject's parent(s)/caregiver(s) in local language. Due to shelf-life limitations, an additional dispensing visit is foreseen at visit 9/week 36 for subjects receiving mirabegron oral suspension. This dispensing visit does not need to be accompanied by the subject.

## 4.1.2 Comparative Drug(s)

Not applicable.

## 4.2 Packaging and Labeling

All study drugs used in this study will be prepared, packaged, and labeled under the responsibility of qualified staff at Astellas Pharma Europe B.V. (APEB) or Sponsor's designee in accordance with APEB or Sponsor's designee Standard Operating Procedures (SOPs), Good Manufacturing Practice (GMP) guidelines, International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines, and applicable local laws/regulations.

Each study drug package will bear a label conforming to regulatory guidelines, GMP and local laws and regulations that identifies the contents as an investigational drug.

A qualified person of APEB or Sponsor's designee will perform the final release of the study drugs according to Directive 2003/94/EC annex 13.

## 4.3 Study Drug Handling

Current ICH GCP Guidelines require the investigator to ensure that study drug deliveries from the Sponsor are received by the investigator/or designee and

- That such deliveries are recorded.
- That study drug is handled and stored according to labeled storage conditions,
- That study drug is with appropriate expiry/retest and is only dispensed to study subjects in accordance with the protocol, and
- That any unused study drug is returned to the Sponsor.

Drug inventory and accountability records for the study drugs will be kept by the investigator/ or designee. Study drug accountability throughout the study must be documented and reconciled. The following guidelines are therefore pertinent:

- The investigator agrees not to supply study drugs to any persons except the subject or subject's parent(s)/caregiver(s) of the eligible subjects in this study in accordance with the protocol.
- The investigator or designee will keep the study drugs in a pharmacy or other locked and secure storage facility under controlled storage conditions, accessible only to those authorized by the investigator to dispense these test drugs.
- A study drug inventory will be maintained by the investigator or designee. The inventory
  will include details of material received and a clear record of when they were dispensed
  and to which subject.

**Sponsor: APEB**EudraCT number 2015-002876-25


At the conclusion or termination of this study, the investigator or designee agrees to
conduct a final drug supply inventory and to record the results of this inventory on the
drug accountability record. It must be possible to reconcile delivery records with those of
used and/or returned study drugs. Any discrepancies must be accounted for and
documented. Appropriate forms of deliveries and returns must be signed by the site staff
delegated this responsibility.

 The site must return study drug to the Sponsor or designee at the end of the study or upon expiration. If due to institutional policy or local law, used drug cannot be returned to the Sponsor or designee the drug may be destroyed according to local law.

## 4.4 Blinding

This section is not applicable as this is an open-label study.

## 4.5 Assignment and Allocation

All subjects will receive active mirabegron treatment (open-label).

Subject number assignment will be coordinated centrally by using an interactive response system.

## 4.5.1 Subject Numbering

Subjects will be assigned a subject number at study entry. The full subject number will consist of 10 digits; 5 for the site number (provided by the Sponsor) and 5 for the consecutive subject number.

## 4.5.2 Subject Replacement

An enrolled subject who withdraws or discontinues before dosing will be considered a screening failure and will be replaced. If a subject discontinues treatment after dosing, this subject will be replaced at the discretion of the Sponsor.

#### 5 TREATMENTS AND EVALUATION

## 5.1 Dosing and Administration of Study Drug

## 5.1.1 Dose/Dose Regimen and Administration Period

The initial dose will be PED25 [Section 2.2.2]. The dose must be up-titrated to PED50 according to the titration criteria. Study drug will be taken orally, once a day in the morning around the same time of day and around time of food intake (i.e., within 1 hour before or after breakfast).

On visit days where a pharmacokinetic sample is planned in the clinic, completion of breakfast and study drug dosing should occur in the clinic and dosing will be done under supervision of the investigator.

Mirabegron tablets will be taken with a sip of water. The tablet should be taken as a whole and should not be chewed, divided or crushed.

02 Nov 2016 Astellas 

EudraCT number 2015-002876-25


Mirabegron prolonged-release granules will be reconstituted with water to prepare a mirabegron oral suspension of 8 mg/mL. Administration will be via an oral syringe with a sip of water afterwards. Detailed information on the preparation of the suspension will be provided to the subject and subject's parent(s)/caregiver(s) in local language. For subjects receiving mirabegron oral suspension, an additional (optional) dispensing visit is scheduled at visit 9/week 36.

#### Selection of the formulation:

Subjects with a body weight < 35 kg: mirabegron oral suspension.

Subjects with a body weight  $\geq$  35 kg: mirabegron tablets.

#### Selection of the dose:

Doses are calculated weight-based. The bodyweight at visit 3/baseline determines the weight range for the starting dose (PED25) and the up-titration dose (PED50) to be used Table 4.

Table 4 Weight-based Doses for Tablets or Suspension

| | Weight Range | Suspension Volume † | <b>Tablet Dose</b> |
|-------|--------------|---------------------|--------------------|
| PED25 | 11 - < 22 kg | 3 mL | - |
| | 22 - < 35 kg | 4 mL | - |
| | ≥ 35 kg | 6 mL | 25 mg |
| PED50 | 11 - < 22 kg | 6 mL | - |
| | 22 - < 35 kg | 8 mL | - |
| | ≥ 35 kg | 11 mL | 50 mg |

PED25: Pediatric equivalent dose 25 mg; PED50: Pediatric equivalent dose 50 mg

#### Further dosing information:

- For subjects with a body weight  $\geq$  35 kg who do not want to or are unable to take tablets, the oral suspension can be supplied.
- At visit 8/week 24 subjects on mirabegron oral suspension may switch to tablets if the body weight turns to be ≥ 35 kg.
- Subjects receiving mirabegron tablets can switch to mirabegron oral suspension (and vice versa) for acceptability reasons after Sponsor's prior approval and on a case-by-case basis.

#### 5.1.2 Increase or Reduction in Dose of the Study Drug(s)

The aim is to obtain a safe low pressure bladder, to inhibit overactive detrusor contractions and to reach continence. Subject discontinuation rules apply (see [Section 6.1]).

Dose up-titration to PED50 must be performed at visit 4/week 2, visit 5/week 4 or visit 6/week 8, unless:

- 1. The investigator considers the subject to be effectively treated with PED25, based on urodynamics and the e-diary;
- 2. There are safety or tolerability issues with PED25.

<sup>†</sup> Suspension strength: 8 mg/mL

EudraCT number 2015-002876-25


Dose down-titration to PED25 can be performed at any time if there is a safety issue.

If an insufficient control of the NDO is observed at the highest tolerated mirabegron dose due to insufficient effect (based on, for example, ultrasound showing upper tract dilation; the appearance of a high grade reflux; high intravesical pressures; high detrusor pressures or high amplitude overactive contractions), the investigator should reconsider the subject's further participation in the study and consider an alternative treatment.

# 5.1.3 Previous and Concomitant Treatment (Medication and Nonmedication Therapy)

Please refer to [Appendix 12.1] for drug classes or specific medications that are prohibited during participation in the study.

#### **5.1.4** Treatment Compliance

The investigator or designee should instruct the subject and/or subject's parent(s)/caregiver(s) to meet 100% compliance with study drug intake throughout the entire study period. If compliance is around 80% or 120%, the investigator or designee is to counsel the subject and/or subject's parent(s)/caregiver(s) and ensure steps are taken to improve compliance.

Compliance of the study drug taken outside the clinic will be monitored at each subsequent visit at the clinic by the accounting of used and unused study drugs returned by the subject.

Subjects and their parent(s)/caregiver(s) will be clearly instructed to return all study drugs to the clinic at each clinic visit. This includes empty study drug containers.

## 5.1.5 Restrictions for Foods and Drinks During the Study

Restrictions for foods and drinks are not applicable. On visit days where a pharmacokinetic sample is planned in the clinic, completion of breakfast and study drug dosing should occur in the clinic.

## 5.2 Demographics and Baseline Characteristics

#### 5.2.1 Demographics

Demographics and baseline characteristics will be collected at visit 1/screening. Demographics will include date of birth (or year depending on the country), age, sex and race/ethnicity.

Measurements for height and weight will be taken at visit 1/screening, visit 3/baseline, visit 8/week 24 and at visit 10/week 52 (EOT/EOS).

#### **5.2.2** Medical History

A complete medical history including a detailed NDO history will be collected at visit 1/screening. All relevant past and present conditions, as well as prior surgical procedures will be recorded for the main body systems.

#### 5.2.3 Diagnosis of the Target Disease, Severity, and Duration of Disease

A detailed NDO history for each subject will be collected at visit 1/screening. This history includes the date of start of symptoms, underlying condition, comorbidities associated with NDO and treatment history for NDO.

## 5.3 Efficacy and Pharmacokinetics Assessment

#### **5.3.1** Urodynamic Assessments

Urodynamic assessments will be performed at visit 3/baseline, and at visit 5/week 4, visit 8/week 24.

Additional urodynamic assessments can be performed at e.g. visit 10/week 52 (EOT/EOS), or at any other time point when deemed necessary by the investigator.

Computerized urodynamic equipment should be used to allow central analysis. A manual with detailed SOPs will be provided to the investigators to ensure standardization of the procedure. On-site assessment and evaluation of the urodynamic assessments are to be conducted by a medically qualified & trained person.

Every effort should be taken to ensure that the rectum is free of stool. The evening before the urodynamic investigation, bowel preparation should be performed with the existing bowel regimen or when a subject is not an a bowel management program a suppository or enema should be applied to cleanse the rectum and increase accuracy of rectal pressure recordings [Bauer et al, 2015]. If digital evacuation of stool is required for the subject, this should be performed prior to the procedure.

The subject is placed in a stable position. The position should be the same for all procedures throughout the study. The bladder is then filled with room-warm saline via a pump with a filling rate of 10% of the mean of the catheterized volumes collected in the bladder diary prior to baseline. All urodynamic investigations in each subject should be done at the same filling rate for all visits. If the filling rate was accidentally too high or too low at the baseline visit, that same filling rate should be used throughout the study for this individual subject. Minor deviations in the filling rate (no more than 1 or 2 mL/min) caused by inaccuracy of the pump are accepted.

The following parameters will be determined:

- MCC at end of filling
- Bladder compliance
- Filling volume until first detrusor contraction (> 15 cm H<sub>2</sub>O)
- Filling volume at 20 cm, 30 cm and 40 cm H<sub>2</sub>O detrusor pressure (if reached)
- Number of overactive detrusor contractions (> 15 cm H<sub>2</sub>O) until end of filling
- Detrusor pressure at end of filling

Filling will be stopped (end of filling) when:

- Major leakage occurs (the rate of leakage exceeds the rate of infusion)
- 135% of maximum catheterized volume has been reached
- The subject experiences pain or discomfort at filling which does not resolve after temporary stop of filling
- The detrusor pressure exceeds 100 cm H<sub>2</sub>0 or is considered dangerously high by the investigator or urodynamicist (for instance a prolonged passive detrusor pressure > 40 cm H<sub>2</sub>O).

The results of the urodynamic assessments, including the position of the subject during the assessments will be entered in the eCRF.

#### 5.3.2 Bladder Diary

The bladder diary is part of the subject's e-diary. After a successful visit 1/screening, all subjects start with the completion of a 2-day weekend e-diary visit to get acquainted with the e-diary and the assessments. Completion of this diary should start in the weekend prior to visit 2.

The e-diary data is reviewed by the investigator prior to the start of visit 2 and discussed and confirmed with the subject or the subject's parent(s)/caregiver(s) during the (telephone) visit. If the investigator is under the impression that the subject and/or the subject's parent(s)/caregiver(s) can perform all the required assessments and are able to complete all required forms with credible data, completion is considered successful.

If this is not the case, the investigator should counsel/re-train the subject or the subject's parent(s)/caregiver(s) prior to the start of the 7-day baseline e-diary. In case the subject and/or the subject's parent(s)/caregiver(s) are still not able to complete the 7-day baseline e-diary satisfactorily, the subject should be excluded from further participation in the study.

If successful completion of the 2-day weekend e-diary is confirmed at visit 2:

- Subjects from group A start with collection of the 7-day baseline e-diary, followed by visit 3/baseline.
- Subjects in group B start with a 14-day washout. In the second week of the washout period collection of their 7-day baseline e-diary starts, followed by visit 3/baseline.

Subsequent bladder diaries will be completed by the subject or the subject's parent(s)/caregiver(s) in the week prior to visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS). Completion of 7-day bladder diaries should start approximately 7 days prior to the indicated visit (or telephone contact).

The following information will be collected in the bladder diary.

Daily during the 7-day period:

- Time of CICs
- Presence of leakage between CICs
- Sleep time and wake-up time

**Sponsor: APEB** EudraCT number 2015-002876-25


On 2 consecutive weekend days within the 7-day period:

- Catheterized volume
- Grade of leakage between CICs
- Weight of diaper/pad (visit 3/baseline and visit 8/week 24)
- SMIP [Section 5.4.6]

The Investigator must guide the subject and subject's parent(s)/caregiver(s) to ensure that on the evening before and during the two weekend days of collection of catheterized volume and SMIP, the subject's fluid intake should be regulated to an appropriate level taking e.g. age, sex and subject's condition into account. The intake must remain as consistent as possible on these volume collecting days throughout the entire study. Detailed on-site training of the bladder diary and a booklet with operating instructions in local language will be provided to the subject and subject's parent(s)/caregiver(s).

To ensure consistency in collection of the data and subject's routine, assessments must be performed over the weekend and by the same person. As an exception, it is possible to perform the weekend assessments on 2 other days in the collection week (e.g., during a holiday period) if the subject can maintain his/her standard weekend routine for catheterizations and fluid intake.

Results will be directly entered by the subject or subject's parent(s)/caregiver(s) in the e-diary [Section 8.1.1].

#### 5.3.3 Questionnaires

Questionnaires will be completed as described below.

The following questionnaires will be used:

- The PIN-Q [Appendix 12.4] will be completed on one weekend day preceding visit 3/baseline, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The PGI-S [Appendix 12.5] will be completed on one weekend day preceding visit 3/baseline, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The Acceptability Questionnaire [Appendix 12.6] will be completed on one weekend day preceding at visit 5/week 4, visit 8/week 24 and visit 10/week 52 (EOT/EOS). For each formulation a separate questionnaire is available [Appendix 12.6] and Appendix 12.7].
- The CGI-C [Appendix 12.8] will be completed at visit 8/week 24 and at visit 10/week 52 (EOT/EOS).

The PIN-Q was chosen as the most appropriate cross-cultural pediatric quality of life measurement tool in this population. A Likert scale adopted for 20 measures is used [Bower et al, 2006].

Questionnaires to be completed by the subject or the subject's parent(s)/caregiver(s) (i.e., PIN-Q, PGI-S and the Acceptability Questionnaire) will be available in the local language and provided via the e-diary. Results will be directly entered in the e-diary by the subject or subject's parent(s)/caregiver(s) [Section 8.1.1].

**Sponsor: APEB** EudraCT number 2015-002876-25


The CGI-C will completed by the investigator and the results will be entered in the eCRF. Clinically relevant adverse changes will be recorded as an AE [Section 5.5.1].

#### 5.3.4 Pharmacokinetics

Samples of venous blood for pharmacokinetic assessments will be taken when the subject has reached steady state at the optimal dose (considered to be reached after 10 days of daily dosing). A total of 4 pharmacokinetic samples will be collected, divided over 2 sampling days. These 2 days can be selected from any of the options given in the schedule of assessments (i.e., on visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36, or visit 10/week 52) and do not have to be in a specific (consecutive) order:

- Sampling day 1: 1 trough sample (i.e., predose sample).
- Sampling day 2: 1 trough and 2 postdose samples taken between 2h and 5h postdose, with at least 1 hour in between the samples.

To allow for an early assessment of the dose-response relationship by the DSMB, it is preferred the pharmacokinetic sampling takes place as early in the study as possible.

On visit days where a pharmacokinetic sample is planned in the clinic, completion of breakfast and study drug dosing should occur in the clinic. Dosing on a sampling day with postdose samples must occur within 1 hour after completion of breakfast.

In case there is a dose change within 10 days prior to a planned pharmacokinetic sampling visit, the subject is not considered to be at steady state, and samples should be postponed to another visit as per the schedule of assessments.

Trough samples must be taken within 1 hour prior to dosing. Dosing time on the sampling day and dosing time of the previous day will be collected in the eCRF/e-diary respectively. Postdose samples must be taken between 2h and 5h postdose, with at least 1 hour in between the samples. In addition to the dosing time, the time of completion of breakfast, and type of breakfast will be collected in the eCRF on this sampling day.

A topical anesthetic cream or plaster must be offered at the point of venipuncture to minimize distress of the subject. For sampling, the arm opposite to the arm used for blood pressure measurements should be used (i.e. preferably the left arm). Blood sampling should occur after vital signs and ECG measurements.

Operational aspects of sample collection, storage and shipment of frozen samples are described in the protocol [Section 5.6] and in the laboratory manual.

EudraCT number 2015-002876-25


### 5.4 Safety Assessments

## 5.4.1 Vital Signs

#### **5.4.1.1** Clinic Measurement of Vital Signs

Triplicate blood pressure and pulse measurements and single body temperature measurements (ear thermometer) will be performed at visit 1/screening, visit 3/baseline, and on visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS). Clinic measurements of vital signs at visit 1/screening and visit 3/baseline will be used to assess eligibility.

The preferred method of measurement is via the auscultatory technique. If this method is not available at the site, measurements will be per standard clinic practices. The method for measuring vital signs should be consistent for all visits. For each subject the correct size of the blood pressure cuff must be determined and used when assessing blood pressures. Blood pressure and pulse will be measured with approximately 2-minute intervals, after the subject has been calm and without distress for at least 5 minutes.

The subject should be seated with the back supported, feet on the floor and right arm supported, legs uncrossed and the cubital fossa at heart level. If sitting is not possible, supine is allowed, but measurements should always be taken in the same position. The subject should not move and should remain silent during the reading, as moving and talking can affect the reading.

The right arm is preferred in repeated measures of blood pressure for consistency and comparison to standard tables. The same arm should be used throughout the study whenever possible. Vital sign measurements should be performed prior to blood sampling.

The method of body temperature measurement is via an ear thermometer and should be consistent for all visits.

Clinically relevant adverse changes in vital signs will be recorded as an AE [Section 5.5.1].

#### 5.4.1.2 Self-measurement of Vital Signs

Triplicate SBPM (blood pressure and pulse rate) will be performed on the 2 weekend days prior to each visit. Additional SBPM is done on 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50 (visit 4/week 2, visit 5/week 4 or visit 6/week 8), if not already covered by the scheduled visit 4/week 2 and/or visit 5/week 4 SBPM.

Following successful completion [see Section 5.3.2] of the first 2-day weekend e-diary, confirmed at visit 2, subsequent measurements will be performed in the weekend preceding visit 3/baseline, visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS).

Devices for measuring blood pressure and pulse rate will be provided to subjects for home measurements. Detailed on-site training to use the SBPM device and a booklet with operating instructions in local language will be provided to the subject and the subject's parent(s)/caregiver(s).

EudraCT number 2015-002876-25


For each subject the correct cuff size will be determined by the investigator by measuring the circumference of the subject's upper arm in order to give the subject the device with the best cuff type. Ideally, the bladder length of the cuff should be 80% to 100% of the arm's circumference and the width of the bladder approximately 40% (the bladder is the inflatable part of the cuff). The cuff should be put on according to the instructions given by investigator.

Morning measurements should be taken after waking up, before breakfast and before study drug intake, evening measurements should be taken prior to bedtime. If deemed necessary by the Investigator, subjects may be asked to perform additional measurements.

Self-measurements should, where possible, be performed in the same position as the clinic measurements for vital signs.

Results will be directly entered by the subject or subject's parent(s)/caregiver(s) in the e-diary [Section 8.1.1].

#### 5.4.2 Adverse Events

AEs will be collected from visit 1/screening until visit 10/week 52 (EOT/EOS). See [Section 5.5] for information regarding AE collection and data handling.

#### 5.4.2.1 Adverse Events of Possible Hepatic Origin

See [Appendix 12.2] for detailed information on monitoring and assessment of suspected liver abnormalities, if an AE for a subject enrolled in a study and receiving study drug is due to circulating liver enzymes (AST, ALT, ALP) or bilirubin, or if the AE is suspected to be due to hepatic dysfunction.

Subjects with AEs of hepatic origin accompanied by liver function test (LFT) abnormalities should be carefully monitored.

#### 5.4.3 Laboratory Assessments

Hematology and biochemistry assessments will be taken at visit 1/screening, visit 7/week 12 and visit 10/week 52 (EOT/EOS). In the event that an AE related to hematology/biochemistry parameters is found at visit 1/screening, an additional hematology/biochemistry assessment is to be taken at visit 3/baseline.

Urinalysis is to be assessed at visit 1/screening, at visit 3/baseline, and at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS).

To allow for an early DSMB safety assessment, the first 5-10 subjects who reach study visit 5/week 4 will have an additional blood draw at this visit [see Section 1.4].

A topical anesthetic cream or plaster must be offered at the point of venipuncture to minimize distress of the subject. For sampling the arm opposite to the arm used for blood pressure measurements should be used (i.e. preferably the left arm). Blood sampling should occur after vital signs and ECG measurements.

EudraCT number 2015-002876-25


All safety laboratory assessments will be performed at a central laboratory, except for urine pregnancy testing, which is done locally. Pregnancy test in female subjects of childbearing potential will be performed in serum (if blood is drawn for hematology/biochemistry) or urine (at the other visits).

Specimen collection and shipping procedures will be described in a laboratory manual. All laboratory results, including ULNs used in exclusion and discontinuation criteria, will be compared to age-appropriate norms. The investigator may decide to repeat the safety laboratory assessments, should the results be important for safety reasons and considered clinically relevant. Repeating safety laboratory assessments for re-screening is not allowed.

The clinical significance of out-of-range laboratory findings is to be determined and documented by the investigator/sub-investigator who is a qualified physician. Clinically significant adverse changes will be recorded as an AE [Section 5.5.1].

The laboratory parameters that will be assessed during the conduct of the study are listed in [Appendix 12.3].

#### 5.4.4 Physical Examination

Physical examinations will be performed at visit 1/screening and at visit 10/week 52 (EOT/EOS).

The physical examination will be performed per clinic standards and clinically significant findings at screening will be recorded as part of the subject's medical history. Clinically significant findings discovered after visit 1/screening will be recorded as an AE [Section 5.5.1].

#### 5.4.5 Electrocardiograms

Triplicate 12-lead ECG will be performed at visit 1/screening, visit 3/baseline, visit 5/week 4, visit 7/week 12, visit 8/week 24 and at visit 10/week 52 (EOT/EOS).

ECGs will be taken in the supine position (when possible, but always in the same position), after the subject has been lying quietly for at least 5 minutes. ECG machines will be provided to the site by a central laboratory to allow for central reading (ECG recordings will be performed according to ICH guidelines E14 [CPMP/ICH/2711/99] to make them readable and interpretable for potential later assessment by an independent cardiologist).

ECGs will be recorded with an interval of about 30 seconds to 5 minutes between each ECG. Recordings will be made at a speed of 25 mm/s and all leads have to include at least 4 complexes. This is according to the standard settings on the machines. The ECGs should be transmitted from the machine to the central laboratory (following the steps indicated in the user manual). In addition, 2 prints of the original ECG traces should be made on normal, nonheat sensitive paper. These should be clearly marked with the subject identification number (in such a way that they are anonymized), include date and time, and should be kept with the source documents.

**Sponsor: APEB** EudraCT number 2015-002876-25


The ECG machine will produce automatically calculated interval duration measurements for intervals of QT, QTcB, QTcF, etc., and an evaluation on the printed ECG. For a final safety assessment the manually read analysis reports of the central ECG readings (from cardiologists) will be made available to the investigators within 72 hours. The final ECG reports sent by the central laboratory must be reviewed by the investigator since there might be relevant differences from the initial analysis produced by the ECG machines.

For analysis the mean values of the triplicate readings will be used (not the highest or lowest value). In case of incomplete triplicates, mean values of the available ECG readings will be taken.

Please refer to [Section 6.1] for discontinuation criteria based on centrally read results from the QTcB mean from the visit 1 and visit 3 ECG triplicates (at least 2 ECGs of each triplicate reading must be available).

The ECG report itself will not be captured on the electronic case report from (eCRF), but will be captured in the central ECG laboratory database. Only the visit, ECG date and time, overall ECG interpretation and relevant comments will be captured in the eCRF. If specific concerns regarding the cardiac safety of a subject exist, a dual approach is recommended:

- On-site evaluation of the ECGs are to be conducted by a medically qualified person.
- In addition, the central ECG laboratory can be contacted (24 hours a day) to provide the final centrally read ECG analysis results within a shorter timeframe than the usual 72 hours (for contact details see the ECG Study Manual provided by the central ECG laboratory).

Any abnormalities must be evaluated in clinical context (based on subject's medical history and concomitant medication) and the investigator should determine if it is clinically significant. Clinically significant abnormalities should be reported as an AE [Section 5.5.1].

Detailed instructions and procedures for ECG recordings will be described in a separate manual.

#### 5.4.6 Self-measurement of Intravesical Pressure

SMIP will be performed as part of the bladder diary [Section 5.3.2]. In case the measuring device is not available/approved for use at the site, the subject or parent(s)/caregiver(s) are not able or willing to perform the SMIP, or there is a technical problem, the SMIP may be omitted.

Following successful completion of the first 2-day weekend e-diary, confirmed at visit 2, subsequent measurements will be performed in the weekend preceding visit 3/baseline, visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS).

SMIP is a method to measure the intravesical pressure at home. The pressure in the bladder can be measured by the subject or subject's parent(s)/caregiver(s) at the moment the subject catheterizes him/herself in the course of using CIC as a therapeutic intervention.

Measurements will be performed on a full and emptied bladder.

EudraCT number 2015-002876-25


The aim of this method is to verify that the intravesical pressure is in a safe range and particularly if the pressure at the time of CIC (the end-filling pressure), where intravesical pressure can be expected to be at its greatest, is at an acceptable level.

To start measurements, the SMIP device is connected to a CIC catheter with a 3-way stopcock via an air tube. By switching the handle on the stopcock, a closed circuit can be established between the SMIP device and the CIC catheter. The urine from the subject exerts pressure to the trapped air in the closed circuit and this pressure is transferred to a sensor in the SMIP device. The signal from the sensor is interpreted by a microprocessor which then displays the pressure numerically in centimeters  $H_2O$ . The zero is set to atmospheric pressure.

Once a stable read-out has been obtained, the handle on the stopcock can be switched again and the urine can now flow out of the catheter attached to the other outlet of the 3-way stopcock.

After the bladder has been emptied, the intravesical pressure is measured a second time by switching the handle of the stopcock again, establishing a closed circuit between the SMIP catheter and the SMIP device.

| Devices (Peritron+, | for measuring intravesical |
|---|---|
| pressure will be provided to subjects along with required auxiliar | ies such as special catheters |
| and connectors (Air Trap Tubing, | Detailed |
| on-site training of the SMIP and a booklet with operating instruct | tions in local language will |
| be provided to the subject and the subject's parent(s)/caregiver(s) | ). |

Results will be entered by the subject or subject's parent(s)/caregiver(s) in the e-diary [Section 8.1.1].

## 5.4.7 Estimated Glomerular Filtration Rate and Upper Urinary Tract Ultrasound

Renal function will be assessed via monitoring plasma creatinine and cystatin C levels at visit 1/screening, visit 7/week 12 and visit 10/week 52 (EOT/EOS).

The presence or absence of structural abnormalities of the urinary tract, upper tract dilation, vesicoureteral reflux, or obstruction at the ureterovesical or ureteropelvic junction will be assessed with an ultrasound of the upper urinary tract at visit 3/baseline, and at visit 10/week 52 (EOT/EOS).

For the first group of subjects (minimum of 5, maximum of 10) who reach study visit 5/week 4, the renal function will also be determined at visit 5/week 4 to allow for the early DSMB safety assessment.

Clinically significant abnormalities should be reported as an AE [Section 5.5.1].

Sponsor: APEB
EudraCT number 2015-002876-25


## 5.5 Adverse Events and Other Safety Aspects

#### **5.5.1** Definition of Adverse Events

An AE is defined as any untoward medical occurrence in a subject administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

Some countries may have additional local requirements for events that are required to be reported as AEs or in an expedited manner similar to a serious adverse event (SAE). In these cases, it is the investigator's responsibility to ensure these AEs or other reporting requirements are followed and the information is appropriately recorded in the eCRF accordingly.

An abnormality identified during a medical test (e.g., laboratory parameter, vital sign, ECG data, physical exam) should be defined as an AE only if the abnormality meets 1 of the following criteria:

- Induces clinical signs or symptoms
- Requires active intervention
- Requires interruption or discontinuation of study drug intake
- The abnormality or investigational value is clinically significant in the opinion of the investigator.

#### **5.5.2** Definition of Serious Adverse Events

An AE is considered "serious" if, in the view of either the investigator or Sponsor, it results in any of the following outcomes:

- Results in death
- Is life-threatening (an AE is considered "life-threatening" if, in the view of either the investigator or Sponsor, its occurrence places the subject at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death)
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly, or birth defect
- Requires inpatient hospitalization or leads to prolongation of hospitalization (hospitalization for treatment/observation/examination caused by AE is to be considered as serious)
- Other medically important events

Medical and scientific judgment should be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent 1 of the other outcomes listed in the definition above. These events, including those that may result in disability/incapacity, should also

EudraCT number 2015-002876-25


usually be considered serious. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

Safety events of interest on the medicinal products administered to the subject as part of the study (e.g., study drug, comparator, background therapy) that may require expedited reporting and/or safety evaluation include, but are not limited to:

- Overdose of the medicinal product(s)
- Suspected abuse/misuse of the medicinal product(s)
- Inadvertent or accidental exposure to the medicinal product(s)
- Medication error involving the medicinal product(s) (with or without subject exposure to the Sponsor medicinal product, e.g., name confusion)

All of the events of interest noted above should be recorded on the eCRF. Any situation involving these events of interest that also meets the criteria for an SAE should be recorded on the AE page of the eCRF and marked 'serious' and the SAE worksheet.

The Sponsor has a list of events that they classify as "always serious" events. If an AE is reported that is considered to be an event per this classification as "always serious", additional information on the event may be requested.

#### 5.5.3 Criteria for Causal Relationship to the Study Drug

AEs that fall under either "Possible" or "Probable" should be defined as "AEs whose relationship to the study drugs could not be ruled out".

| Causal relationship | Criteria for causal relationship |
|---|---|
| to the study drug | |
| Not Related | A clinical event, including laboratory test abnormality, with a |
| | temporal relationship to drug administration which makes a causal |
| | relationship improbable, and/or in which other drugs, chemicals o |
| | underlying disease provide plausible explanations. |
| Possible | A clinical event, including laboratory test abnormality, with a |
| | reasonable time sequence to administration of the drug, but which |
| | could also be explained by concurrent disease or other drugs or |
| | chemicals. Information on drug withdrawal may be lacking or |
| | unclear. |
| Probable | A clinical event, including laboratory test abnormality, with a |
| | reasonable time sequence to administration of the drug, unlikely to |
| | be attributed to concurrent disease or other drugs or chemicals, and |
| | which follows a clinically reasonable response on re- administration |
| | (rechallenge) or withdrawal (dechallenge). |

**Sponsor: APEB**EudraCT number 2015-002876-25


#### 5.5.4 Criteria for Defining the Severity of an Adverse Event

The investigator will use the following definitions to rate the severity of each AE

• Mild: No disruption of normal daily activities

Moderate: Affects normal daily activities
 Severe: Inability to perform daily activities

#### 5.5.5 Reporting of Serious Adverse Events

In the case of an SAE, the investigator must contact the CRO by telephone or fax/e-mail immediately (within 1 working day of awareness).

The investigator should complete and submit an SAE Worksheet containing all information that is required by the Regulatory Authorities to CRO by fax/e-mail immediately (within 1 working day of awareness). If the faxing/e-mailing of an SAE Worksheet is not possible or is not possible within 1 working day, the local drug safety contact should be informed by phone. Within 1 working day during weekdays or within 60 hours during weekends, whatever is shorter, after receipt of the information, the CRO will forward the SAE details to the Sponsor.

SAEs must be reported up to 28 days after the EOS visit or up to 28 days after early discontinuation of dosing.

For contact details, see [Section II Contact Details of Key Sponsor's Personnel. Please fax/email to:

Safety & Pharmacovigilance

Please use the country specific toll-free fax number provided on the SAE Fax cover sheet.

In case of fax failure, email:

If there are any questions, or if clarification is needed regarding the SAE, please contact the Sponsor's Medical Monitor/Expert or his/her designee (Section II).

Follow-up information for the event should be sent promptly (within 7 days of the initial notification).

Full details of the SAE should be recorded on the medical records and on the eCRF.

The following minimum information is required:

- International Study Number (ISN)
- Subject number, sex and age
- The date of report
- A description of the SAE (event, seriousness of the event) and
- Causal relationship to the study drug

Where required by local requirements, the Sponsor or Sponsor's designee will submit expedited safety reports (e.g., IND Safety Reports) to the regulatory agencies (e.g., FDA) as necessary, and will inform the investigators of such regulatory reports. Investigators must 02 Nov 2016

Astellas


EudraCT number 2015-002876-25


submit safety reports as required by their IEC/IRB within timelines set by regional regulations (i.e., EU, (e)CTD, FDA). Documentation of the submission to and receipt by the IEC/IRB of expedited safety reports should be retained by the site.

The delegated CRO will notify all investigators responsible for ongoing clinical studies with the study drug of all SAEs which require submission per local requirements.

The investigators should provide written documentation of IEC/IRB notification for each report to the Sponsor, where required by local requirements.

You may contact the Sponsor's Medical Monitor/Expert for any other problem related to the safety, welfare, or rights of the subject.

#### 5.5.6 Follow-up of Adverse Events

All AEs occurring during or after the subject has discontinued the study are to be followed up until resolved or judged to be no longer clinically significant, or until they become chronic to the extent that they can be fully characterized.

If during AE follow-up, the AE progresses to an SAE, or if a subject experiences a new SAE, the investigator must immediately report the information to the Sponsor.

Please refer to [Appendix 12.2] for detailed instructions on Drug Induced Liver Injury.

#### 5.5.7 Monitoring of Common Serious Adverse Events

Common serious adverse events are SAEs commonly anticipated to occur in the study population independent of drug exposure. For this protocol, there is no list of common serious adverse events that the Sponsor considers to be associated with the disease state being studied for which a single occurrence will be excluded from safety reporting.

## 5.5.8 Procedure in Case of Pregnancy

If a female subject or partner of a male subject becomes pregnant during the study dosing period or within 28 days from the discontinuation of dosing, the investigator should report the information to the CRO as if it is an SAE. The expected date of delivery or expected date of the end of the pregnancy, last menstruation, estimated conception date, pregnancy result and neonatal data etc., should be included in this information.

The investigator will follow the medical status of the mother, as well as the fetus, as if the pregnancy is an SAE and will report the outcome to the Sponsor.

When the outcome of the pregnancy falls under the criteria for SAEs [spontaneous abortion, induced abortion, stillbirth, death of newborn, congenital anomaly (including anomaly in a miscarried fetus)], the investigator should respond in accordance with the report procedure for SAEs.

Additional information regarding the outcome of a pregnancy (which is categorized as an SAE) is mentioned below.

• "Spontaneous abortion" includes miscarriage, abortion and missed abortion

- Death of an infant within 1 month after birth should be reported as an SAE regardless of its relationship with the study drug
- If an infant dies more than 1 month after the birth, it should be reported if a relationship between the death and intrauterine exposure to the study drug is judged as "possible" by the investigator
- In the case of a delivery of a living newborn, the "normality" of the infant is evaluated at the birth
- Unless a congenital anomaly is identified prior to spontaneous abortion or miscarriage, the embryo or fetus should be assessed for congenital defects by visual examination

## 5.5.9 Emergency Procedures and Management of Overdose

In the event of suspected mirabegron overdose, the subject should receive supportive care and monitoring. Heart rate, blood pressure and ECG monitoring are recommended. The Medical Monitor/Expert should be contacted as applicable.

#### 5.5.10 Supply of New Information Affecting the Conduct of the Study

When new information becomes available necessary for conducting the clinical study properly, the Sponsor will inform all investigators involved in the clinical study as well as the regulatory authorities. Investigators should inform the IEC/IRB of such information when needed.

## 5.6 Test Drug Concentration

Samples will be collected as per local standards, however a topical anesthetic cream or plaster must be offered at the point of venipuncture to minimize distress of the subject. Venous blood (2 mL) for bioanalysis of mirabegron will be collected in properly labeled tubes containing sodium-heparin as anticoagulant and sodium fluoride as stabilizer.

Blood samples will be kept on melting-ice until ready for centrifugation, which must be done within 30 minutes after collection. Blood samples will be centrifuged at 1500 g for 10 minutes at ambient temperature in order to obtain plasma. Plasma will be harvested and transferred into a properly labeled polypropylene tube and stored at -20°C or below (preferably at -70°C) within 30 minutes after centrifugation.

Plasma samples will be sent to the central laboratory, packed with sufficient dry ice, to keep the samples frozen during shipment. Bioanalysis of mirabegron in plasma will be done at a designated CRO using a validated liquid chromatography-tandem mass spectrometry method.

## 5.7 Other Measurements, Assessments or Methods

If deemed relevant, the remaining plasma may be used for retrospective mirabegron metabolite profiling, identification and/or quantification studies. Analysis of these metabolites will be done at Astellas or at a designated CRO using LC-MS/MS or other appropriate analytical techniques. The results from these tests will be described in (a) separate report(s) and will not be incorporated in the integrated clinical study report.

**Sponsor: APEB** EudraCT number 2015-002876-25


#### **5.8 Total Amount of Blood**

The total amount of blood that is to be taken as foreseen over the entire study period is approximately 25 to 30 mL per subject Table 5:

Table 5 Total Amount of Blood Volume per Subject During the Study Period

| Amount for pharmacokinetic sampling (2.0 mL/sample x 4 samples) | 8 mL |
|---|---|
| Amount for safety hematology & biochemistry † (5.5 mL/sample x 3‡ samples) | 16.5 mL |
| Total § | 24.5 mL |

- If applicable, pregnancy test will be done from the same sample; no additional blood is required.
- The first group of subjects (minimum of 5, maximum of 10) who reach study visit 5/week 4 will have an additional blood draw of about 5 mL at study visit 5/week 4 for DSMB safety monitoring. The total amount of blood drawn from these subjects will thus be approximately 30.0 mL
- Volume does not take any unscheduled visits or re-tests into account (e.g., follow-up of AEs)

#### 6 DISCONTINUATION

#### **Discontinuation of Individual Subject(s)** 6.1

A discontinuation is a subject who received study drugs and for whom study treatment is permanently discontinued prematurely for any reason.

The subject is free to withdraw from the study treatment and/or study for any reason and at any time without giving reason for doing so and without penalty or prejudice. The investigator is also free to terminate a subject's involvement in the study at any time if the subject's clinical condition warrants it.

If a subject is discontinued from the study with an ongoing AE or an unresolved laboratory result that is significantly outside of the reference range, the investigator will attempt to provide follow-up until the condition stabilizes or no longer is clinically significant.

Discontinuation criteria from treatment for individual subjects:

- If, within 7 days of the first dose of mirabegron:
  - The centrally read urodynamic trace reveals no evidence of NDO
  - The centrally read ECG has an average QTcB interval greater than 450 ms, based on the QTcB mean from the visit 1 and visit 3 ECG triplicates
- If signs or symptoms of hypersensitivity to mirabegron are observed (e.g., anaphylactic reaction, erytheme multiforme or exfoliative dermatitis).
- Discontinuation of treatment should be considered if:
  - $\circ$  ALT or AST  $> 8 \times ULN$
  - ALT or AST  $> 5 \times ULN$  for more than 2 weeks
  - ALT or AST  $> 3 \times$  ULN and TBL  $> 2 \times$  ULN or INR > 1.5) (If INR testing is applicable/evaluated)

02 Nov 2016 Astellas 

- $\circ$  ALT or AST > 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia ( > 5%).
- o In addition, if close monitoring for a subject with moderate or severe hepatic laboratory tests is not possible, the drug should be discontinued.

#### 6.2 Discontinuation of the Site

If an investigator intends to discontinue participation in the study, the investigator must immediately inform the Sponsor.

## 6.3 Discontinuation of the Study

The Sponsor may terminate this study prematurely, either in its entirety or at any study site, for reasonable cause provided that written notice is submitted in advance of the intended termination. Advance notice is not required if the study is stopped due to safety concerns. If the Sponsor terminates the study for safety reasons, the Sponsor will immediately notify the investigator and subsequently provide written instructions for study termination.

#### 7 STATISTICAL METHODOLOGY

The statistical analysis will be coordinated by the responsible biostatistician of Astellas. A Statistical Analysis Plan (SAP) will be written to provide details of the analysis, along with specifications for tables, listings and figures (TLFs) to be produced. The SAP will be finalized before the database soft lock at the latest. Any changes from the analyses planned in SAP will be justified in the clinical study report (CSR).

Prior to database lock, a final meeting will be held to allow a review of the clinical trial data and (TLFs) and to verify the data that will be used for analysis set classification. If required, consequences for the statistical analysis will be discussed and documented. A meeting to determine analysis set classifications may also be held prior to database lock.

In general, all data will be summarized with descriptive statistics (number of subjects, mean, standard deviation, minimum, median and maximum) for continuous endpoints, and frequency and percentage for categorical endpoints.

## 7.1 Sample Size

The primary endpoint will be the change from baseline in MCC after 24 weeks of mirabegron treatment. There are data from previous studies that indicate the effect size that can be expected as a result of the treatment with mirabegron. Franco et al. (2005) analyzed 2 age groups (1 to 5 years, and 6 to 15 years) and reported mean (SD) MCC changes from baseline of 71.5 (88) mL and 75.4 (102.7) mL respectively after 24 weeks treatment with oxybutynin. Goessl et al. (2000) reported an increase of 52.8 mL after 3 months treatment with tolterodine. Cartwright et al. (2009) reported an increase of 98 mL after 14 weeks treatment with oxybutynin and a corresponding SD of 87 mL.

EudraCT number 2015-002876-25


A study with 44 evaluable subjects who have valid (as by the central reviewer's assessment) nonmissing MCC measurements at visit 8/week 24 and at baseline would have a 90 percent power to detect a statistical significant change from baseline, if the real change from baseline in the subject population is at least 52 mL and the real SD for change from baseline is  $\leq 103$  mL. The power calculation was done assuming a paired t-test with 2-sided significance level of 0.05.

Assuming 30% of enrolled subjects will discontinue or will not be evaluable for the primary endpoint, a total of approximately 63 subjects may need to be enrolled so that 44 subjects are evaluable in total.

These sample size considerations should allow sufficient precision for the assessment of the primary objective in this nonrandomized pediatric trial.

Detailed criteria for analysis sets will be laid out in Classification Specifications and the allocation of subjects to analysis sets will be determined prior to database hard-lock.

## 7.2 Analysis Set

Detailed criteria for analysis sets will be laid out in Classification Specifications and the allocation of subjects to analysis sets will be determined prior to database hard-lock.

## 7.2.1 Full Analysis Set

The full analysis set (FAS) will consist of all subjects who:

- Took at least 1 dose of study drug, and
- Had a valid (as by the central reviewer's assessment) nonmissing MCC measurement at baseline and at a postbaseline visit for the primary efficacy endpoint.

The FAS will be used for primary analyses of efficacy data, for sensitivity and subgroup analyses [Section 7.4.1.3] and for summaries of some demographic and baseline characteristics.

#### 7.2.2 Per Protocol Set

The per protocol set (PPS) will include all subjects of the FAS who fulfill the protocol in terms of their eligibility, interventions and outcome assessments, and for whom valid MCC measurements at visit 3/baseline and at visit 8/week 24 are reported.

A list of the protocol deviations that may result in a subject in the FAS being excluded from the PPS will be provided in the SAP. The final selection of subjects for the PPS will be confirmed in the Analysis Set Classification Meeting based upon a review of all the pertinent data.

The PPS will be used for secondary analyses of efficacy data. Also, selected demographic and baseline characteristics may also be summarized for the PPS.

**Sponsor: APEB** EudraCT number 2015-002876-25


#### 7.2.3 Safety Analysis Set

The safety analysis set (SAF) will consist of all subjects who took at least 1 dose of study drug.

The SAF will be used for all summaries of demographic and baseline characteristics and all safety and tolerability related variables.

#### 7.2.4 Pharmacokinetics Analysis Set

The pharmacokinetics analysis set (PKAS) consists of the subset of subjects of the SAF for whom plasma concentration data are available to facilitate derivation of at least 1 pharmacokinetic parameter and for whom the time of last dose prior to sampling is known.

Additional subjects may be excluded from the PKAS at the discretion of the pharmacokineticist. Any formal definitions for exclusion of subjects or time points from the PKAS will be documented in the Classification Specifications.

Since the actual bioanalytical results may only become available after the data review meeting, additional data points may be excluded at the time of pharmacokinetic analysis at the discretion of the pharmacokineticist. These data points will be reported in the CSR.

## 7.3 Demographics and Other Baseline Characteristics

Demographic and other baseline characteristics will be summarized by using descriptive statistics. Summaries of demographic data will be provided for each analysis set within and across age groups.

## 7.4 Analysis of Efficacy

Efficacy analysis will be conducted on the FAS. The interpretation of results from statistical tests will be based on the FAS. The PPS will be used to assess the robustness of the results from the statistical tests based on the FAS.

## 7.4.1 Analyses of Primary Endpoint

#### 7.4.1.1 Primary Analysis

Baseline for efficacy variables is the last assessment made prior to the first intake of study drug at visit 3 (day -1).

The primary efficacy variable is change from baseline in MCC after 24 weeks of treatment (based on filling urodynamics). The primary analysis will be a paired t-test for the change from baseline to week 24 to test the hypothesis that the change from baseline in MCC is not equal to zero with a 2-sided alpha level of 0.05. A 95% CI will be calculated for mean change from baseline. It will be assessed whether the estimated lower bound of the 95% CI excludes 0 mL. No adjustment for multiplicity will be made.

Missing MCC observations at visit 8/week 24 will be imputed using the last observation carried forward method (LOCF). The data will be summarized with descriptive statistics as a continuous variable (n, mean, SD, SEM, 95% CI, min, median, max).

02 Nov 2016 Astellas 

EudraCT number 2015-002876-25


#### 7.4.1.2 Secondary Analyses

A repeat of the primary analysis will be performed on the FAS without imputing missing data as well as based on the PPS.

A repeated measures analysis of covariance (ANCOVA) will be performed considering the change from baseline (without LOCF) and baseline MCC. This analysis will serve as a sensitivity analysis to the LOCF methods used in the primary model to assess robustness of those findings. For this analysis, data will be windowed according to predefined study visit windows.

Details of these analyses, including study visit windows, will be provided in the SAP.

#### 7.4.1.3 Subgroup and Sensitivity Analyses of Primary Endpoint

For the primary efficacy endpoint, MCC, 95% CI will be calculated for mean change from baseline per age group, per formulation, and per dosing regimen (with and without LOCF).

Dosing regimen here refers to whether the subjects had been up-titrated to PED50 at least once or maintained at PED25 for safety reasons at least until visit 8/week 24.

A subgroup analysis of the primary efficacy endpoint by whether NDO medication treatment was received at screening/prior to start of washout for both groups of subjects will be performed if there are sufficient subject numbers (with and without LOCF) on the FAS.

A subgroup analysis of the primary efficacy endpoint of subjects with insufficient efficacy under antimuscarinics specifically intended for NDO treatment (i.e. stopping the medication for lack of efficacy prior to start of treatment) will be performed if there are sufficient subject numbers (with and without LOCF) on the FAS.

The following sensitivity analyses of the primary efficacy endpoint will be performed if there are sufficient subject numbers (without LOCF only) on the FAS:

- Excluding those subjects who had a positive urine culture at visit 3/baseline and/or visit 8/week 24.
- For any of the subgroups specified, at least 10 subjects by stratum are required.

#### 7.4.2 Analysis of Secondary Endpoints

Each of the secondary efficacy endpoints will be summarized and, if applicable, plotted by visit.

The change from baseline for secondary endpoint based on urodynamic assessments, the subject's e-diary (including bladder diary) and questionnaires will be summarized and analyzed using similar primary statistical methods as for the primary endpoint, where appropriate.

CGI-C and acceptability results will be tabulated per time point of assessment.

These analyses of secondary endpoints will be produced for subjects in the FAS. Details of these analyses and of any further analyses will be defined in the SAP.

**Sponsor: APEB** EudraCT number 2015-002876-25


#### 7.4.3 Analysis of Exploratory Endpoints

Each of the exploratory efficacy endpoints will be summarized and analyzed in the same way as the secondary efficacy endpoints [Section 7.4.2].

Details of these analyses and of any further analyses will be defined in the SAP.

### 7.5 Analysis of Safety

The baseline for safety variables is the last assessment made prior to first intake of study drug (visit 3/day -1).

For safety variables relating to the ECG intervals, baseline values are taken from the mean of the visit 1 and visit 3 mean values.

All safety data will be summarized descriptively based on the SAF. The continuous safety data will be summarized using the following descriptive statistics: n, mean, SD, min, median, max, at each time point and for change from baseline. Categorical data will be summarized by absolute and relative frequencies. All safety data from subjects in the SAF will be listed.

Safety parameters such as vital signs and weight will also be summarized with respect to height- and sex-specific percentiles. Height will also be summarized with respect to age- and sex-specific percentiles.

Subgroup presentations regarding age (children and adolescents), formulation (tablets and suspension) and dosing regimen (PED25 and PED 50) will be tabulated for the following parameters: AEs, vital signs and ECGs. For any of the subgroups specified, at least 10 subjects by stratum are required.

#### 7.5.1 Vital Signs

Descriptive statistics will be used to summarize vital sign results and changes from baseline by treatment group and time. For clinic measurements Z-scores and percentiles for SBP and DBP will be calculated and summarized based on a comparison with age and height norms supplied by the Center for Disease Control and Prevention.

Z-scores and percentiles for pulse rate will be calculated and summarized based on a comparison with age norms based on Fleming [Fleming et al, 2011].

#### 7.5.2 Adverse Events

AEs will be coded using MedDRA. The number and percentage of AEs, SAEs, AEs leading to discontinuation, and AEs related to study drug will be summarized by system organ class and preferred term. The number and percentage of AEs by severity will also be summarized.

#### 7.5.3 Laboratory Assessments

For quantitative laboratory measurements descriptive statistics will be used to summarize results and change from baseline time point. Shifts relative to normal ranges from baseline to each time point during treatment period in lab tests will also be tabulated.

#### 7.5.4 Physical Examination

Abnormal findings/conditions identified during the physical examinations will be summarized and listed as part of the medical history for the screening visit, or as AEs at later visits.

#### 7.5.5 Electrocardiograms

12-lead ECG parameters (QT, QT interval corrected by Fridericia's formula [QTcF], HR, PR, QRS and RR) and their changes from baseline will be summarized with descriptive statistics by visit. The following thresholds will be used to characterize an individual subject's QTcF data: QTcF interval > 440 ms for children, and QTcF interval > 450 ms and >500 ms for male adolescents and >480 ms and >500 ms for female adolescents. These categories are cumulative in that subjects satisfying criterion for a more extreme category will also be counted in each applicable less extreme category. A summary of normal, abnormal not clinical significant and abnormal clinical significant findings will be provided.

In addition for QTcF, the impact of concomitant medications potentially prolonging QTc will be evaluated.

To perform this analysis, all QTcF post-baseline values will be presented (regardless of time point). If anomalies occur, an additional presentation will be provided using only QTcF values not under the influence of respective concomitant medications.

Details on how these will be derived, will be described in the SAP.

### 7.5.6 Estimated Glomerular Filtration Rate and Upper Urinary Tract Ultrasound

For eGFR and upper urinary tract ultrasound, descriptive statistics will be used to summarize results and change from baseline by time point. The eGFR results will be summarized based upon the Larsson, the modified Schwartz 2009 (for children < 12 years old) and the Cockcroft-Gault equation (for adolescents).

#### 7.5.7 Analysis of Exploratory Endpoints

Each of the exploratory safety endpoints will be summarized and analyzed in the same way as the safety endpoints [Sections 7.5.1] to 7.5.6]. For SMIP descriptive statistics will be used to summarize results and change from baseline by time point.

All analyses of exploratory safety endpoints will be produced for subjects in the SAF.

Details of these analyses and of any further analyses will be defined in the SAP.

## 7.6 Analysis of Pharmacokinetics

Descriptive statistics (N, mean, SD, minimum, median, maximum, coefficient of variation and geometric mean) will be provided for plasma concentration data. Further details will be specified in the SAP.

EudraCT number 2015-002876-25


#### 7.6.1 Estimation of Pharmacokinetic Parameters

The plasma concentrations will be analyzed with nonlinear mixed effects modeling (population pharmacokinetics) using NONMEM (version 7.3 or higher, USA).

The following plasma pharmacokinetic parameters of mirabegron will be calculated for each subject:

• C<sub>max</sub>, t<sub>max</sub>, AUC<sub>24</sub>, C<sub>trough</sub>, CL/F and V<sub>z</sub>/F.

## 7.7 Protocol Deviations and Other Analyses

Protocol deviations as defined in [Section 8.1.6] will be summarized for all subjects by site. A data listing will be provided by site and subject.

The protocol deviation criteria will be uniquely identified in the summary table and listing. The unique identifiers will be as follows:

- PD1 Entered into the study even though they did not satisfy entry criteria,
- PD2 Developed withdrawal criteria during the study and was not withdrawn,
- PD3 Received wrong treatment or incorrect dose,
- PD4 Received excluded concomitant treatment.

Descriptive statistics will be used to explore whether there is an association between certain subject characteristics (such as medical history) and the final titrated mirabegron doses. Collected data on study drug compliance rates and maintenance of treatment will be analyzed using descriptive statistics.

# 7.8 Interim Analysis (and Early Discontinuation of the Clinical Study)

No formal interim analysis is planned.

# 7.9 Handling of Missing Data, Outliers, Visit Windows, and Other Information

As a general principle, no imputation of missing data (with exception of visit 8/week 24, LOCF analysis for MCC) will be performed. Values lower than the limit of quantification for laboratory parameters will be set to 0 for the calculation of descriptive statistics.

See the SAP for details of the definitions for windows to be used for analyses by visit.
#### 8 OPERATIONAL AND ADMINISTRATIVE CONSIDERATIONS

#### 8.1 Procedure for Clinical Study Quality Control

#### 8.1.1 Data Collection

The investigator or site designee will enter data collected using an Electronic Data Capture system. In the interest of collecting data in the most efficient manner, the investigator or site designee should record data (including laboratory values, if applicable) in the eCRF within 5 working days after the subject visit.

The investigator or site designee is responsible to ensure that all data in the eCRFs and queries are accurate and complete and that all entries are verifiable with source documents. These documents should be appropriately maintained by the site.

The monitor should verify the data in the eCRFs with source documents and confirm that there are no inconsistencies between them.

Laboratory tests (except for the locally performed pregnancy tests) are performed at a central laboratory and results are visible for the site shortly after analysis has been completed. Laboratory data will be transferred electronically to the Sponsor or designee at predefined intervals during the study. The laboratory will provide the Sponsor or designee with a complete and clean copy of the data.

ECG analysis and interpretation are performed at a central ECG reading vendor and results are visible for the site shortly after analysis has been completed. Central ECG read data will be transferred electronically to the Sponsor or designee at predefined intervals during the study. The central ECG vendor will provide the Sponsor or designee with a complete and clean copy of the data.

For Screen failures the demographic data, reason for failing, informed consent, inclusion and exclusion criteria and AEs will be collected in the eCRF and listed.

#### **8.1.1.1** Electronic Patient Reported Outcomes

Subject bladder diaries, questionnaires and other data completed by the subject or the subject's parent(s)/caregiver(s) will be entered on an electronic device (e-diary). The information on the electronic device will be automatically uploaded to a central website. The investigator or site designee should review the diaries and questionnaire data on the website for correct completion before each planned visit of the subject (on site or phone visit) and discuss the results or retrain the subject and/or subject's parent(s)/caregiver(s) if applicable. In case clinically relevant adverse changes are noticed during review of the e-diary, these will be recorded as an AE [Section 5.5.1].

The bladder diary, questionnaire results and other data collected in the e-diary will be transferred electronically to Sponsor or designee at predefined intervals during the study. The vendor will provide Sponsor or designee with a complete and clean copy of the data.


For this study the following information will be collected and entered by the subject or subject's parent(s)/caregiver(s) in the e-diary (see [Sections 5.3.2 5.3.3] and 5.4.1.2] for detailed information per visit):

- Bladder diary:
  - o Each day for 7 days: time of CICs
  - Each day for 7 days: presence of leakage between CICs
  - o Each day for 7 days: sleep time and wake-up time
  - o On the 2 weekend days: catheterized volume
  - o On the 2 weekend days: SMIP (if applicable)
  - o On the 2 weekend days: grade and number of leakages between CICs
  - o On the 2 weekend days (selected visits): weight of diaper/pad
- SBPM (blood pressure and pulse rate):
  - o On the 2 weekend days: triplicate measurements in the morning and evening
  - On 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM.
- Questionnaires: on 1 weekend day at selected visits
  - o PIN-Q
  - o PGI-S
  - Acceptability
- Confirmation of study drug intake: daily

The Investigator must guide the subject and subject's parent(s)/caregiver(s) to ensure that on the evening before and during the two weekend days of collection of catheterized volume and SMIP (if applicable), the subject's fluid intake should be regulated to an appropriate level taking e.g. age, sex and subject's condition into account. The intake must remain as consistent as possible on these volume collecting days throughout the entire study.

#### 8.1.2 Specification of Source Documents

Source data must be available at the site to document the existence of the study subjects and to substantiate the integrity of study data collected. Source data must include the original documents relating to the study, as well as the medical treatment and medical history of the subject.

The following information should be included in the source medical records (not exhaustive):

- Demographic data (e.g., date of birth/age, sex, race/ethnicity, height and body weight)
- Subject number
- Inclusion and exclusion criteria details
- Participation in study and original signed and dated informed consent forms (ICFs)
- Visit dates
- Dispensing and return of study drug details
- Medical history and physical examination details
- Key efficacy and safety data (as specified in the protocol)

Sponsor: APEB

EudraCT number 2015-002876-25


- AEs and concomitant medication
- Results of relevant examinations (e.g., ECG printouts, physical examination)
- Laboratory printouts
- Reason for premature discontinuation (if applicable)

#### 8.1.3 Clinical Study Monitoring

The Sponsor or delegated CRO is responsible for monitoring the clinical study to ensure that subject's human rights, safety, and well-being are protected, that the study is properly conducted in adherence to the current protocol and GCP, and study data reported by the investigator/sub-investigator are accurate and complete and that they are verifiable with study-related records such as source documents. The Sponsor is responsible for assigning study monitor(s) to this study for proper monitoring. They will monitor the study in accordance with planned monitoring procedures.

#### 8.1.4 Direct Access to Source Data/Documents

The investigator and the study site must accept monitoring and auditing by the Sponsor or delegated CRO as well as inspections from the IEC/IRB and relevant regulatory authorities. In these instances, they must provide all study-related records, such as source documents [Section 8.1.2] when they are requested by the Sponsor monitors and auditors, the IEC/IRB, or regulatory authorities. The confidentiality of the subjects' identities shall be well protected consistent with local and national regulations when the source documents are subject to direct access.

#### 8.1.5 Data Management

Data Management will be coordinated by the Global Data Science Department of the Sponsor in accordance with the SOPs for data management. All study-specific processes and definitions will be documented by Data Management. eCRF completion will be described in the eCRF instructions. Coding of medical terms and medications will be performed using MedDRA and the World Health Organization Drug Dictionary respectively.

#### **8.1.6** Protocol Deviations

A protocol deviation is generally an unplanned excursion from the protocol that is not implemented or intended as a systematic change. The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol and must protect the rights, safety, and welfare of subjects. The investigator should not implement any deviation from, or changes of, the protocol, unless it is necessary to eliminate an immediate hazard to trial subjects.

A protocol waiver is a documented prospective approval of a request from an investigator to deviate from the protocol. Protocol waivers are strictly prohibited.

ISN/Protocol 178-CL-206A

Sponsor: APEB
EudraCT number 2015-002876-25


For the purposes of this protocol, deviations requiring notification to Sponsor are defined as any subject who:

- Entered into the study even though they did not satisfy entry criteria†
- Developed withdrawal criteria during the study and not withdrawn
- Received wrong treatment or incorrect dose
- Received excluded concomitant treatment
- † Subjects who are discontinued within the first 7 days of dosing, after the centrally read urodynamic trace or the ECG results from visit 3/baseline show the subject is no longer fulfilling the eligibility criteria, will not result in a protocol deviation.

When a deviation from the protocol is identified for an individual subject, the investigator or designee must ensure the Sponsor is notified. The Sponsor will follow-up with the investigator, as applicable, to assess the deviation and the possible impact to the safety and/or efficacy of the subject to determine subject continuation in the study.

If a deviation impacts the safety of a subject, the investigator must contact the Sponsor immediately.

The investigator will also assure that deviations meeting IEC/IRB and applicable regulatory authorities' criteria are documented and communicated appropriately. All documentation and communications to the IEC/IRB and applicable regulatory authorities will be provided to the Sponsor and maintained within the Trial Master File.

NOTE: Other deviations outside of the categories defined above will be reported to the IEC/IRB as required in accordance with local requirements, as applicable.

#### **8.1.7** End of Trial in All Participating Countries

The end of trial in all participating countries is defined as the last subject's last visit.

### 8.2 Ethics and Protection of Subject Confidentiality

#### 8.2.1 Independent Ethics Committee/Competent Authorities

GCP requires that the clinical protocol, any protocol amendments, the IB, the informed consent/assent and all other forms of subject information related to the study (e.g., advertisements used to recruit subjects) and any other necessary documents be reviewed by an IEC/IRB. The IEC/IRB will review the ethical, scientific and medical appropriateness of the study before it is conducted. IEC/IRB approval of the protocol, informed consent/assent and subject information and/or advertising, as relevant, will be obtained prior to the authorization of drug shipment to a study site.

Any substantial amendments to the protocol will require IEC/IRB approval prior to implementation of the changes made to the study design at the site. The investigator will be required to submit, maintain and archive study essential documents according to ICH-GCP.

Any SAEs that meet reporting criteria, as dictated by local regulations, will be reported to both responsible Ethics Committees and Regulatory Agencies, as required. During the conduct of the study, the investigator should promptly provide written reports (e.g., ICH

Expedited Reports, and any additional reports required by local regulations) to the IEC/IRB of any changes that affect the conduct of the study and/or increase the risk to subjects. Written documentation of the submission to the IEC/IRB should also be provided to Sponsor.

If required by local regulations, the investigator shall make accurate and adequate written progress reports to the IEC/IRB at appropriate intervals, not exceeding 1 year. The investigator shall make an accurate and adequate final report to the IEC/IRB within 1 year after last subject out or termination of the study.

#### 8.2.2 Ethical Conduct of the Study

The study will be conducted in accordance with the protocol, ICH guidelines, applicable regulations and guidelines governing clinical study conduct and the ethical principles that have their origin in the Declaration of Helsinki.

#### 8.2.3 Informed Consent of Subjects

#### 8.2.3.1 Subject Information and Consent

For this pediatric study in subjects aged 3 to less than 18 years, in addition to information sheets and consent/assent forms for subjects (according to applicable local regulations), parent/legal guardian information sheets and consent forms will also be prepared.

Prior to any study-related screening procedures being performed on the subject, the informed consent statement will be reviewed and signed and dated by the subject, the subject's parent(s) or legal guardian(s), the person who administered the informed consent/assent, and any other signatories according to local requirements.

The following general rules apply but these may vary by local regulations for pediatric studies:

- The investigator/sub-investigator is responsible for explaining the nature and purpose of the study as well as other study-related matters to subjects and their parents or legal guardians, using the written information, and for obtaining the child's assent and the parent(s)'/guardian(s)' full understanding and written consent to participate in the study of their own free will.
- In cases where there might be an explicit wish of a minor or an incapacitated adult, who is capable of forming an opinion and assessing this information, to refuse to participate or to be withdrawn from the clinical trial at any time, this will have to be considered by the investigator, even if consent is given by the parent(s)/legal guardian(s). Every effort should be made to understand and respect differences of opinion between the subject and their parent(s)/legal guardian(s). Strong and definitive objections from the child should be respected.
- The investigator or other responsible personnel who provided explanations (including collaborators who gave supportive information, if applicable) and the subject and parent(s)/legal guardian(s) should sign and date the written information, or write down his/her name, and date the form.

- Informed consent/assent must be obtained prior to any study-related procedures (including discontinuation of prohibited medication, if applicable). Consent should be obtained from the subject and his/her parent(s)/legal guardian(s), before start of pre-investigational period. Assent and consent will be obtained per local regulations.
- The investigator or other responsible personnel must give a copy of the signed consent/assent form to the subject and parent(s)/legal guardian(s), and store the original appropriately in accordance with the rules at the study site concerned.
- The investigator or other responsible personnel should note the following when obtaining consent/assent from subjects and parent(s)/legal guardian(s):
  - No subject may be subjected to undue influence, such as compulsory enrollment into a study.
  - The language and expressions used in the written information should be as plain and understandable as possible. Subjects and their parent(s)/legal guardian(s) should be given the opportunity to ask questions and receive satisfactory answers to the inquiry, and should have adequate time to decide whether or not to participate in the study. Written information should not contain any language or contents that causes the subject to waive or appears to waive any legal rights, or that releases/mitigates or appears to release/mitigate the study site, the investigator/sub-investigator, collaborators, or the Sponsor from liability for negligence.

The signed consent forms will be retained by the investigator and made available (for review only) to the study monitor and auditor regulatory authorities and other applicable individuals upon request.

## 8.2.3.2 Supply of New and Important Information Influencing the Subject's Consent and Revision of the Written Information

- The investigator or his/her representative will immediately inform the subject or subject's parent(s)/guardian(s) orally whenever new information becomes available that may be relevant to the subject's consent or may influence the subject's willingness to continue to participate in the study (e.g., report of serious drug adverse drug reaction). The communication must be documented in the subject's medical records and must document whether the subject is willing to remain in the study or not.
- The investigator must update their ICF and submit it for approval to the IEC/IRB. The investigator or his/her representative must obtain written informed consent from the subject on all updated ICFs throughout their participation in the study. The investigator or his/her designee must reconsent subjects with the updated ICF even if relevant information was provided orally. The investigator or his/her representative who obtained the written informed consent and the subject should sign and date the informed consent form. A copy of the signed ICF will be given to the subject and the original will be placed in the subject's medical record. An entry must be made in the subject's records documenting the re-consent process.

#### 8.2.4 Subject Confidentiality

Individual subject medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited. Such medical information may be given only after approval of the subject to the subject's physician or to other appropriate medical personnel responsible for the subject's well-being.

The Sponsor shall not disclose any confidential information on subjects obtained during the performance of their duties in the clinical study without justifiable reasons.

The Sponsor affirms the subject's right to protection against invasion of privacy. Only a subject identification number and/or initials will identify subject data retrieved by the Sponsor. However, the Sponsor requires the investigator to permit the Sponsor, Sponsor's representative(s), the IEC/IRB and when necessary, representatives of the regulatory health authorities to review and/or to copy any medical records relevant to the study.

The Sponsor will ensure that the use and disclosure of protected health information obtained during a research study complies with the federal and/or regional legislation related to the privacy and protection of personal information.

#### **8.3** Administrative Matters

#### 8.3.1 Arrangement for Use of Information and Publication of the Clinical Study

Information concerning the study drug, patent applications, processes, unpublished scientific data, the IB and other pertinent information is confidential and remains the property of the Sponsor. Details should be disclosed only to the persons involved in the approval or conduct of the study. The investigator may use this information for the purpose of the study only. It is understood by the investigator that the Sponsor will use the information obtained during the clinical study in connection with the development of the drug and therefore may disclose it as required to other clinical investigators or to regulatory agencies. In order to allow for the use of the information derived from this clinical study, the investigator understands that he/she has an obligation to provide the Sponsor with all data obtained during the study.

Publication of the study results is discussed in the Clinical Study Agreement.

#### 8.3.2 Documents and Records Related to the Clinical Study

The investigator will archive all study data (e.g., Subject Identification Code List, source data, CRFs, and Investigator's File) and relevant correspondence. These documents are to be kept on file for the appropriate term determined by local regulation (for US sites, 2 years after approval of the NDA or discontinuation of the IND). The Sponsor will notify the site/investigator if the MAA is approved or if the IND/IMPD is discontinued. The investigator agrees to obtain the Sponsor's agreement prior to disposal, moving, or transferring of any study-related records. The Sponsor will archive and retain all documents pertaining to the study according to local regulations.

Data generated by the methods described in the protocol will be recorded in the subjects' medical records and/or study progress notes. All data will be entered on the eCRFs supplied for each subject.

The documents of the Efficacy and Safety Evaluation Committee (minutes and SOPs and others) and the judgment committee outside the study sites (minutes and SOPs and others) shall be retained by the Sponsor.

#### 8.3.3 Protocol Amendment and/or Revision

Any changes to the study that arise after approval of the protocol must be documented as protocol amendments: substantial amendments and/or nonsubstantial amendments. Depending on the nature of the amendment, either IEC/IRB, Competent Authority approval or notification may be required. The changes will become effective only after the approval of the Sponsor, the investigator, the regulatory authority, and the IEC/IRB (if applicable).

Amendments to this protocol must be signed by the Sponsor and the investigator. Written verification of IEC/IRB approval will be obtained before any amendment is implemented which affects subject safety or the evaluation of safety, and/or efficacy. Modifications to the protocol that are administrative in nature do not require IEC/IRB approval, but will be submitted to the IEC/IRB for their information, if required by local regulations.

If there are changes to the Informed Consent, written verification of IEC/IRB approval must be forwarded to the Sponsor. An approved copy of the new ICF must also be forwarded to the Sponsor.

#### 8.3.4 Insurance of Subjects and Others

The Sponsor has covered this study by means of an insurance of the study according to national requirements. The name and address of the relevant insurance company, the certificate of insurance, the policy number and the sum insured are provided in the Investigator's File.

#### 8.3.5 Signatory Investigator for Clinical Study Report

ICH E3 guidelines recommend and EU Directive 2001/83/EC requires that a final study report which forms part of a marketing authorization application be signed by the representative for the Coordinating Investigator(s) or the Principal Investigator(s). The representative for the Coordinating Investigator (s) or the Principal Investigator(s) will have the responsibility to review the final study results to confirm to the best of his/her knowledge it accurately describes the conduct and results of the study. The representative for Coordinating Investigator(s) or the Principal Investigator(s) will be selected from the participating investigators by the Sponsor prior to database lock.

**Sponsor: APEB** 

EudraCT number 2015-002876-25


#### 9 QUALITY ASSURANCE

The Sponsor is implementing and maintaining quality assurance and quality control systems with written SOPs to ensure that trials are conducted and data are generated, documented, recorded, and reported in compliance with the protocol, GCP, and applicable regulatory requirement(s).

The Sponsor or Sponsor's designee may arrange to audit the clinical study at any or all investigational sites and facilities. The audit may include on-site review of regulatory documents, case report forms, and source documents. Direct access to these documents will be required by the auditors.

#### 10 STUDY ORGANIZATION

# 10.1 Independent Data-Monitoring Committee | Data and Safety Monitoring Board | Monitoring Committee | Other Evaluation Committee(s)

A DSMB will be installed to act in an advisory capacity to the Sponsor to monitor participant safety and data quality.

Subject safety will be reviewed on a regular basis by the DSMB, who will advise the Sponsor on appropriate steps to protect study participants, which may include the early termination of the study.

A separate charter will describe the responsibilities, remit and timing of DSMB meetings.

#### 10.2 Other Study Organization

Not applicable.

#### 11 REFERENCES

- Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, et al. The standardization of terminology of lower urinary tract function in children and adolescents: update report from the Standardization Committee of the International Children's Continence Society. J. Urol. 2014;191:1863-5.
- Bauer SB, Austin PF, Rawashdeh YF, de Jong TP, Franco I, Siggard C, et al. International Children's Continence Society's recommendations for initial diagnostic evaluation and follow-up in congenital neuropathic bladder and bowel dysfunction in children. Neurourol Urodyn 2012;31:610-14.
- Bauer SB, Nijman RJ, Drzewiecki BA, Sillen U, Hoebeke P. International Children's Continence Society standardization report on urodynamic studies of the lower urinary tract in children. Neurourol Urodyn. 2015 May 21. doi:10.1002/nau.22783.
- Bower WF, Sit FK, Bluyssen N, Wong EM, Yeung CK. PinQ: a valid, reliable and reproducible quality-of-life measure in children with bladder dysfunction. J Pediatr Urol. 2006;2:185-9.
- Cartwright PC, Coplen DE, Kogan BA, Volinn W, Finan E, Hoel G. Efficacy and safety of transdermal and oral oxybutynin in children with neurogenic detrusor overactivity. J Urol. 2009;182:1548–54.
- Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. (1976); 16(1):31–41. doi:10.1159/000180580. PMID 1244564.
- de Zwart L, Scholten M, Monbaliu JG, Annaert PP, Van Houdt JM, Van den Wyngaert I, et al. The ontogeny of drug metabolizing enzymes and transporters in the rat. Reprod Toxicol. 2008;26:220-30.
- Food and Agriculture Organization of the United Nations; Food Safety and Quality: Online Edition: 'Combined compendium of food additive specifications'; 2015. Available from: <a href="http://www.fao.org/food/food-safety-quality/scientific-advice/jecfa-additivies/en/">http://www.fao.org/food/food-safety-quality/scientific-advice/jecfa-additivies/en/</a>
- Fleming S, Thompson M, Stevens R, Heneghan C, Plüddemann A, Maconochie I, et al. Normal ranges of heart rate and respiratory rate in children from birth to 18 years of age: a systematic review of observational studies. Lancet. 2011;377:1011-18.
- Franco I, Horowitz M, Grady R, Adams RC, de Jong TP, Lindert K, et al. Efficacy and safety of oxybutynin in children with detrusor hyperreflexia secondary to neurogenic bladder dysfunction. J. Urol. 2005;173:221-5.
- Goessl C, Sauter T, Michael T, Bergé B, Staehler M, Miller K. Efficacy and tolerability of tolterodine in children with detrusor hyperreflexia. Urology. 2000;55:414-8.
- Lafontan M, Berlan M. Fat cell adrenergic receptors and the control of white and brown fat cell function. J Lipid Res. 1993;34:1057-91.
- Larsson A, Malm J, Grubb A, Hansson LO. Calculation of glomerular filtration rate expressed in mL/min from plasma cystatin C values in mg/L. Scand J Clin Lab Invest 2004;64:25-30.
- McDowell MA, Fryar CD, Ogden CL, Flegal KM. Anthropometric reference data for children and adults: United States, 2003–2006. Natl Health Stat Report. 2008;22(10):1-48.
- Momper JD, Mulugeta Y, Green DJ, Karesh A, Krudys KM, Sachs HC, et al. Adolescent Dosing and Labeling Since the Food and Drug Administration Amendments Act of 2007. JAMA Pediatr. 2013;167(10):926-932. doi:10.1001/jamapediatrics.2013.465.

- Rawashdeh YF, Austin P, Siggaard C, Bauer SB, Franco I, de Jong TP, et al. International Children's Continence Society's Recommendations for Therapeutic Intervention in Congenital Neuropathic Bladder and Bowel Dysfunction in Children. Neurourol Urodyn 2012;31:615-20.
- Saghir SA, Khan SA, McCoy AT. Ontogeny of mammalian metabolizing enzymes in humans and animals used in toxicological studies. Crit Rev Toxicol 2012;42:323-57.
- Schwartz GJ, Muñoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, et al. New Equations to Estimate GFR in Children with CKD. J Am Soc Nephrol. 2009;20:629–37.
- Skobejko L. Mirabegron in management of neurogenic patients with resistance to anticholinergic medicaments. Paper presented at ICS2014 44th Annual Meeting of the International Continence Society (ICS), October 20-24, 2014, Rio de Janeiro, Brazil.
- Temple R. Hy's law: predicting serious hepatotoxicity. Pharmacoepidemiol Drug Saf. 2006;15:241-3.
- The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. U.S. Department of Health and Human Services, National Institutes of Health National Heart, Lung, and Blood Institute. NIH Publication No. 05-5267 Originally printed September 1996 (96-3790) Revised May 2005. Available from: https://www.nhlbi.nih.gov/files/docs/resources/heart/hbp\_ped.pdf
- Verpoorten C, Buyse GM. The neurogenic bladder: medical treatment. Pediatr Nephrol. 2008 May;23(5):717-25. Epub 2007 Dec 19.
- Wada N, Okazaki S, Kobayashi S, Hashizume K, Kita M, Matsumoto S, et al. Efficacy of combination therapy with mirabegron for anticholinergic-resistant neurogenic bladder: videourodynamic evaluation. Hinyokika Kiyo. 2015 Jan;61(1):7-11.
- Wöllner J, Pannek J. Initial experience with the treatment of neurogenic detrusor overactivity with a new β-3 agonist (mirabegron) in patients with spinal cord injury. Spinal Cord. 2015 Oct 27. doi: 10.1038/sc.2015.195. [Epub ahead of print].

#### 12 APPENDICES

#### 12.1 List of Excluded Concomitant Medications

Any medication used for the management of NDO (including tricyclic antidepressants, 1<sup>st</sup> generation H1-antagonists and alpha-blockers) and any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index and sensitive P-gp substrates.

Strong CYP3A4 inhibitors are excluded for subjects with mild to moderate renal impairment (mild: eGFR 60 to 89 mL/min; moderate: eGFR 30 to 59 mL/min).

Use of these medications is not permitted during the study phase. This list is <u>not exhaustive</u>. In case of doubt, the investigator should contact the local study monitor.

| Anticholinergics/ | Tricyclic antidepressants | 1 <sup>st</sup> generation H1- |
|---|---|---|
| antimuscarinics | | antagonists <sup>†</sup> |
| Darifenacin | Alimemazine / Trimipramine | Tripelennamine |
| Dicyclomine/Dicycloverine | Amitriptyline | Dimenhydrinate |
| Fesoterodine | Amoxapine | Clemastine |
| Flavoxate | Clomipramine | Bromazine |
| Isopropamide | Desipramine | Orphenadrine |
| Oxybutynin | Dosulepin/ Dothiepin | Doxylamine |
| Oxyphencyclimine | Doxepine | Carbinoxamine |
| Propantheline | Imipramine | Diphenhydramine |
| Propiverine | Lofepramine | Cyclizine |
| Tolterodine | Maprotiline | Chlorcyclizine |
| Trospium | Mianserin | Hydroxyzine |
| Solifenacin | Mirtazapine | Meclizine |
| | Nortriptyline | |
| | Protriptyline | |
| Alpha-blockers | CYP2D6 with narrow | Sensitive P-gp substrates |
| | therapeutic index | |
| Tamsulosin | Thioridazine | Digoxin |
| Alfuzosin | Flecainide | Dabigatran |
| Doxazosin | Propafenone | |
| Terazosin | Imipramine | |
| Silodosin | Desipramine | |
| Strong CYP3A4 inhibitors | Other | |
| Itraconazole | Mirabegron (except for study drug) | |
| Ketoconazole | Botulinum toxin | |
| Ritonavir | | |
| Clarthromycin | | |

<sup>†</sup> Incidental use for motion sickness is accepted.

#### 12.2 Liver Safety Monitoring and Assessment

Any subject enrolled in a clinical study with active drug therapy and reveals an increase of serum aminotransferases to  $> 3 \times \text{ULN}$ , or bilirubin  $> 2 \times \text{ULN}$ , should undergo detailed testing for liver enzymes (including at least ALT, AST, ALP) and TBL. Testing should be repeated within 48-72 hours of notification of the test results. For studies for which a central laboratory is used, alerts will be generated by the central lab regarding moderate and severe liver abnormality to inform the investigator, study monitor and study team. Subjects or his/her parent(s)/caregiver(s) should be asked if they have any symptoms suggestive of hepatobiliary dysfunction.

#### **Definition of Liver Abnormalities**

Confirmed abnormalities will be characterized as moderate and severe where ULN:

| Moderate | ALT or AST<br>> 3× ULN | or | Total Bilirubin > 2× ULN |
|----------|------------------------|-----|--------------------------|
| Severe* | > 3× ULN | and | > 2× ULN |

In addition, the subject should be considered to have severe hepatic abnormalities for any of the following:

- ALT or AST  $> 8 \times ULN$
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks
- ALT or AST > 3× ULN and International Normalized Ratio (INR) > 1.5 (If INR testing is applicable/evaluated).
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%).

The investigator may determine that abnormal liver function results, other than as described above, may qualify as moderate or severe abnormalities and require additional monitoring and follow-up.

#### **Follow-up Procedures**

Confirmed moderate and severe abnormalities in hepatic functions should be thoroughly characterized by obtaining appropriate expert consultations, detailed pertinent history, physical examination and laboratory tests. The site should complete the Liver Abnormality Case Report Form (LA-CRF) that has been developed globally and can be activated for any study or an appropriate document. Subjects with confirmed abnormal liver function testing should be followed as described below.

Confirmed moderately abnormal LFTs should be repeated 2-3 times weekly then weekly or less frequently if abnormalities stabilize or the study drug has been discontinued and the subject is asymptomatic.

Severe hepatic liver function abnormalities as defined above, in the absence of another etiology, may be considered an important medical event and may be reported as an SAE.

The Sponsor should be contacted and informed of all subjects for whom severe hepatic liver function abnormalities possibly attributable to study drug are observed.

To further assess abnormal hepatic laboratory findings, the investigator is expected to:

- Obtain a more detailed history of symptoms and prior or concurrent diseases. Symptoms and new onset-diseases should be recorded as 'adverse events' on the AE page of the eCRF. Illnesses and conditions such as hypotensive events, and decompensated cardiac disease that may lead to secondary liver abnormalities should be noted. Nonalcoholic steatohepatitis is seen in obese hyperlipoproteinemic, and/or diabetic subjects and may be associated with fluctuating aminotransferase levels. The investigator should ensure that the medical history form captures any illness that predates study enrollment that may be relevant in assessing hepatic function.
- Obtain a history of concomitant drug use (including nonprescription medication, complementary and alternative medications), alcohol use, recreational drug use, and special diets. Medications, including dose, should be entered on the concomitant medication page of the eCRF. Information on alcohol, other substance use, and diet should be entered on the LA-CRF or an appropriate document.
- Obtain a history of exposure to environmental chemical agents.
- Based on the subject's history, other testing may be appropriate including:
  - o acute viral hepatitis (A,B, C, D, E or other infectious agents)
  - o ultrasound or other imaging to assess biliary tract disease
  - o other laboratory tests including INR, direct bilirubin
- Consider gastroenterology or hepatology consultations.
- Submit results for any additional testing and possible etiology on the LA-CRF or an appropriate document.

#### **Study Discontinuation**

In the absence of an explanation for increased LFTs, such as viral hepatitis, pre-existing or acute liver disease or exposure to other agents associated with liver injury, the subject may be discontinued from the study. The investigator may determine that it is not in the subject's best interest to continue study enrollment. Discontinuation of treatment should be considered if:

- ALT or AST  $> 8 \times ULN$
- ALT or AST  $> 5 \times ULN$  for more than 2 weeks
- ALT or AST > 3  $\times$  ULN and TBL > 2  $\times$  ULN or INR > 1.5) (If INR testing is applicable/evaluated)
- ALT or AST > 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%).

In addition, if close monitoring for a subject with moderate or severe hepatic laboratory tests is not possible, the drug should be discontinued.

\*Hy's Law Definition-Drug-induced jaundice caused by hepatocellular injury, without a significant obstructive component, has a high rate of bad outcomes, from 10–50% mortality (or transplant). The 2 "requirements" for Hy's Law are:

Sponsor: APEB

EudraCT number 2015-002876-25


1) Evidence that a drug can cause hepatocellular-type injury, generally shown by an increase in transaminase elevations higher 3 times the upper limit of normal ("2 x ULN elevations are too common in treated and untreated subjects to be discriminating");

2) Cases of increased bilirubin (at least 2 x ULN) with concurrent transaminase elevations at least 3x ULN and no evidence of intra- or extra-hepatic bilirubin obstruction (elevated alkaline phosphatase) or Gilbert's syndrome [Temple 2006].

#### **Reference**

Guidance for Industry titled "Drug-Induced Liver Injury: Premarketing Clinical Evaluation" issued by FDA on July 2009.


#### 12.3 Laboratory Assessments

| | By Central | Laboratory |
|---|---|---|
| Assessment | Collecting tube | Parameters to be analyzed |
| Hematology | EDTA tube | HbA1c |
| | | Hemoglobin |
| | | Hematocrit |
| | | Platelets |
| | | Red blood cells |
| | | White blood cells |
| | | Differential white blood cell count |
| Biochemistry | Serum tube | Alanine aminotransferase |
| - | | Albumin |
| | | Alkaline phosphatase |
| | | Aspartate aminotransferase |
| | | Calcium |
| | | Chloride |
| | | Creatine phosphokinase |
| | | Creatinine |
| | | Cystatin C |
| | | Estimated glomerular filtration rate (Larsson, |
| | | modified Schwartz and Cockcroft-Gault) |
| | | Gamma-glutamyl transaminase |
| | | Glucose |
| | | hCG † |
| | | Lactate dehydrogenase |
| | | Potassium |
| | | Sodium |
| | | Total bilirubin |
| | | Total protein |
| | | Urea |
| | | Uric acid |
| Urinalysis | Dipstick | Protein |
| · | - | Glucose |
| | | pH |
| | | Urobilinogen |
| | | Bilirubin |
| | | Ketones |
| | | Nitrite |
| | Polypropylene tube | Casts |
| | | Crystals |
| | | Bacteria |
| | | Epithelial cells |
| | | Small round cells |
| | | Yeasts |
| | | Red blood cells |
| | | White blood cells <sup>‡</sup> |
| | Done I | Locally |
| Pregnancy | Urine | hCG <sup>†</sup> |

HbA1c: glycosylated hemoglobin A1c; hCG: human chorionic gonadotropin;

- † Only in female subjects of childbearing potential
- ‡ If white blood cell count is >100/μL (or '++' for semi-quantitative results) a urine culture will be done including an antibiotic sensitivity test.

Sponsor: APEB

EudraCT number 2015-002876-25


## 12.4 Pediatric Incontinence Questionnaire

| 1. I get shy because of my bladder problem |
|---|
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 2. People in my family treat me in a different way because of my bladder proble |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 3. I am worried that people might think my clothes smell of wee |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 4. I think that my bladder problem won't get better |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 5. Mum and Dad worry about me because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 6. I would feel better about myself if I didn't have a bladder problem |
| □ No □ Maybe □ Probably □ Yes □ Definitely |
| 7. My bladder problem makes me feel nervous |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 8. Mum or Dad sometimes seem a bit cranky because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 9. My bladder problem stops me going on sleepovers or holidays |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 10. My bladder problem makes me feel bad about myself |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 11. I wake up during my sleep because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 12. I miss out on doing things because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 13. I feel unhappy because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 14. My bladder problem makes me feel sad |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 15. I think about my bladder problem when choosing which sport to play |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 16. I have to go to the toilet when I'm watching a movie |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 17. If my bladder problem was fixed I would invite more friends to my house |
| □ No □ Maybe □ Probably □ Yes □ Definitely |
| 18. I choose hobbies that won't be spoiled by stopping to go to the toilet |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 19. My bladder problem makes me feel different to other people |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 20. I miss out on being with friends because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |

PINQ (UK-English) Astellas Pharma Europe Ltd FINAL V1 Oxford, Version 30NOV2011

Sponsor: APEB

EudraCT number 2015-002876-25


## 12.5 Patient Global Impression of Severity Scale

| How did you feel about your bladder condition <u>DURING THE PAST 3 DAYS?</u> | | | | |
|---|---|---|---|---|
| 0 | 1 | 2 | 3 | 4 |
| | | | ( <u>:</u> | $\odot$ |
| Really bad | Bad | Not bad, not<br>good | Good | Really good |

## 12.6 Acceptability Questionnaire for Tablets

| | | Questions | | |
|---|---|---|---|---|
| 1. How was t | 1. How was the <u>TASTE</u> of the study drug? | | | |
| 0 | 1 | 2 | 3 | 4 |
| Really bad | Bad | Not bad, not | Good | Really good |
| | | good | | |
| 2. How was i | t to <u>SWALLOV</u> | V the study drug | ? | |
| 0 | 1 | 2 | 3 | 4 |
| | | 2 | 3 | 4 |
| Really difficult | Difficult | Not difficult, not easy | Easy | 4 Really easy |

## 12.7 Acceptability Questionnaire for Oral Suspension

| Questions | | | | |
|---|---|---|---|---|
| 1. How was t | the <u>TASTE</u> of th | e study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| | $(\widehat{})$ | $\left(\frac{3}{2}\right)$ | $(\mathbb{Z})$ | |
| Really bad | Bad | Not bad, not<br>good | Good | Really good |
| 2. How was t | the <u>SMELL</u> of t | he study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| (••) | (·•) | | (••) | |
| D 11 1 1 | D. 1 | <u> </u> | Con-1 | |
| Really bad | Bad | Not bad, not<br>good | Good | Really Good |
| 3. How was i | t to <u>TAKE</u> the s | study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| (••) | $(\bullet \bullet)$ | | (· ·) | |
| | | ) | | |
| Really difficult | Difficult | Not difficult,<br>not easy | Easy | Really easy |

EudraCT number 2015-002876-25


| 4. How was it to PREPARE the study drug? | | | | |
|---|---|---|---|---|
| 0 1 2 3 4 | | | | |
| | $(\widetilde{})$ | ( <u>••</u> ) | ( | |
| Really difficult | Difficult | Not difficult,<br>not easy | Easy | Really easy |
| | | not easy | | |


## 12.8 Clinical Global Impression of Change Scale

| | Clinical Global Impression of Change Scale |
|---|---|
| Please rate the degree of change in the subject's overall bladder symptoms since the start of the study on day 1 (tick 1 box) | |
| | Very much improved |
| | Much improved |
| | Minimally improved |
| | No change |
| | Minimally worse |
| | Much worse |
| | Very much worse |

#### 12.9 Centiles of heart rate for normal children from birth to 18 years of age [Fleming et al, 2011]




## 12.10 CDC Data Table of Stature-for-age Chart for Males

Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 24 | 79.91084 | 80.72977 | 81.99171 | 84.10289 | 86.4522 | 88.80525 | 90.92619 | 92.19688 | 93.02265 |
| 24.5 | 80.26037 | 81.08868 | 82.36401 | 84.49471 | 86.86161 | 89.22805 | 91.35753 | 92.63177 | 93.45923 |
| 25.5 | 81.00529 | 81.83445 | 83.11387 | 85.25888 | 87.65247 | 90.05675 | 92.22966 | 93.53407 | 94.38278 |
| 26.5 | 81.73416 | 82.56406 | 83.84716 | 86.00517 | 88.42326 | 90.8626 | 93.07608 | 94.40885 | 95.27762 |
| 27.5 | 82.44846 | 83.27899 | 84.56534 | 86.73507 | 89.17549 | 91.64711 | 93.89827 | 95.25754 | 96.14512 |
| 28.5 | 83.14945 | 83.98045 | 85.26962 | 87.44977 | 89.91041 | 92.41159 | 94.69757 | 96.08149 | 96.98663 |
| 29.5 | 83.83819 | 84.66948 | 85.96098 | 88.15028 | 90.62908 | 93.15719 | 95.47522 | 96.88198 | 97.80345 |
| 30.5 | 84.51558 | 85.34694 | 86.64027 | 88.83745 | 91.33242 | 93.88496 | 96.23239 | 97.66027 | 98.59691 |
| 31.5 | 85.18238 | 86.01357 | 87.3082 | 89.51202 | 92.02127 | 94.59585 | 96.97022 | 98.41758 | 99.36828 |
| 32.5 | 85.83925 | 86.66999 | 87.9654 | 90.17464 | 92.69638 | 95.2908 | 97.68978 | 99.15514 | 100.1189 |
| 33.5 | 86.48678 | 87.3168 | 88.61244 | 90.82592 | 93.35847 | 95.97068 | 98.39218 | 99.87416 | 100.8501 |
| 34.5 | 87.12552 | 87.95452 | 89.24986 | 91.46645 | 94.00823 | 96.63637 | 99.07848 | 100.5759 | 101.5631 |
| 35.5 | 87.75597 | 88.58366 | 89.87816 | 92.0968 | 94.64637 | 97.28875 | 99.74979 | 101.2615 | 102.2593 |
| 36.5 | 88.37864 | 89.20473 | 90.49789 | 92.71756 | 95.27359 | 97.9287 | 100.4072 | 101.9324 | 102.9402 |
| 37.5 | 88.93297 | 89.77301 | 91.08608 | 93.3344 | 95.91475 | 98.58525 | 101.069 | 102.593 | 103.5983 |
| 38.5 | 89.47916 | 90.33306 | 91.66589 | 93.94268 | 96.54734 | 99.23358 | 101.7234 | 103.247 | 104.2503 |
| 39.5 | 90.01766 | 90.88532 | 92.23779 | 94.54291 | 97.17191 | 99.87426 | 102.3709 | 103.8948 | 104.8967 |
| 40.5 | 90.54891 | 91.43025 | 92.80225 | 95.13557 | 97.78898 | 100.5078 | 103.012 | 104.537 | 105.538 |
| 41.5 | 91.07337 | 91.96832 | 93.35972 | 95.72115 | 98.39903 | 101.1348 | 103.6473 | 105.1739 | 106.1747 |
| 42.5 | 91.59152 | 92.49999 | 93.91068 | 96.30009 | 99.00254 | 101.7556 | 104.2771 | 105.8061 | 106.8071 |
| 43.5 | 92.10382 | 93.0257 | 94.45556 | 96.87286 | 99.59998 | 102.3708 | 104.9021 | 106.434 | 107.4357 |
| 44.5 | 92.61073 | 93.54592 | 94.99482 | 97.43989 | 100.1918 | 102.9807 | 105.5225 | 107.0579 | 108.0609 |
| 45.5 | 93.11271 | 94.06109 | 95.52888 | 98.00159 | 100.7783 | 103.5858 | 106.1387 | 107.6784 | 108.683 |
| 46.5 | 93.61022 | 94.57166 | 96.05817 | 98.55838 | 101.36 | 104.1865 | 106.7513 | 108.2956 | 109.3024 |
| 47.5 | 94.10371 | 95.07806 | 96.5831 | 99.11064 | 101.9373 | 104.7831 | 107.3604 | 108.9101 | 109.9193 |
| 48.5 | 94.59361 | 95.5807 | 97.10407 | 99.65875 | 102.5105 | 105.3759 | 107.9665 | 109.522 | 110.5342 |
| 49.5 | 95.08035 | 96.08 | 97.62147 | 100.2031 | 103.0799 | 105.9654 | 108.5698 | 110.1317 | 111.1473 |
| 50.5 | 95.56435 | 96.57635 | 98.13566 | 100.7439 | 103.6459 | 106.5518 | 109.1706 | 110.7394 | 111.7588 |
| 51.5 | 96.046 | 97.07013 | 98.64701 | 101.2817 | 104.2087 | 107.1354 | 109.7693 | 111.3454 | 112.369 |
| 52.5 | 96.52568 | 97.5617 | 99.15585 | 101.8166 | 104.7687 | 107.7165 | 110.366 | 111.95 | 112.9781 |
| 53.5 | 97.00376 | 98.05141 | 99.6625 | 102.3491 | 105.3262 | 108.2953 | 110.9609 | 112.5533 | 113.5863 |
| 54.5 | 97.48058 | 98.53958 | 100.1673 | 102.8792 | 105.8813 | 108.872 | 111.5543 | 113.1555 | 114.1937 |
| 55.5 | 97.95648 | 99.02654 | 100.6705 | 103.4074 | 106.4343 | 109.4469 | 112.1464 | 113.7568 | 114.8006 |


#### Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 56.5 | 98.43175 | 99.51256 | 101.1723 | 103.9339 | 106.9855 | 110.0201 | 112.7374 | 114.3574 | 115.4072 |
| 57.5 | 98.90667 | 99.99791 | 101.6731 | 104.4588 | 107.535 | 110.5919 | 113.3273 | 114.9575 | 116.0134 |
| 58.5 | 99.38151 | 100.4828 | 102.173 | 104.9825 | 108.083 | 111.1623 | 113.9164 | 115.557 | 116.6194 |
| 59.5 | 99.8565 | 100.9676 | 102.6723 | 105.505 | 108.6296 | 111.7316 | 114.5047 | 116.1561 | 117.2254 |
| 60.5 | 100.3318 | 101.4523 | 103.1712 | 106.0265 | 109.1751 | 112.2998 | 115.0924 | 116.755 | 117.8314 |
| 61.5 | 100.8077 | 101.9372 | 103.6697 | 106.5472 | 109.7196 | 112.8671 | 115.6795 | 117.3536 | 118.4374 |
| 62.5 | 101.2843 | 102.4225 | 104.1682 | 107.0673 | 110.2631 | 113.4335 | 116.2661 | 117.9521 | 119.0435 |
| 63.5 | 101.7618 | 102.9082 | 104.6666 | 107.5868 | 110.8058 | 113.9992 | 116.8522 | 118.5505 | 119.6498 |
| 64.5 | 102.2401 | 103.3945 | 105.1651 | 108.1058 | 111.3477 | 114.5641 | 117.438 | 119.1487 | 120.2562 |
| 65.5 | 102.7195 | 103.8814 | 105.6638 | 108.6244 | 111.889 | 115.1284 | 118.0234 | 119.7469 | 120.8627 |
| 66.5 | 103.2 | 104.369 | 106.1627 | 109.1427 | 112.4296 | 115.6921 | 118.6084 | 120.345 | 121.4694 |
| 67.5 | 103.6815 | 104.8574 | 106.6619 | 109.6607 | 112.9696 | 116.2551 | 119.1931 | 120.943 | 122.0761 |
| 68.5 | 104.1642 | 105.3466 | 107.1614 | 110.1785 | 113.509 | 116.8176 | 119.7774 | 121.5408 | 122.6829 |
| 69.5 | 104.6479 | 105.8364 | 107.6611 | 110.696 | 114.0479 | 117.3794 | 120.3613 | 122.1384 | 123.2897 |
| 70.5 | 105.1326 | 106.327 | 108.1612 | 111.2132 | 114.5861 | 117.9407 | 120.9447 | 122.7359 | 123.8965 |
| 71.5 | 105.6183 | 106.8182 | 108.6614 | 111.7302 | 115.1238 | 118.5012 | 121.5277 | 123.333 | 124.5031 |
| 72.5 | 106.1048 | 107.3099 | 109.1619 | 112.2469 | 115.6609 | 119.0611 | 122.1101 | 123.9297 | 125.1095 |
| 73.5 | 106.5921 | 107.8021 | 109.6624 | 112.7631 | 116.1973 | 119.6203 | 122.6918 | 124.526 | 125.7156 |
| 74.5 | 107.0799 | 108.2946 | 110.1629 | 113.2789 | 116.7329 | 120.1786 | 123.2729 | 125.1217 | 126.3212 |
| 75.5 | 107.5682 | 108.7873 | 110.6633 | 113.7942 | 117.2678 | 120.7361 | 123.8532 | 125.7168 | 126.9263 |
| 76.5 | 108.0566 | 109.2801 | 111.1634 | 114.3089 | 117.8018 | 121.2926 | 124.4327 | 126.3111 | 127.5307 |
| 77.5 | 108.5451 | 109.7727 | 111.6631 | 114.8229 | 118.3348 | 121.848 | 125.0111 | 126.9045 | 128.1344 |
| 78.5 | 109.0335 | 110.2649 | 112.1623 | 115.336 | 118.8668 | 122.4024 | 125.5884 | 127.4969 | 128.7371 |
| 79.5 | 109.5214 | 110.7566 | 112.6608 | 115.8481 | 119.3977 | 122.9555 | 126.1646 | 128.0882 | 129.3387 |
| 80.5 | 110.0086 | 111.2476 | 113.1583 | 116.3592 | 119.9272 | 123.5073 | 126.7394 | 128.6782 | 129.9391 |
| 81.5 | 110.495 | 111.7375 | 113.6548 | 116.869 | 120.4554 | 124.0576 | 127.3128 | 129.2668 | 130.5381 |
| 82.5 | 110.9801 | 112.2263 | 114.1499 | 117.3774 | 120.9821 | 124.6064 | 127.8846 | 129.8538 | 131.1356 |
| 83.5 | 111.4638 | 112.7135 | 114.6436 | 117.8842 | 121.5072 | 125.1535 | 128.4547 | 130.4392 | 131.7314 |
| 84.5 | 111.9459 | 113.1991 | 115.1356 | 118.3893 | 122.0305 | 125.6987 | 129.023 | 131.0226 | 132.3253 |
| 85.5 | 112.4259 | 113.6827 | 115.6257 | 118.8926 | 122.552 | 126.2421 | 129.5893 | 131.6041 | 132.9172 |
| 86.5 | 112.9036 | 114.1642 | 116.1136 | 119.3938 | 123.0714 | 126.7834 | 130.1535 | 132.1834 | 133.507 |
| 87.5 | 113.3789 | 114.6431 | 116.5992 | 119.8927 | 123.5886 | 127.3225 | 130.7154 | 132.7605 | 134.0943 |
| 88.5 | 113.8513 | 115.1194 | 117.0822 | 120.3893 | 124.1035 | 127.8594 | 131.275 | 133.335 | 134.6792 |


#### Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 89.5 | 114.3206 | 115.5927 | 117.5625 | 120.8833 | 124.616 | 128.3937 | 131.8321 | 133.907 | 135.2615 |
| 90.5 | 114.7867 | 116.0629 | 118.0398 | 121.3746 | 125.1259 | 128.9256 | 132.3865 | 134.4763 | 135.8409 |
| 91.5 | 115.2491 | 116.5297 | 118.5139 | 121.863 | 125.6331 | 129.4547 | 132.9381 | 135.0426 | 136.4173 |
| 92.5 | 115.7077 | 116.9928 | 118.9847 | 122.3483 | 126.1374 | 129.981 | 133.4868 | 135.606 | 136.9906 |
| 93.5 | 116.1623 | 117.4521 | 119.4519 | 122.8305 | 126.6388 | 130.5044 | 134.0325 | 136.1662 | 137.5607 |
| 94.5 | 116.6127 | 117.9074 | 119.9153 | 123.3092 | 127.137 | 131.0247 | 134.5751 | 136.7231 | 138.1274 |
| 95.5 | 117.0587 | 118.3585 | 120.3749 | 123.7845 | 127.632 | 131.5419 | 135.1144 | 137.2767 | 138.6906 |
| 96.5 | 117.5 | 118.8053 | 120.8305 | 124.2562 | 128.1237 | 132.0559 | 135.6504 | 137.8267 | 139.2502 |
| 97.5 | 117.9366 | 119.2475 | 121.2819 | 124.7242 | 128.6119 | 132.5664 | 136.1829 | 138.3731 | 139.806 |
| 98.5 | 118.3683 | 119.6851 | 121.729 | 125.1882 | 129.0966 | 133.0736 | 136.7118 | 138.9159 | 140.358 |
| 99.5 | 118.7949 | 120.1179 | 122.1716 | 125.6484 | 129.5777 | 133.5771 | 137.2371 | 139.4548 | 140.9062 |
| 100.5 | 119.2165 | 120.5459 | 122.6099 | 126.1045 | 130.055 | 134.0771 | 137.7587 | 139.9899 | 141.4503 |
| 101.5 | 119.633 | 120.969 | 123.0435 | 126.5565 | 130.5286 | 134.5734 | 138.2765 | 140.5211 | 141.9904 |
| 102.5 | 120.0442 | 121.3872 | 123.4726 | 127.0044 | 130.9983 | 135.066 | 138.7905 | 141.0484 | 142.5263 |
| 103.5 | 120.4502 | 121.8004 | 123.897 | 127.4481 | 131.4641 | 135.5548 | 139.3006 | 141.5716 | 143.0582 |
| 104.5 | 120.851 | 122.2086 | 124.3168 | 127.8876 | 131.926 | 136.0397 | 139.8069 | 142.0908 | 143.586 |
| 105.5 | 121.2467 | 122.6119 | 124.7319 | 128.3228 | 132.384 | 136.5209 | 140.3093 | 142.6061 | 144.1096 |
| 106.5 | 121.6372 | 123.0103 | 125.1425 | 128.7539 | 132.8381 | 136.9982 | 140.8077 | 143.1173 | 144.6291 |
| 107.5 | 122.0228 | 123.4039 | 125.5485 | 129.1807 | 133.2882 | 137.4717 | 141.3023 | 143.6245 | 145.1445 |
| 108.5 | 122.4034 | 123.7928 | 125.9501 | 129.6035 | 133.7345 | 137.9414 | 141.793 | 144.1278 | 145.656 |
| 109.5 | 122.7793 | 124.1771 | 126.3473 | 130.0222 | 134.1769 | 138.4073 | 142.28 | 144.6272 | 146.1634 |
| 110.5 | 123.1506 | 124.5569 | 126.7402 | 130.4369 | 134.6155 | 138.8696 | 142.7632 | 145.1228 | 146.6671 |
| 111.5 | 123.5175 | 124.9325 | 127.1291 | 130.8477 | 135.0504 | 139.3282 | 143.2428 | 145.6148 | 147.167 |
| 112.5 | 123.8803 | 125.304 | 127.514 | 131.2548 | 135.4818 | 139.7833 | 143.7188 | 146.1032 | 147.6633 |
| 113.5 | 124.2391 | 125.6717 | 127.8953 | 131.6584 | 135.9097 | 140.235 | 144.1915 | 146.5882 | 148.1562 |
| 114.5 | 124.5943 | 126.0358 | 128.273 | 132.0585 | 136.3343 | 140.6835 | 144.661 | 147.0699 | 148.6459 |
| 115.5 | 124.9462 | 126.3966 | 128.6474 | 132.4555 | 136.7557 | 141.1289 | 145.1273 | 147.5486 | 149.1325 |
| 116.5 | 125.295 | 126.7544 | 129.0189 | 132.8495 | 137.1742 | 141.5713 | 145.5909 | 148.0245 | 149.6163 |
| 117.5 | 125.6413 | 127.1096 | 129.3876 | 133.2407 | 137.5899 | 142.0111 | 146.0518 | 148.4979 | 150.0977 |
| 118.5 | 125.9852 | 127.4624 | 129.754 | 133.6295 | 138.0032 | 142.4484 | 146.5103 | 148.9689 | 150.5767 |
| 119.5 | 126.3272 | 127.8132 | 130.1183 | 134.0161 | 138.4143 | 142.8835 | 146.9668 | 149.438 | 151.0539 |
| 120.5 | 126.6678 | 128.1625 | 130.4809 | 134.4008 | 138.8234 | 143.3168 | 147.4214 | 149.9053 | 151.5294 |
| 121.5 | 127.0073 | 128.5106 | 130.8422 | 134.7841 | 139.231 | 143.7484 | 147.8747 | 150.3714 | 152.0038 |


#### Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 122.5 | 127.3462 | 128.8579 | 131.2026 | 135.1663 | 139.6373 | 144.1789 | 148.3268 | 150.8365 | 152.4773 |
| 123.5 | 127.6851 | 129.2051 | 131.5625 | 135.5477 | 140.0427 | 144.6085 | 148.7782 | 151.301 | 152.9504 |
| 124.5 | 128.0243 | 129.5524 | 131.9224 | 135.9288 | 140.4477 | 145.0377 | 149.2294 | 151.7655 | 153.4235 |
| 125.5 | 128.3643 | 129.9004 | 132.2828 | 136.3101 | 140.8527 | 145.4669 | 149.6808 | 152.2303 | 153.8972 |
| 126.5 | 128.7058 | 130.2496 | 132.6441 | 136.692 | 141.2582 | 145.8965 | 150.1329 | 152.696 | 154.3718 |
| 127.5 | 129.0491 | 130.6005 | 133.0068 | 137.075 | 141.6646 | 146.3272 | 150.5861 | 153.1631 | 154.848 |
| 128.5 | 129.3949 | 130.9536 | 133.3714 | 137.4597 | 142.0725 | 146.7593 | 151.041 | 153.6321 | 155.3263 |
| 129.5 | 129.7436 | 131.3094 | 133.7386 | 137.8466 | 142.4824 | 147.1936 | 151.4982 | 154.1035 | 155.8072 |
| 130.5 | 130.0958 | 131.6686 | 134.1089 | 138.2362 | 142.8949 | 147.6305 | 151.9583 | 154.578 | 156.2913 |
| 131.5 | 130.452 | 132.0316 | 134.4828 | 138.6292 | 143.3107 | 148.0707 | 152.4218 | 155.0562 | 156.7792 |
| 132.5 | 130.8127 | 132.399 | 134.8608 | 139.0262 | 143.7304 | 148.5147 | 152.8894 | 155.5386 | 157.2715 |
| 133.5 | 131.1785 | 132.7714 | 135.2437 | 139.4278 | 144.1545 | 148.9633 | 153.3617 | 156.0258 | 157.7688 |
| 134.5 | 131.5498 | 133.1491 | 135.6318 | 139.8346 | 144.5838 | 149.4172 | 153.8394 | 156.5186 | 158.2717 |
| 135.5 | 131.9272 | 133.5329 | 136.026 | 140.2472 | 145.019 | 149.8769 | 154.323 | 157.0174 | 158.7806 |
| 136.5 | 132.311 | 133.9232 | 136.4266 | 140.6664 | 145.4607 | 150.3433 | 154.8133 | 157.5229 | 159.2964 |
| 137.5 | 132.7018 | 134.3205 | 136.8343 | 141.0928 | 145.9097 | 150.8169 | 155.3109 | 158.0356 | 159.8193 |
| 138.5 | 133.1 | 134.7252 | 137.2496 | 141.5269 | 146.3665 | 151.2984 | 155.8164 | 158.5562 | 160.35 |
| 139.5 | 133.5059 | 135.1378 | 137.673 | 141.9694 | 146.832 | 151.7885 | 156.3303 | 159.0851 | 160.889 |
| 140.5 | 133.9199 | 135.5588 | 138.105 | 142.4209 | 147.3066 | 152.2878 | 156.8532 | 159.6228 | 161.4365 |
| 141.5 | 134.3423 | 135.9885 | 138.5461 | 142.882 | 147.7911 | 152.7969 | 157.3857 | 160.1697 | 161.993 |
| 142.5 | 134.7733 | 136.4271 | 138.9968 | 143.3532 | 148.2859 | 153.3164 | 157.928 | 160.7262 | 162.5588 |
| 143.5 | 135.2132 | 136.8751 | 139.4573 | 143.835 | 148.7917 | 153.8466 | 158.4807 | 161.2924 | 163.1339 |
| 144.5 | 135.6621 | 137.3326 | 139.928 | 144.3277 | 149.3088 | 154.3881 | 159.0439 | 161.8686 | 163.7185 |
| 145.5 | 136.1202 | 137.7998 | 140.4091 | 144.8317 | 149.8376 | 154.941 | 159.6179 | 162.4549 | 164.3126 |
| 146.5 | 136.5875 | 138.2769 | 140.9009 | 145.3473 | 150.3784 | 155.5056 | 160.2026 | 163.0511 | 164.916 |
| 147.5 | 137.064 | 138.7638 | 141.4034 | 145.8746 | 150.9313 | 156.0819 | 160.7981 | 163.6571 | 165.5285 |
| 148.5 | 137.5496 | 139.2605 | 141.9167 | 146.4137 | 151.4964 | 156.6699 | 161.4041 | 164.2726 | 166.1497 |
| 149.5 | 138.0442 | 139.767 | 142.4407 | 146.9645 | 152.0735 | 157.2694 | 162.0203 | 164.8972 | 166.7791 |
| 150.5 | 138.5477 | 140.2831 | 142.9752 | 147.5269 | 152.6624 | 157.88 | 162.6462 | 165.5302 | 167.416 |
| 151.5 | 139.0597 | 140.8085 | 143.52 | 148.1005 | 153.2627 | 158.5012 | 163.2811 | 166.1711 | 168.0596 |
| 152.5 | 139.5799 | 141.3429 | 144.0746 | 148.6849 | 153.8738 | 159.1324 | 163.9243 | 166.8187 | 168.7091 |
| 153.5 | 140.108 | 141.8859 | 144.6388 | 149.2795 | 154.4951 | 159.7725 | 164.5748 | 167.4723 | 169.3634 |
| 154.5 | 140.6435 | 142.4369 | 145.2117 | 149.8836 | 155.1255 | 160.4207 | 165.2314 | 168.1305 | 170.0213 |


#### Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 155.5 | 141.1858 | 142.9955 | 145.7928 | 150.4962 | 155.7642 | 161.0758 | 165.893 | 168.7923 | 170.6817 |
| 156.5 | 141.7345 | 143.5608 | 146.3813 | 151.1165 | 156.4099 | 161.7364 | 166.5581 | 169.4561 | 171.343 |
| 157.5 | 142.2889 | 144.1322 | 146.9763 | 151.7433 | 157.0612 | 162.401 | 167.2253 | 170.1205 | 172.004 |
| 158.5 | 142.8482 | 144.7089 | 147.5767 | 152.3754 | 157.7168 | 163.0682 | 167.8929 | 170.784 | 172.663 |
| 159.5 | 143.4118 | 145.29 | 148.1815 | 153.0113 | 158.3751 | 163.7363 | 168.5594 | 171.445 | 173.3186 |
| 160.5 | 143.9788 | 145.8746 | 148.7896 | 153.6498 | 159.0344 | 164.4035 | 169.2231 | 172.1018 | 173.9691 |
| 161.5 | 144.5483 | 146.4615 | 149.3998 | 154.2892 | 159.6931 | 165.0681 | 169.8822 | 172.7528 | 174.6131 |
| 162.5 | 145.1196 | 147.0498 | 150.0107 | 154.928 | 160.3493 | 165.7283 | 170.535 | 173.3965 | 175.249 |
| 163.5 | 145.6915 | 147.6385 | 150.621 | 155.5647 | 161.0015 | 166.3823 | 171.1798 | 174.0312 | 175.8753 |
| 164.5 | 146.2633 | 148.2262 | 151.2295 | 156.1977 | 161.6478 | 167.0284 | 171.8151 | 174.6554 | 176.4906 |
| 165.5 | 146.8339 | 148.812 | 151.8348 | 156.8253 | 162.2865 | 167.665 | 172.4393 | 175.2677 | 177.0935 |
| 166.5 | 147.4023 | 149.3947 | 152.4355 | 157.4462 | 162.9161 | 168.2905 | 173.0509 | 175.8668 | 177.6829 |
| 167.5 | 147.9674 | 149.9731 | 153.0304 | 158.0587 | 163.535 | 168.9033 | 173.6486 | 176.4515 | 178.2575 |
| 168.5 | 148.5284 | 150.5461 | 153.6181 | 158.6615 | 164.1418 | 169.5022 | 174.2313 | 177.0206 | 178.8165 |
| 169.5 | 149.0842 | 151.1127 | 154.1975 | 159.2532 | 164.7352 | 170.0859 | 174.7978 | 177.5733 | 179.3589 |
| 170.5 | 149.6338 | 151.6717 | 154.7674 | 159.8327 | 165.314 | 170.6535 | 175.3473 | 178.1088 | 179.884 |
| 171.5 | 150.1763 | 152.2221 | 155.3268 | 160.3988 | 165.8771 | 171.2039 | 175.879 | 178.6264 | 180.3913 |
| 172.5 | 150.7107 | 152.763 | 155.8746 | 160.9506 | 166.4236 | 171.7364 | 176.3923 | 179.1256 | 180.8804 |
| 173.5 | 151.2363 | 153.2935 | 156.4099 | 161.4872 | 166.9528 | 172.2504 | 176.8868 | 179.6061 | 181.3509 |
| 174.5 | 151.7521 | 153.8127 | 156.9319 | 162.0078 | 167.4641 | 172.7455 | 177.3622 | 180.0676 | 181.8027 |
| 175.5 | 152.2575 | 154.32 | 157.4399 | 162.5118 | 167.9571 | 173.2213 | 177.8183 | 180.5102 | 182.2358 |
| 176.5 | 152.7517 | 154.8147 | 157.9334 | 162.9988 | 168.4313 | 173.6778 | 178.2551 | 180.9338 | 182.6503 |
| 177.5 | 153.2342 | 155.2961 | 158.4118 | 163.4685 | 168.8867 | 174.1148 | 178.6727 | 181.3385 | 183.0463 |
| 178.5 | 153.7043 | 155.7638 | 158.8747 | 163.9205 | 169.3231 | 174.5324 | 179.0712 | 181.7247 | 183.4242 |
| 179.5 | 154.1615 | 156.2174 | 159.3218 | 164.3547 | 169.7405 | 174.9309 | 179.451 | 182.0927 | 183.7842 |
| 180.5 | 154.6056 | 156.6566 | 159.7529 | 164.7713 | 170.1393 | 175.3105 | 179.8124 | 182.4429 | 184.127 |
| 181.5 | 155.036 | 157.0811 | 160.168 | 165.1701 | 170.5195 | 175.6716 | 180.1559 | 182.7757 | 184.4528 |
| 182.5 | 155.4526 | 157.4907 | 160.5669 | 165.5514 | 170.8815 | 176.0146 | 180.482 | 183.0918 | 184.7624 |
| 183.5 | 155.8552 | 157.8853 | 160.9498 | 165.9154 | 171.2257 | 176.34 | 180.7912 | 183.3916 | 185.0562 |
| 184.5 | 156.2436 | 158.265 | 161.3167 | 166.2625 | 171.5525 | 176.6483 | 181.0841 | 183.6757 | 185.3349 |
| 185.5 | 156.6178 | 158.6298 | 161.6679 | 166.5929 | 171.8626 | 176.9402 | 181.3614 | 183.9449 | 185.599 |
| 186.5 | 156.9777 | 158.9798 | 162.0035 | 166.9072 | 172.1563 | 177.2163 | 181.6236 | 184.1997 | 185.8493 |
| 187.5 | 157.3235 | 159.315 | 162.3239 | 167.2057 | 172.4343 | 177.4771 | 181.8715 | 184.4408 | 186.0863 |


#### Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 188.5 | 157.6551 | 159.6359 | 162.6294 | 167.489 | 172.6972 | 177.7234 | 182.1056 | 184.6687 | 186.3107 |
| 189.5 | 157.9729 | 159.9425 | 162.9204 | 167.7576 | 172.9456 | 177.9558 | 182.3267 | 184.8843 | 186.5231 |
| | 158.277 | 160.2352 | 163.1973 | 168.012 | 173.1801 | 178.175 | 182.5353 | 185.0879 | 186.724 |
| 191.5 | 158.5676 | 160.5143 | 163.4605 | 168.2528 | 173.4014 | 178.3815 | 182.7322 | 185.2804 | 186.9142 |
| 192.5 | 158.845 | 160.7802 | 163.7104 | 168.4805 | 173.6101 | 178.5762 | 182.9179 | 185.4623 | 187.0941 |
| 193.5 | 159.1095 | 161.0332 | 163.9476 | 168.6958 | 173.8067 | 178.7595 | 183.0931 | 185.6341 | 187.2643 |
| 194.5 | 159.3614 | 161.2738 | 164.1725 | 168.8991 | 173.992 | 178.9321 | 183.2583 | 185.7965 | 187.4254 |
| 195.5 | 159.6011 | 161.5023 | 164.3856 | 169.0911 | 174.1665 | 179.0946 | 183.414 | 185.9498 | 187.5779 |
| 196.5 | 159.829 | 161.7191 | 164.5873 | 169.2722 | 174.3308 | 179.2476 | 183.5609 | 186.0948 | 187.7222 |
| 197.5 | 160.0455 | 161.9247 | 164.7782 | 169.4431 | 174.4854 | 179.3915 | 183.6995 | 186.2318 | 187.8588 |
| 198.5 | 160.2508 | 162.1196 | 164.9587 | 169.6041 | 174.631 | 179.5271 | 183.8302 | 186.3613 | 187.9881 |
| 199.5 | 160.4456 | 162.3041 | 165.1292 | 169.756 | 174.768 | 179.6547 | 183.9535 | 186.4837 | 188.1106 |
| 200.5 | 160.63 | 162.4786 | 165.2903 | 169.8991 | 174.8969 | 179.7748 | 184.0699 | 186.5995 | 188.2267 |
| 201.5 | 160.8046 | 162.6437 | 165.4424 | 170.0339 | 175.0182 | 179.888 | 184.1797 | 186.7091 | 188.3368 |
| 202.5 | 160.9697 | 162.7997 | 165.586 | 170.1608 | 175.1323 | 179.9946 | 184.2835 | 186.8128 | 188.4411 |
| 203.5 | 161.1258 | 162.947 | 165.7214 | 170.2804 | 175.2398 | 180.095 | 184.3815 | 186.911 | 188.54 |
| 204.5 | 161.2733 | 163.086 | 165.8491 | 170.3931 | 175.341 | 180.1896 | 184.4741 | 187.004 | 188.6338 |
| 205.5 | 161.4125 | 163.2172 | 165.9694 | 170.4991 | 175.4362 | 180.2789 | 184.5617 | 187.0922 | 188.7229 |
| 206.5 | 161.5438 | 163.3409 | 166.0828 | 170.599 | 175.5259 | 180.3631 | 184.6446 | 187.1757 | 188.8075 |
| 207.5 | 161.6676 | 163.4575 | 166.1897 | 170.693 | 175.6104 | 180.4426 | 184.723 | 187.255 | 188.8878 |
| 208.5 | 161.7843 | 163.5673 | 166.2903 | 170.7816 | 175.6901 | 180.5176 | 184.7972 | 187.3302 | 188.9642 |
| 209.5 | 161.8942 | 163.6708 | 166.3851 | 170.865 | 175.7652 | 180.5885 | 184.8676 | 187.4016 | 189.0368 |
| 210.5 | 161.9977 | 163.7682 | 166.4743 | 170.9436 | 175.836 | 180.6555 | 184.9343 | 187.4694 | 189.1058 |
| 211.5 | 162.0951 | 163.8598 | 166.5583 | 171.0176 | 175.9028 | 180.7189 | 184.9975 | 187.5338 | 189.1715 |
| 212.5 | 162.1866 | 163.9461 | 166.6373 | 171.0873 | 175.9658 | 180.7789 | 185.0576 | 187.5951 | 189.234 |
| 213.5 | 162.2727 | 164.0272 | 166.7116 | 171.1529 | 176.0254 | 180.8357 | 185.1146 | 187.6534 | 189.2936 |
| 214.5 | 162.3537 | 164.1034 | 166.7816 | 171.2148 | 176.0816 | 180.8895 | 185.1687 | 187.7088 | 189.3503 |
| 215.5 | 162.4297 | 164.1751 | 166.8474 | 171.2732 | 176.1348 | 180.9405 | 185.2202 | 187.7617 | 189.4044 |
| 216.5 | 162.5011 | 164.2424 | 166.9094 | 171.3282 | 176.185 | 180.9889 | 185.2692 | 187.812 | 189.456 |
| 217.5 | 162.5681 | 164.3057 | 166.9676 | 171.3801 | 176.2326 | 181.0348 | 185.3159 | 187.86 | 189.5052 |
| 218.5 | 162.631 | 164.3651 | 167.0224 | 171.429 | 176.2776 | 181.0784 | 185.3603 | 187.9057 | 189.5522 |
| 219.5 | 162.69 | 164.4209 | 167.074 | 171.4752 | 176.3202 | 181.1199 | 185.4026 | 187.9494 | 189.5971 |
| 220.5 | 162.7453 | 164.4733 | 167.1224 | 171.5188 | 176.3606 | 181.1593 | 185.443 | 187.9911 | 189.6399 |

http://www.cdc.gov/growthcharts/html\_charts/statage.htm/#males


#### Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 221.5 | 162.7972 | 164.5224 | 167.168 | 171.5599 | 176.3989 | 181.1968 | 185.4815 | 188.0309 | 189.6809 |
| 222.5 | 162.8458 | 164.5686 | 167.2109 | 171.5988 | 176.4352 | 181.2325 | 185.5182 | 188.069 | 189.7201 |
| 223.5 | 162.8914 | 164.6119 | 167.2513 | 171.6355 | 176.4697 | 181.2666 | 185.5534 | 188.1054 | 189.7575 |
| 224.5 | 162.9341 | 164.6526 | 167.2892 | 171.6701 | 176.5024 | 181.299 | 185.5869 | 188.1402 | 189.7934 |
| 225.5 | 162.9741 | 164.6907 | 167.325 | 171.7029 | 176.5335 | 181.33 | 185.619 | 188.1736 | 189.8277 |
| 226.5 | 163.0115 | 164.7265 | 167.3585 | 171.7339 | 176.563 | 181.3595 | 185.6497 | 188.2055 | 189.8606 |
| 227.5 | 163.0465 | 164.76 | 167.3902 | 171.7632 | 176.5911 | 181.3877 | 185.6791 | 188.236 | 189.8922 |
| 228.5 | 163.0793 | 164.7915 | 167.4199 | 171.791 | 176.6179 | 181.4147 | 185.7073 | 188.2653 | 189.9224 |
| 229.5 | 163.11 | 164.821 | 167.4479 | 171.8172 | 176.6433 | 181.4405 | 185.7343 | 188.2934 | 189.9513 |
| 230.5 | 163.1387 | 164.8487 | 167.4742 | 171.8421 | 176.6676 | 181.4651 | 185.7601 | 188.3204 | 189.9791 |
| 231.5 | 163.1656 | 164.8746 | 167.499 | 171.8657 | 176.6907 | 181.4887 | 185.7849 | 188.3462 | 190.0058 |
| 232.5 | 163.1907 | 164.8989 | 167.5224 | 171.888 | 176.7127 | 181.5113 | 185.8087 | 188.3711 | 190.0314 |
| 233.5 | 163.2142 | 164.9217 | 167.5444 | 171.9091 | 176.7337 | 181.533 | 185.8316 | 188.3949 | 190.056 |
| 234.5 | 163.2361 | 164.9431 | 167.5651 | 171.9292 | 176.7538 | 181.5538 | 185.8535 | 188.4178 | 190.0797 |
| 235.5 | 163.2566 | 164.9631 | 167.5846 | 171.9483 | 176.773 | 181.5737 | 185.8746 | 188.4399 | 190.1024 |
| 236.5 | 163.2757 | 164.9819 | 167.6029 | 171.9663 | 176.7913 | 181.5928 | 185.8949 | 188.461 | 190.1242 |
| 237.5 | 163.2936 | 164.9995 | 167.6203 | 171.9835 | 176.8088 | 181.6111 | 185.9144 | 188.4814 | 190.1452 |
| 238.5 | 163.3103 | 165.016 | 167.6366 | 171.9998 | 176.8255 | 181.6287 | 185.9331 | 188.501 | 190.1654 |
| 239.5 | 163.3259 | 165.0315 | 167.6519 | 172.0153 | 176.8415 | 181.6456 | 185.9512 | 188.5198 | 190.1849 |
| 240 | 163.3333 | 165.0389 | 167.6593 | 172.0227 | 176.8492 | 181.6538 | 185.9599 | 188.529 | 190.1943 |

## 12.11 CDC Data Table of Stature-for-age Chart for Females

#### Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 24 | 78.43754 | 79.25982 | 80.52476 | 82.63524 | 84.97556 | 87.31121 | 89.40951 | 90.66355 | 91.47729 |
| 24.5 | 78.82133 | 79.64777 | 80.91946 | 83.04213 | 85.39732 | 87.74918 | 89.86316 | 91.12707 | 91.94741 |
| 25.5 | 79.60198 | 80.44226 | 81.73541 | 83.8943 | 86.29026 | 88.68344 | 90.83505 | 92.12168 | 92.95685 |
| 26.5 | 80.37555 | 81.22666 | 82.53699 | 84.72592 | 87.15714 | 89.58751 | 91.77421 | 93.08254 | 93.93209 |
| 27.5 | 81.1357 | 81.9954 | 83.31968 | 85.53389 | 87.99602 | 90.46018 | 92.67969 | 94.00873 | 94.87215 |
| 28.5 | 81.87746 | 82.74411 | 84.07998 | 86.31589 | 88.80551 | 91.30065 | 93.55097 | 94.89974 | 95.77649 |
| 29.5 | 82.59712 | 83.46957 | 84.81532 | 87.07028 | 89.58477 | 92.10859 | 94.38793 | 95.75551 | 96.64505 |
| 30.5 | 83.29206 | 84.16953 | 85.52398 | 87.79609 | 90.33342 | 92.88403 | 95.19083 | 96.57635 | 97.47814 |
| 31.5 | 83.96065 | 84.84264 | 86.205 | 88.49291 | 91.05154 | 93.62741 | 95.9603 | 97.36295 | 98.27646 |
| 32.5 | 84.6021 | 85.4883 | 86.85807 | 89.16084 | 91.73964 | 94.33951 | 96.69729 | 98.11632 | 99.04107 |
| 33.5 | 85.2163 | 86.10656 | 87.48344 | 89.80045 | 92.39854 | 95.0214 | 97.40303 | 98.83778 | 99.77332 |
| 34.5 | 85.80379 | 86.69803 | 88.08186 | 90.4127 | 93.02945 | 95.67446 | 98.07904 | 99.52891 | 100.4748 |
| 35.5 | 86.36557 | 87.26379 | 88.6545 | 90.99891 | 93.63382 | 96.30029 | 98.72705 | 100.1915 | 101.1474 |
| 36.5 | 86.90307 | 87.80528 | 89.20285 | 91.56066 | 94.21336 | 96.90071 | 99.34899 | 100.8276 | 101.7931 |
| 37.5 | 87.43482 | 88.34236 | 89.74875 | 92.12298 | 94.79643 | 97.50724 | 99.97896 | 101.4726 | 102.4485 |
| 38.5 | 87.95945 | 88.87256 | 90.28811 | 92.67925 | 95.37392 | 98.10855 | 100.604 | 102.1129 | 103.0991 |
| 39.5 | 88.4785 | 89.39733 | 90.82228 | 93.2307 | 95.94693 | 98.70568 | 101.2251 | 102.7494 | 103.746 |
| 40.5 | 88.9933 | 89.91797 | 91.35246 | 93.7784 | 96.51645 | 99.29957 | 101.8432 | 103.383 | 104.3901 |
| 41.5 | 89.50502 | 90.43559 | 91.87972 | 94.32334 | 97.08337 | 99.89104 | 102.459 | 104.0144 | 105.032 |
| 42.5 | 90.01466 | 90.95115 | 92.40497 | 94.86634 | 97.64848 | 100.4808 | 103.0732 | 104.6444 | 105.6727 |
| 43.5 | 90.52307 | 91.46549 | 92.92901 | 95.40817 | 98.21247 | 101.0696 | 103.6866 | 105.2736 | 106.3126 |
| 44.5 | 91.031 | 91.97932 | 93.45252 | 95.94946 | 98.77593 | 101.6579 | 104.2996 | 105.9025 | 106.9523 |
| 45.5 | 91.53905 | 92.49325 | 93.97609 | 96.49076 | 99.3394 | 102.2462 | 104.9128 | 106.5316 | 107.5922 |
| 46.5 | 92.04774 | 93.00778 | 94.50021 | 97.03254 | 99.90331 | 102.835 | 105.5264 | 107.1613 | 108.2328 |
| 47.5 | 92.55748 | 93.52333 | 95.02528 | 97.57519 | 100.4681 | 103.4247 | 106.141 | 107.7919 | 108.8744 |
| 48.5 | 93.06862 | 94.04022 | 95.55164 | 98.11905 | 101.0339 | 104.0154 | 106.7567 | 108.4238 | 109.5172 |
| 49.5 | 93.58141 | 94.55872 | 96.07954 | 98.66436 | 101.6012 | 104.6075 | 107.3737 | 109.057 | 110.1614 |
| 50.5 | 94.09605 | 95.07903 | 96.60918 | 99.21132 | 102.17 | 105.2012 | 107.9924 | 109.6918 | 110.8073 |
| 51.5 | 94.61267 | 95.60128 | 97.14072 | 99.76009 | 102.7406 | 105.7965 | 108.6127 | 110.3283 | 111.4548 |
| 52.5 | 95.13134 | 96.12555 | 97.67423 | 100.3108 | 103.313 | 106.3936 | 109.2347 | 110.9665 | 112.1041 |
| 53.5 | 95.65211 | 96.65189 | 98.20976 | 100.8634 | 103.8873 | 106.9925 | 109.8585 | 111.6066 | 112.7552 |
| 54.5 | 96.17495 | 97.18029 | 98.74731 | 101.418 | 104.4635 | 107.5933 | 110.4841 | 112.2483 | 113.4079 |
| 55.5 | 96.69982 | 97.71069 | 99.28686 | 101.9745 | 105.0415 | 108.1958 | 111.1114 | 112.8917 | 114.0624 |


#### Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 56.5 | 97.22663 | 98.24303 | 99.82832 | 102.5329 | 105.6213 | 108.8001 | 111.7404 | 113.5368 | 114.7184 |
| 57.5 | 97.75525 | 98.77719 | 100.3716 | 103.093 | 106.2029 | 109.406 | 112.3709 | 114.1833 | 115.3759 |
| 58.5 | 98.28555 | 99.31303 | 100.9165 | 103.6549 | 106.7861 | 110.0134 | 113.0028 | 114.8312 | 116.0347 |
| 59.5 | 98.81735 | 99.85039 | 101.463 | 104.2182 | 107.3707 | 110.6222 | 113.6359 | 115.4802 | 116.6945 |
| 60.5 | 99.35047 | 100.3891 | 102.0109 | 104.7829 | 107.9566 | 111.2321 | 114.2701 | 116.1301 | 117.3552 |
| 61.5 | 99.8847 | 100.9289 | 102.5599 | 105.3488 | 108.5436 | 111.8431 | 114.9052 | 116.7808 | 118.0166 |
| 62.5 | 100.4198 | 101.4696 | 103.1098 | 105.9156 | 109.1316 | 112.4548 | 115.5408 | 117.432 | 118.6783 |
| 63.5 | 100.9555 | 102.011 | 103.6604 | 106.4831 | 109.7202 | 113.0671 | 116.1768 | 118.0834 | 119.3402 |
| 64.5 | 101.4916 | 102.5529 | 104.2115 | 107.0512 | 110.3092 | 113.6797 | 116.813 | 118.7348 | 120.0019 |
| 65.5 | 102.0279 | 103.0948 | 104.7628 | 107.6194 | 110.8984 | 114.2923 | 117.449 | 119.3858 | 120.6632 |
| 66.5 | 102.564 | 103.6367 | 105.3141 | 108.1877 | 111.4876 | 114.9048 | 118.0845 | 120.0362 | 121.3238 |
| 67.5 | 103.0996 | 104.1782 | 105.865 | 108.7556 | 112.0764 | 115.5167 | 118.7193 | 120.6857 | 121.9832 |
| 68.5 | 103.6346 | 104.7191 | 106.4154 | 109.323 | 112.6646 | 116.1278 | 119.3531 | 121.334 | 122.6413 |
| 69.5 | 104.1685 | 105.259 | 106.9648 | 109.8895 | 113.2519 | 116.7379 | 119.9855 | 121.9807 | 123.2977 |
| 70.5 | 104.7012 | 105.7976 | 107.5131 | 110.4549 | 113.838 | 117.3466 | 120.6163 | 122.6256 | 123.9521 |
| 71.5 | 105.2323 | 106.3348 | 108.0599 | 111.0189 | 114.4226 | 117.9537 | 121.2452 | 123.2684 | 124.6042 |
| 72.5 | 105.7615 | 106.8701 | 108.605 | 111.5812 | 115.0055 | 118.5588 | 121.8718 | 123.9086 | 125.2536 |
| 73.5 | 106.2886 | 107.4033 | 109.148 | 112.1415 | 115.5863 | 119.1616 | 122.4959 | 124.5461 | 125.9 |
| 74.5 | 106.8132 | 107.9342 | 109.6888 | 112.6996 | 116.1648 | 119.7619 | 123.1171 | 125.1804 | 126.5432 |
| 75.5 | 107.3351 | 108.4624 | 110.227 | 113.255 | 116.7406 | 120.3594 | 123.7352 | 125.8114 | 127.1827 |
| 76.5 | 107.8541 | 108.9877 | 110.7623 | 113.8077 | 117.3136 | 120.9537 | 124.3499 | 126.4387 | 127.8184 |
| 77.5 | 108.3698 | 109.5099 | 111.2944 | 114.3572 | 117.8833 | 121.5447 | 124.9608 | 127.062 | 128.45 |
| 78.5 | 108.882 | 110.0285 | 111.8232 | 114.9034 | 118.4496 | 122.132 | 125.5678 | 127.6811 | 129.0771 |
| 79.5 | 109.3905 | 110.5435 | 112.3483 | 115.446 | 119.0123 | 122.7154 | 126.1705 | 128.2957 | 129.6996 |
| 80.5 | 109.8949 | 111.0545 | 112.8696 | 115.9847 | 119.571 | 123.2946 | 126.7688 | 128.9056 | 130.3171 |
| 81.5 | 110.3952 | 111.5613 | 113.3867 | 116.5193 | 120.1254 | 123.8695 | 127.3623 | 129.5105 | 130.9295 |
| 82.5 | 110.8909 | 112.0638 | 113.8995 | 117.0496 | 120.6755 | 124.4397 | 127.951 | 130.1103 | 131.5365 |
| 83.5 | 111.3821 | 112.5616 | 114.4077 | 117.5754 | 121.221 | 125.0051 | 128.5345 | 130.7047 | 132.138 |
| 84.5 | 111.8684 | 113.0546 | 114.9112 | 118.0964 | 121.7617 | 125.5655 | 129.1127 | 131.2936 | 132.7338 |
| 85.5 | 112.3496 | 113.5427 | 115.4097 | 118.6125 | 122.2974 | 126.1207 | 129.6855 | 131.8768 | 133.3238 |
| 86.5 | 112.8257 | 114.0256 | 115.9031 | 119.1235 | 122.8279 | 126.6706 | 130.2526 | 132.4542 | 133.9077 |
| 87.5 | 113.2963 | 114.5031 | 116.3913 | 119.6293 | 123.3531 | 127.215 | 130.814 | 133.0256 | 134.4857 |
| 88.5 | 113.7615 | 114.9752 | 116.874 | 120.1297 | 123.8728 | 127.7539 | 131.3696 | 133.5911 | 135.0574 |


#### Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 89.5 | 114.2211 | 115.4418 | 117.3512 | 120.6246 | 124.387 | 128.287 | 131.9194 | 134.1505 | 135.623 |
| 90.5 | 114.6749 | 115.9026 | 117.8228 | 121.1138 | 124.8956 | 128.8144 | 132.4631 | 134.7038 | 136.1824 |
| 91.5 | 115.123 | 116.3577 | 118.2886 | 121.5974 | 125.3985 | 129.3359 | 133.0009 | 135.251 | 136.7356 |
| 92.5 | 115.5651 | 116.8069 | 118.7486 | 122.0753 | 125.8956 | 129.8516 | 133.5328 | 135.7922 | 137.2826 |
| 93.5 | 116.0012 | 117.2502 | 119.2028 | 122.5473 | 126.3869 | 130.3615 | 134.0587 | 136.3273 | 137.8236 |
| 94.5 | 116.4314 | 117.6875 | 119.6511 | 123.0135 | 126.8724 | 130.8656 | 134.5787 | 136.8565 | 138.3585 |
| 95.5 | 116.8555 | 118.1189 | 120.0935 | 123.4739 | 127.3522 | 131.364 | 135.093 | 137.3798 | 138.8876 |
| 96.5 | 117.2737 | 118.5443 | 120.53 | 123.9285 | 127.8263 | 131.8567 | 135.6015 | 137.8975 | 139.411 |
| 97.5 | 117.6858 | 118.9638 | 120.9607 | 124.3774 | 128.2947 | 132.3438 | 136.1046 | 138.4097 | 139.9289 |
| 98.5 | 118.092 | 119.3774 | 121.3855 | 124.8207 | 128.7576 | 132.8255 | 136.6024 | 138.9166 | 140.4415 |
| 99.5 | 118.4924 | 119.7852 | 121.8047 | 125.2584 | 129.2152 | 133.302 | 137.095 | 139.4184 | 140.9492 |
| 100.5 | 118.8869 | 120.1873 | 122.2182 | 125.6906 | 129.6675 | 133.7734 | 137.5828 | 139.9155 | 141.4521 |
| 101.5 | 119.2757 | 120.5838 | 122.6263 | 126.1177 | 130.1148 | 134.2401 | 138.066 | 140.4082 | 141.9507 |
| 102.5 | 119.659 | 120.9748 | 123.0291 | 126.5396 | 130.5574 | 134.7023 | 138.545 | 140.8968 | 142.4454 |
| 103.5 | 120.037 | 121.3606 | 123.4268 | 126.9568 | 130.9954 | 135.1604 | 139.0201 | 141.3817 | 142.9364 |
| 104.5 | 120.4097 | 121.7413 | 123.8196 | 127.3694 | 131.4293 | 135.6146 | 139.4918 | 141.8633 | 143.4244 |
| 105.5 | 120.7775 | 122.1171 | 124.2078 | 127.7777 | 131.8593 | 136.0654 | 139.9604 | 142.3422 | 143.9098 |
| 106.5 | 121.1405 | 122.4884 | 124.5916 | 128.1822 | 132.2859 | 136.5132 | 140.4265 | 142.8188 | 144.393 |
| 107.5 | 121.4991 | 122.8555 | 124.9715 | 128.5831 | 132.7094 | 136.9585 | 140.8906 | 143.2937 | 144.8747 |
| 108.5 | 121.8537 | 123.2186 | 125.3478 | 128.9808 | 133.1304 | 137.4018 | 141.3532 | 143.7674 | 145.3555 |
| 109.5 | 122.2044 | 123.5782 | 125.7208 | 129.3759 | 133.5493 | 137.8437 | 141.8149 | 144.2406 | 145.8359 |
| 110.5 | 122.5518 | 123.9347 | 126.0911 | 129.7689 | 133.9667 | 138.2847 | 142.2764 | 144.7139 | 146.3167 |
| 111.5 | 122.8963 | 124.2885 | 126.4592 | 130.1603 | 134.3832 | 138.7256 | 142.7382 | 145.1879 | 146.7984 |
| 112.5 | 123.2384 | 124.6402 | 126.8255 | 130.5506 | 134.7995 | 139.1669 | 143.2012 | 145.6634 | 147.2818 |
| 113.5 | 123.5785 | 124.9902 | 127.1907 | 130.9406 | 135.2163 | 139.6094 | 143.666 | 146.141 | 147.7676 |
| 114.5 | 123.9173 | 125.3393 | 127.5554 | 131.3309 | 135.6342 | 140.0538 | 144.1333 | 146.6215 | 148.2564 |
| 115.5 | 124.2553 | 125.688 | 127.9203 | 131.7223 | 136.054 | 140.501 | 144.6039 | 147.1056 | 148.7491 |
| 116.5 | 124.5933 | 126.0371 | 128.2861 | 132.1156 | 136.4766 | 140.9516 | 145.0785 | 147.594 | 149.2461 |
| 117.5 | 124.932 | 126.3872 | 128.6537 | 132.5115 | 136.9027 | 141.4065 | 145.5579 | 148.0874 | 149.7484 |
| 118.5 | 125.2721 | 126.7392 | 129.0238 | 132.9109 | 137.3333 | 141.8665 | 146.0429 | 148.5865 | 150.2564 |
| 119.5 | 125.6144 | 127.094 | 129.3973 | 133.3147 | 137.7691 | 142.3324 | 146.5341 | 149.092 | 150.7707 |
| 120.5 | 125.9599 | 127.4524 | 129.7752 | 133.7239 | 138.2112 | 142.8051 | 147.0322 | 149.6044 | 151.292 |
| 121.5 | 126.3095 | 127.8154 | 130.1584 | 134.1394 | 138.6602 | 143.2852 | 147.5379 | 150.1242 | 151.8205 |


#### Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 122.5 | 126.6641 | 128 184 | 130.5479 | 134.562 | 139.1172 | 143.7735 | 148.0517 | 150.652 | 152.3568 |
| 123.5 | 127.0248 | 128.5591 | 130.9446 | 134.9929 | 139.5829 | 144.2707 | 148.5741 | 151.188 | 152.9011 |
| | 127.3926 | 128.9419 | 131.3496 | 135.4328 | 140.0581 | 144.7773 | 149.1054 | 151.7325 | 153,4534 |
| | 127.7687 | 129.3334 | 131.7639 | 135.8826 | 140.5435 | 145.2938 | 149.646 | 152.2856 | 154.0139 |
| | 128.1541 | 129.7346 | 132.1885 | 136.3433 | 141.0397 | 145.8206 | 150.196 | 152.8473 | 154.5824 |
| | 128.5499 | 130.1467 | 132.6243 | 136.8154 | 141.5472 | 146.3579 | 150.7552 | 153,4174 | 155.1586 |
| 128.5 | 128.9573 | 130.5705 | 133.0721 | 137.2997 | 142.0664 | 146.9059 | 151.3236 | 153,9955 | 155.742 |
| | 129.3772 | 131.0071 | 133.5329 | 137.7967 | 142.5974 | 147.4643 | 151.9008 | 154.5812 | 156.3321 |
| | 129.8106 | 131.4573 | 134.0072 | 138.3067 | 143.1404 | 148.0329 | 152.4861 | 155.1737 | 156.928 |
| 131.5 | 130.2585 | 131.9218 | 134.4955 | 138.83 | 143.695 | 148.6111 | 153.079 | 155.7721 | 157.5288 |
| 132.5 | 130.7217 | 132.4013 | 134.9983 | 139.3664 | 144.2609 | 149.1984 | 153.6783 | 156.3755 | 158.1335 |
| 133.5 | 131.2006 | 132.8962 | 135.5157 | 139.9157 | 144.8376 | 149.7937 | 154.283 | 156.9825 | 158.7407 |
| 134.5 | 131.6958 | 133.4067 | 136.0476 | 140.4775 | 145.424 | 150.3959 | 154.8918 | 157.5918 | 159.3491 |
| 135.5 | 132.2074 | 133.9328 | 136.5937 | 141.051 | 146.0192 | 151.0036 | 155.5032 | 158.202 | 159.9571 |
| 136.5 | 132.7354 | 134.4742 | 137.1534 | 141.6352 | 146.6217 | 151.6153 | 156.1156 | 158.8115 | 160.5633 |
| 137.5 | 133.2795 | 135.0304 | 137.7259 | 142.2288 | 147.23 | 152.2293 | 156.7273 | 159.4185 | 161.166 |
| 138.5 | 133.8388 | 135.6004 | 138.31 | 142.8304 | 147.8424 | 152.8438 | 157.3365 | 160.0213 | 161.7634 |
| 139.5 | 134.4125 | 136.1831 | 138.9043 | 143.4381 | 148.4569 | 153.4568 | 157.9413 | 160.6182 | 162.3541 |
| 140.5 | 134.9993 | 136.7769 | 139.507 | 144.0501 | 149.0714 | 154.0662 | 158.5398 | 161.2075 | 162.9363 |
| 141.5 | 135.5973 | 137.3801 | 140.1161 | 144.6641 | 149.6839 | 154.67 | 159.1302 | 161.7874 | 163.5084 |
| 142.5 | 136.2047 | 137.9905 | 140.7295 | 145.278 | 150.292 | 155.2663 | 159.7107 | 162.3564 | 164.069 |
| 143.5 | 136.8191 | 138.6058 | 141.3448 | 145.8893 | 150.8936 | 155.8529 | 160.2796 | 162.9129 | 164.6167 |
| 144.5 | 137.4381 | 139.2236 | 141.9594 | 146.4958 | 151.4866 | 156.428 | 160.8353 | 163.4555 | 165.1503 |
| 145.5 | 138.0588 | 139.841 | 142.5709 | 147.0949 | 152.0687 | 156.9899 | 161.3764 | 163.983 | 165.6685 |
| 146.5 | 138.6784 | 140.4554 | 143.1767 | 147.6845 | 152.6381 | 157.5369 | 161.9016 | 164.4943 | 166.1706 |
| 147.5 | 139.2941 | 141.064 | 143.7741 | 148.2623 | 153.193 | 158.0677 | 162.4097 | 164.9885 | 166.6555 |
| 148.5 | 139.9028 | 141.6641 | 144.3607 | 148.8263 | 153.7317 | 158.581 | 162.8999 | 165.4648 | 167.1228 |
| 149.5 | 140.5019 | 142.253 | 144.9342 | 149.3747 | 154.2529 | 159.0758 | 163.3715 | 165.9227 | 167.572 |
| 150.5 | 141.0885 | 142.8283 | 145.4925 | 149.9059 | 154.7555 | 159.5513 | 163.8239 | 166.3618 | 168.0027 |
| 151.5 | 141.6602 | 143.3877 | 146.0338 | 150.4184 | 155.2385 | 160.007 | 164.2568 | 166.7819 | 168.4147 |
| 152.5 | 142.2148 | 143.9294 | 146.5564 | 150.9113 | 155.7012 | 160.4425 | 164.6701 | 167.1829 | 168.808 |
| 153.5 | 142.7504 | 144.4516 | 147.059 | 151.3835 | 156.1432 | 160.8576 | 165.0637 | 167.5648 | 169.1827 |
| 154.5 | 143.2654 | 144.953 | 147.5405 | 151.8346 | 156.5643 | 161.2524 | 165.4378 | 167.9278 | 169.5391 |


#### Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 155.5 | 143.7584 | 145.4325 | 148.0002 | 152.2642 | 156.9644 | 161.627 | 165.7928 | 168.2723 | 169.8773 |
| 156.5 | 144.2287 | 145.8894 | 148.4376 | 152.6721 | 157.3437 | 161.9818 | 166.1289 | 168.5987 | 170.1979 |
| 157.5 | 144.6756 | 146.3232 | 148.8525 | 153.0584 | 157.7025 | 162.3172 | 166.4466 | 168.9074 | 170.5013 |
| 158.5 | 145.0987 | 146.7338 | 149.2449 | 153.4234 | 158.0411 | 162.6338 | 166.7467 | 169.199 | 170.7881 |
| 159.5 | 145.4981 | 147.1213 | 149.615 | 153.7674 | 158.3603 | 162.9321 | 167.0296 | 169.4742 | 171.0587 |
| 160.5 | 145.874 | 147.4859 | 149.9633 | 154.0911 | 158.6606 | 163.2129 | 167.2961 | 169.7335 | 171.314 |
| 161.5 | 146.2269 | 147.8281 | 150.2902 | 154.3951 | 158.9427 | 163.477 | 167.5469 | 169.9777 | 171.5544 |
| 162.5 | 146.5573 | 148.1487 | 150.5966 | 154.6801 | 159.2075 | 163.725 | 167.7826 | 170.2074 | 171.7807 |
| 163.5 | 146.866 | 148.4483 | 150.8831 | 154.947 | 159.4557 | 163.9577 | 168.0042 | 170.4234 | 171.9935 |
| 164.5 | 147.1539 | 148.7279 | 151.1507 | 155.1966 | 159.6882 | 164.1761 | 168.2122 | 170.6263 | 172.1936 |
| 165.5 | 147.4219 | 148.9885 | 151.4003 | 155.4298 | 159.9058 | 164.3808 | 168.4075 | 170.817 | 172.3816 |
| 166.5 | 147.6712 | 149.2309 | 151.6329 | 155.6475 | 160.1094 | 164.5726 | 168.5907 | 170.9959 | 172.5582 |
| 167.5 | 147.9026 | 149.4562 | 151.8494 | 155.8507 | 160.2997 | 164.7523 | 168.7626 | 171.1639 | 172.7239 |
| 168.5 | 148.1173 | 149.6655 | 152.0508 | 156.0401 | 160.4777 | 164.9206 | 168.9239 | 171.3216 | 172.8796 |
| 169.5 | 148.3164 | 149.8598 | 152.2381 | 156.2167 | 160.6441 | 165.0783 | 169.0751 | 171.4696 | 173.0257 |
| 170.5 | 148.5009 | 150.04 | 152.4121 | 156.3813 | 160.7995 | 165.226 | 169.217 | 171.6085 | 173.1628 |
| 171.5 | 148.6717 | 150.2072 | 152.5738 | 156.5348 | 160.9449 | 165.3644 | 169.3501 | 171.7388 | 173.2915 |
| 172.5 | 148.8299 | 150.3621 | 152.7241 | 156.6778 | 161.0808 | 165.4941 | 169.4749 | 171.8611 | 173.4124 |
| 173.5 | 148.9764 | 150.5059 | 152.8638 | 156.8112 | 161.2079 | 165.6157 | 169.5921 | 171.976 | 173.5258 |
| 174.5 | 149.1121 | 150.6392 | 152.9936 | 156.9356 | 161.3268 | 165.7297 | 169.7022 | 172.0839 | 173.6324 |
| 175.5 | 149.2377 | 150.7629 | 153.1143 | 157.0517 | 161.4381 | 165.8366 | 169.8055 | 172.1853 | 173.7326 |
| 176.5 | 149.3542 | 150.8777 | 153.2266 | 157.16 | 161.5423 | 165.9369 | 169.9026 | 172.2806 | 173.8267 |
| 177.5 | 149.4622 | 150.9843 | 153.3312 | 157.2612 | 161.6399 | 166.0312 | 169.9939 | 172.3701 | 173.9152 |
| 178.5 | 149.5623 | 151.0833 | 153.4286 | 157.3558 | 161.7315 | 166.1197 | 170.0798 | 172.4544 | 173.9984 |
| 179.5 | 149.6553 | 151.1754 | 153.5193 | 157.4443 | 161.8174 | 166.2029 | 170.1606 | 172.5337 | 174.0768 |
| 180.5 | 149.7416 | 151.2611 | 153.604 | 157.5271 | 161.898 | 166.2812 | 170.2366 | 172.6084 | 174.1505 |
| 181.5 | 149.8219 | 151.341 | 153.683 | 157.6047 | 161.9738 | 166.3549 | 170.3083 | 172.6787 | 174.22 |
| 182.5 | 149.8967 | 151.4154 | 153.7569 | 157.6775 | 162.045 | 166.4244 | 170.3759 | 172.7451 | 174.2855 |
| 183.5 | 149.9663 | 151.4848 | 153.826 | 157.7458 | 162.112 | 166.4898 | 170.4396 | 172.8076 | 174.3472 |
| 184.5 | 150.0312 | 151.5497 | 153.8907 | 157.8099 | 162.1752 | 166.5516 | 170.4997 | 172.8667 | 174.4055 |
| 185.5 | 150.0918 | 151.6103 | 153.9513 | 157.8702 | 162.2347 | 166.6099 | 170.5566 | 172.9225 | 174.4606 |
| 186.5 | 150.1484 | 151.6671 | 154.0082 | 157.927 | 162.2908 | 166.6649 | 170.6103 | 172.9752 | 174.5125 |
| 187.5 | 150.2014 | 151.7203 | 154.0616 | 157.9804 | 162.3439 | 166.717 | 170.6611 | 173.025 | 174.5617 |

http://www.cdc.gov/growthcharts/html charts/statage.htm/#females


#### Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 188.5 | 150.251 | 151.7702 | 154.1119 | 158.0308 | 162.394 | 166.7663 | 170.7091 | 173.0722 | 174.6082 |
| | 150.2975 | 151.8171 | 154.1592 | 158.0784 | 162.4414 | 166.8129 | 170.7546 | 173.1168 | 174.6522 |
| 190.5 | 150.3412 | 151.8612 | 154.2037 | 158.1234 | 162.4862 | 166.8571 | 170.7978 | 173.1591 | 174.6938 |
| 191.5 | 150.3823 | 151.9027 | 154.2457 | 158.1659 | 162.5287 | 166.899 | 170.8387 | 173.1992 | 174.7333 |
| 192.5 | 150.4209 | 151.9418 | 154.2854 | 158.2061 | 162.569 | 166.9388 | 170.8775 | 173.2373 | 174.7708 |
| 193.5 | 150.4573 | 151.9787 | 154.3229 | 158.2442 | 162.6072 | 166.9766 | 170.9144 | 173.2734 | 174.8063 |
| 194.5 | 150.4917 | 152.0135 | 154.3584 | 158.2803 | 162.6435 | 167.0125 | 170.9494 | 173.3077 | 174.84 |
| 195.5 | 150.5241 | 152.0465 | 154.3919 | 158.3146 | 162.6781 | 167.0466 | 170.9827 | 173.3402 | 174.8721 |
| 196.5 | 150.5547 | 152.0776 | 154.4238 | 158.3472 | 162.7109 | 167.0791 | 171.0144 | 173.3712 | 174.9025 |
| 197.5 | 150.5837 | 152.1072 | 154.454 | 158.3782 | 162.7421 | 167.11 | 171.0446 | 173.4007 | 174.9314 |
| 198.5 | 150.6111 | 152.1352 | 154.4827 | 158.4077 | 162.7719 | 167.1395 | 171.0733 | 173.4288 | 174.959 |
| 199.5 | 150.6372 | 152.1617 | 154.51 | 158.4357 | 162.8002 | 167.1676 | 171.1007 | 173.4555 | 174.9852 |
| 200.5 | 150.6619 | 152.187 | 154.5359 | 158.4625 | 162.8273 | 167.1944 | 171.1268 | 173.481 | 175.0102 |
| 201.5 | 150.6854 | 152.211 | 154.5607 | 158.4879 | 162.8531 | 167.22 | 171.1517 | 173.5053 | 175.034 |
| 202.5 | 150.7077 | 152.2339 | 154.5842 | 158.5123 | 162.8778 | 167.2444 | 171.1754 | 173.5284 | 175.0567 |
| 203.5 | 150.7289 | 152.2556 | 154.6067 | 158.5355 | 162.9013 | 167.2677 | 171.1981 | 173.5505 | 175.0783 |
| 204.5 | 150.7491 | 152.2764 | 154.6281 | 158.5577 | 162.9238 | 167.29 | 171.2198 | 173.5716 | 175.099 |
| 205.5 | 150.7684 | 152.2962 | 154.6486 | 158.5789 | 162.9454 | 167.3114 | 171.2405 | 173.5918 | 175.1187 |
| 206.5 | 150.7868 | 152.3151 | 154.6681 | 158.5992 | 162.966 | 167.3318 | 171.2604 | 173.6111 | 175.1376 |
| 207.5 | 150.8044 | 152.3332 | 154.6868 | 158.6187 | 162.9858 | 167.3514 | 171.2793 | 173.6295 | 175.1556 |
| 208.5 | 150.8211 | 152.3504 | 154.7047 | 158.6373 | 163.0047 | 167.3701 | 171.2975 | 173.6471 | 175.1728 |
| 209.5 | 150.8372 | 152.3669 | 154.7218 | 158.6551 | 163.0228 | 167.3881 | 171.3149 | 173.664 | 175.1892 |
| 210.5 | 150.8525 | 152.3827 | 154.7382 | 158.6722 | 163.0402 | 167.4053 | 171.3315 | 173.6802 | 175.205 |
| 211.5 | 150.8672 | 152.3979 | 154.754 | 158.6886 | 163.0569 | 167.4218 | 171.3475 | 173.6956 | 175.2201 |
| 212.5 | 150.8812 | 152.4124 | 154.769 | 158.7043 | 163.0729 | 167.4376 | 171.3628 | 173.7104 | 175.2345 |
| 213.5 | 150.8947 | 152.4263 | 154.7835 | 158.7194 | 163.0882 | 167.4528 | 171.3775 | 173.7246 | 175.2483 |
| 214.5 | 150.9076 | 152.4396 | 154.7974 | 158.7339 | 163.103 | 167.4674 | 171.3915 | 173.7382 | 175.2616 |
| 215.5 | 150.92 | 152.4524 | 154.8107 | 158.7478 | 163.1172 | 167.4814 | 171.405 | 173.7513 | 175.2742 |
| 216.5 | 150.9319 | 152.4647 | 154.8235 | 158.7612 | 163.1308 | 167.4948 | 171.418 | 173.7638 | 175.2864 |
| | 150.9433 | 152.4765 | 154.8358 | 158.774 | 163.1439 | 167.5078 | 171.4304 | 173.7758 | 175.2981 |
| 218.5 | 150.9542 | 152.4878 | 154.8476 | 158.7864 | 163.1565 | 167.5202 | 171.4424 | 173.7873 | 175.3093 |
| | 150.9647 | 152.4987 | 154.859 | 158.7983 | 163.1686 | 167.5321 | 171.4538 | 173.7984 | 175.32 |
| 220.5 | 150.9749 | 152.5092 | 154.8699 | 158.8097 | 163.1802 | 167.5436 | 171.4649 | 173.809 | 175.3303 |

http://www.cdc.gov/growthcharts/html charts/statage.htm/#females


**Sponsor: APEB** EudraCT number 2015-002876-25


# Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 221.5 | 150.9846 | 152.5192 | 154.8804 | 158.8207 | 163.1914 | 167.5546 | 171.4755 | 173.8192 | 175.3402 |
| 222.5 | 150.9939 | 152.5289 | 154.8905 | 158.8313 | 163.2022 | 167.5653 | 171.4856 | 173.829 | 175.3497 |
| 223.5 | 151.0029 | 152.5382 | 154.9003 | 158.8415 | 163.2126 | 167.5755 | 171.4954 | 173.8384 | 175.3588 |
| 224.5 | 151.0115 | 152.5472 | 154.9096 | 158.8514 | 163.2226 | 167.5853 | 171.5049 | 173.8474 | 175.3675 |
| 225.5 | 151.0198 | 152.5558 | 154.9187 | 158.8608 | 163.2322 | 167.5948 | 171.5139 | 173.8561 | 175.376 |
| 226.5 | 151.0279 | 152.5641 | 154.9273 | 158.8699 | 163.2415 | 167.6039 | 171.5226 | 173.8645 | 175.384 |
| 227.5 | 151.0356 | 152.5721 | 154.9357 | 158.8787 | 163.2504 | 167.6127 | 171.531 | 173.8725 | 175.3918 |
| 228.5 | 151.043 | 152.5798 | 154.9438 | 158.8872 | 163.259 | 167.6211 | 171.5391 | 173.8802 | 175.3993 |
| 229.5 | 151.0501 | 152.5873 | 154.9516 | 158.8953 | 163.2673 | 167.6293 | 171.5468 | 173.8877 | 175.4064 |
| 230.5 | 151.057 | 152.5944 | 154.959 | 158.9032 | 163.2753 | 167.6371 | 171.5543 | 173.8948 | 175.4133 |
| 231.5 | 151.0636 | 152.6013 | 154.9663 | 158.9107 | 163.283 | 167.6446 | 171.5615 | 173.9017 | 175.42 |
| 232.5 | 151.07 | 152.6079 | 154.9732 | 158.918 | 163.2904 | 167.6519 | 171.5684 | 173.9083 | 175.4264 |
| 233.5 | 151.0762 | 152.6143 | 154.9799 | 158.9251 | 163.2976 | 167.6589 | 171.5751 | 173.9147 | 175.4325 |
| 234.5 | 151.0821 | 152.6205 | 154.9864 | 158.9319 | 163.3045 | 167.6657 | 171.5815 | 173.9208 | 175.4384 |
| 235.5 | 151.0879 | 152.6265 | 154.9926 | 158.9384 | 163.3111 | 167.6722 | 171.5877 | 173.9267 | 175.4441 |
| 236.5 | 151.0934 | 152.6322 | 154.9986 | 158.9447 | 163.3175 | 167.6785 | 171.5937 | 173.9324 | 175.4496 |
| 237.5 | 151.0987 | 152.6377 | 155.0044 | 158.9508 | 163.3237 | 167.6845 | 171.5994 | 173.9379 | 175.4548 |
| 238.5 | 151.1038 | 152.6431 | 155.01 | 158.9567 | 163.3297 | 167.6904 | 171.6049 | 173.9432 | 175.4599 |
| 239.5 | 151.1088 | 152.6482 | 155.0154 | 158.9624 | 163.3354 | 167.696 | 171.6103 | 173.9482 | 175.4648 |
| 240 | 151.1112 | 152.6507 | 155.0181 | 158.9651 | 163.3383 | 167.6987 | 171.6129 | 173.9507 | 175.4671 |

http://www.cdc.gov/growthcharts/html charts/statage.htm/#females


# 12.12 Blood Pressure Levels for Boys by Age and Height Percentile [NIH 2005]

# Blood Pressure Levels for Boys by Age and Height Percentile

| | BP | | | Systo | lic BP ( | mmHg) | | | | | Diasto | lic BP | (mmHg | ) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | | + | Perce | ntile of | Height | <b>→</b> | | | + | Perce | ntile of | Height | <b>→</b> | |
| (Year) | 4 | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 1 | 50th | 80 | 81 | 83 | 85 | 87 | 88 | 89 | 34 | 35 | 36 | 37 | 38 | 39 | 39 |
| | 90th | 94 | 95 | 97 | 99 | 100 | 102 | 103 | 49 | 50 | 51 | 52 | 53 | 53 | 54 |
| | 95th | 98 | 99 | 101 | 103 | 104 | 106 | 106 | 54 | 54 | 55 | 56 | 57 | 58 | 58 |
| | 99th | 105 | 106 | 108 | 110 | 112 | 113 | 114 | 61 | 62 | 63 | 64 | 65 | 66 | 66 |
| 2 | 50th | 84 | 85 | 87 | 88 | 90 | 92 | 92 | 39 | 40 | 41 | 42 | 43 | 44 | 44 |
| | 90th | 97 | 99 | 100 | 102 | 104 | 105 | 106 | 54 | 55 | 56 | 57 | 58 | 58 | 59 |
| | 95th | 101 | 102 | 104 | 106 | 108 | 109 | 110 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 99th | 109 | 110 | 111 | 113 | 115 | 117 | 117 | 66 | 67 | 68 | 69 | 70 | 71 | 71 |
| 3 | 50th | 86 | 87 | 89 | 91 | 93 | 94 | 95 | 44 | 44 | 45 | 46 | 47 | 48 | 48 |
| | 90th | 100 | 101 | 103 | 105 | 107 | 108 | 109 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 95th | 104 | 105 | 107 | 109 | 110 | 112 | 113 | 63 | 63 | 64 | 65 | 66 | 67 | 67 |
| | 99th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 71 | 71 | 72 | 73 | 74 | 75 | 75 |
| 4 | 50th | 88 | 89 | 91 | 93 | 95 | 96 | 97 | 47 | 48 | 49 | 50 | 51 | 51 | 52 |
| | 90th | 102 | 103 | 105 | 107 | 109 | 110 | 111 | 62 | 63 | 64 | 65 | 66 | 66 | 67 |
| | 95th | 106 | 107 | 109 | 111 | 112 | 114 | 115 | 66 | 67 | 68 | 69 | 70 | 71 | 71 |
| | 99th | 113 | 114 | 116 | 118 | 120 | 121 | 122 | 74 | 75 | 76 | 77 | 78 | 78 | 79 |
| 5 | 50th | 90 | 91 | 93 | 95 | 96 | 98 | 98 | 50 | 51 | 52 | 53 | 54 | 55 | 55 |
| | 90th | 104 | 105 | 106 | 108 | 110 | 111 | 112 | 65 | 66 | 67 | 68 | 69 | 69 | 70 |
| | 95th | 108 | 109 | 110 | 112 | 114 | 115 | 116 | 69 | 70 | 71 | 72 | 73 | 74 | 74 |
| | 99th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 77 | 78 | 79 | 80 | 81 | 81 | 82 |
| 6 | 50th | 91 | 92 | 94 | 96 | 98 | 99 | 100 | 53 | 53 | 54 | 55 | 56 | 57 | 57 |
| | 90th | 105 | 106 | 108 | 110 | 111 | 113 | 113 | 68 | 68 | 69 | 70 | 71 | 72 | 72 |
| | 95th | 109 | 110 | 112 | 114 | 115 | 117 | 117 | 72 | 72 | 73 | 74 | 75 | 76 | 76 |
| | 99th | 116 | 117 | 119 | 121 | 123 | 124 | 125 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| 7 | 50th | 92 | 94 | 95 | 97 | 99 | 100 | 101 | 55 | 55 | 56 | 57 | 58 | 59 | 59 |
| | 90th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 70 | 70 | 71 | 72 | 73 | 74 | 74 |
| | 95th | 110 | 111 | 113 | 115 | 117 | 118 | 119 | 74 | 74 | 75 | 76 | 77 | 78 | 78 |
| | 99th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 82 | 82 | 83 | 84 | 85 | 86 | 86 |
| 8 | 50th | 94 | 95 | 97 | 99 | 100 | 102 | 102 | 56 | 57 | 58 | 59 | 60 | 60 | 61 |
| 1070 | 90th | 107 | 109 | 110 | 112 | 114 | 115 | 116 | 71 | 72 | 72 | 73 | 74 | 75 | 76 |
| | 95th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 99th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 83 | 84 | 85 | 86 | 87 | 87 | 88 |
| 9 | 50th | 95 | 96 | 98 | 100 | 102 | 103 | 104 | 57 | 58 | 59 | 60 | 61 | 61 | 62 |
| | 90th | 109 | 110 | 112 | 114 | 115 | 117 | 118 | 72 | 73 | 74 | 75 | 76 | 76 | 77 |
| | 95th | 113 | 114 | 116 | 118 | 119 | 121 | 121 | 76 | 77 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 120 | 121 | 123 | 125 | 127 | 128 | 129 | 84 | 85 | 86 | 87 | 88 | 88 | 89 |
| 10 | 50th | 97 | 98 | 100 | 102 | 103 | 105 | 106 | 58 | 59 | 60 | 61 | 61 | 62 | 63 |
| | 90th | 111 | 112 | 114 | 115 | 117 | 119 | 119 | 73 | 73 | 74 | 75 | 76 | 77 | 78 |
| | 95th | 115 | 116 | 117 | 119 | 121 | 122 | 123 | 77 | 78 | 79 | 80 | 81 | 81 | 82 |
| | 99th | 122 | 123 | 125 | 127 | 128 | 130 | 130 | 85 | 86 | 86 | 88 | 88 | 89 | 90 |

EudraCT number 2015-002876-25


## Blood Pressure Levels for Boys by Age and Height Percentile (Continued)

| | ВР | | | Systo | lic BP ( | mmHg) | r. | | | | Diasto | lic BP | (mmHg | ) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | | + | • Perce | ntile of | Height | <b>→</b> | | | + | Perce | ntile of | Height | 90th 95th 63 63 78 78 82 82 90 90 63 64 78 79 82 83 90 91 64 64 79 79 83 83 91 91 65 65 79 80 84 84 92 92 66 66 80 81 85 85 93 93 67 67 82 82 86 87 94 94 69 70 84 84 88 88 | |
| (Year) | 4 | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 11 | 50th | 99 | 100 | 102 | 104 | 105 | 107 | 107 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 90th | 113 | 114 | 115 | 117 | 119 | 120 | 121 | 74 | 74 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 117 | 118 | 119 | 121 | 123 | 124 | 125 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 124 | 125 | 127 | 129 | 130 | 132 | 132 | 86 | 86 | 87 | 88 | 89 | 90 | 90 |
| 12 | 50th | 101 | 102 | 104 | 106 | 108 | 109 | 110 | 59 | 60 | 61 | 62 | 63 | 63 | 64 |
| | 90th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 74 | 75 | 75 | 76 | 77 | 78 | 79 |
| | 95th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 78 | 79 | 80 | 81 | 82 | 82 | 83 |
| | 99th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 86 | 87 | 88 | 89 | 90 | 90 | 91 |
| 13 | 50th | 104 | 105 | 106 | 108 | 110 | 111 | 112 | 60 | 60 | 61 | 62 | 63 | 64 | 64 |
| | 90th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 75 | 75 | 76 | 77 | 78 | 79 | 79 |
| | 95th | 121 | 122 | 124 | 126 | 128 | 129 | 130 | 79 | 79 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 130 | 131 | 133 | 135 | 136 | 137 | 87 | 87 | 88 | 89 | 90 | 91 | 91 |
| 14 | 50th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 60 | 61 | 62 | 63 | 64 | 65 | 65 |
| | 90th | 120 | 121 | 123 | 125 | 126 | 128 | 128 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 95th | 124 | 125 | 127 | 128 | 130 | 132 | 132 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 131 | 132 | 134 | 136 | 138 | 139 | 140 | 87 | 88 | 89 | 90 | 91 | 92 | 92 |
| 15 | 50th | 109 | 110 | 112 | 113 | 115 | 117 | 117 | 61 | 62 | 63 | 64 | 65 | 66 | 66 |
| | 90th | 122 | 124 | 125 | 127 | 129 | 130 | 131 | 76 | 77 | 78 | 79 | 80 | 80 | 81 |
| | 95th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 81 | 81 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 134 | 135 | 136 | 138 | 140 | 142 | 142 | 88 | 89 | 90 | 91 | 92 | 93 | 93 |
| 16 | 50th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 63 | 63 | 64 | 65 | 66 | 67 | 67 |
| | 90th | 125 | 126 | 128 | 130 | 131 | 133 | 134 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 95th | 129 | 130 | 132 | 134 | 135 | 137 | 137 | 82 | 83 | 83 | 84 | 85 | 86 | 87 |
| | 99th | 136 | 137 | 139 | 141 | 143 | 144 | 145 | 90 | 90 | 91 | 92 | 93 | 94 | 94 |
| 17 | 50th | 114 | 115 | 116 | 118 | 120 | 121 | 122 | 65 | 66 | 66 | 67 | 68 | 69 | 70 |
| | 90th | 127 | 128 | 130 | 132 | 134 | 135 | 136 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 95th | 131 | 132 | 134 | 136 | 138 | 139 | 140 | 84 | 85 | 86 | 87 | 87 | 88 | 89 |
| | 99th | 139 | 140 | 141 | 143 | 145 | 146 | 147 | 92 | 93 | 93 | 94 | 95 | 96 | 97 |

BP, blood pressure

For research purposes, the standard deviations in Appendix Table B–1 allow one to compute BP Z-scores and percentiles for boys with height percentiles given in Table 3 (i.e., the 5th,10th, 25th, 50th, 75th, 90th, and 95th percentiles). These height percentiles must be converted to height Z-scores given by (5% = -1.645; 10% = -1.28; 25% = -0.68; 50% = 0; 75% = 0.68; 90% = 1.28%; 95% = 1.645) and then computed according to the methodology in steps 2–4 described in Appendix B. For children with height percentiles other than these, follow steps 1–4 as described in Appendix B.

<sup>\*</sup> The 90th percentile is 1.28 SD, 95th percentile is 1.645 SD, and the 99th percentile is 2.326 SD over the mean.


# 12.13 Blood Pressure Levels for Girls by Age and Height Percentile [NIH 2005]

# Blood Pressure Levels for Girls by Age and Height Percentile

| | BP | | | Systo | lic BP ( | mmHg) | | | | | Diasto | lic BP ( | mmHg | ) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | | + | Perce | ntile of | Height | <b>→</b> | | | + | Perce | ntile of | Height | <b>→</b> | |
| (Year) | 4 | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| ı | 50th | 83 | 84 | 85 | 86 | 88 | 89 | 90 | 38 | 39 | 39 | 40 | 41 | 41 | 42 |
| | 90th | 97 | 97 | 98 | 100 | 101 | 102 | 103 | 52 | 53 | 53 | 54 | 55 | 55 | 56 |
| | 95th | 100 | 101 | 102 | 104 | 105 | 106 | 107 | 56 | 57 | 57 | 58 | 59 | 59 | 60 |
| | 99th | 108 | 108 | 109 | 111 | 112 | 113 | 114 | 64 | 64 | 65 | 65 | 66 | 67 | 67 |
| 2 | 50th | 85 | 85 | 87 | 88 | 89 | 91 | 91 | 43 | 44 | 44 | 45 | 46 | 46 | 47 |
| | 90th | 98 | 99 | 100 | 101 | 103 | 104 | 105 | 57 | 58 | 58 | 59 | 60 | 61 | 61 |
| | 95th | 102 | 103 | 104 | 105 | 107 | 108 | 109 | 61 | 62 | 62 | 63 | 64 | 65 | 65 |
| | 99th | 109 | 110 | 111 | 112 | 114 | 115 | 116 | 69 | 69 | 70 | 70 | 71 | 72 | 72 |
| 3 | 50th | 86 | 87 | 88 | 89 | 91 | 92 | 93 | 47 | 48 | 48 | 49 | 50 | 50 | 51 |
| | 90th | 100 | 100 | 102 | 103 | 104 | 106 | 106 | 61 | 62 | 62 | 63 | 64 | 64 | 65 |
| | 95th | 104 | 104 | 105 | 107 | 108 | 109 | 110 | 65 | 66 | 66 | 67 | 68 | 68 | 69 |
| | 99th | 111 | 111 | 113 | 114 | 115 | 116 | 117 | 73 | 73 | 74 | 74 | 75 | 76 | 76 |
| 4 | 50th | 88 | 88 | 90 | 91 | 92 | 94 | 94 | 50 | 50 | 51 | 52 | 52 | 53 | 54 |
| | 90th | 101 | 102 | 103 | 104 | 106 | 107 | 108 | 64 | 64 | 65 | 66 | 67 | 67 | 68 |
| | 95th | 105 | 106 | 107 | 108 | 110 | 111 | 112 | 68 | 68 | 69 | 70 | 71 | 71 | 72 |
| | 99th | 112 | 113 | 114 | 115 | 117 | 118 | 119 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| 5 | 50th | 89 | 90 | 91 | 93 | 94 | 95 | 96 | 52 | 53 | 53 | 54 | 55 | 55 | 56 |
| | 90th | 103 | 103 | 105 | 106 | 107 | 109 | 109 | 66 | 67 | 67 | 68 | 69 | 69 | 70 |
| | 95th | 107 | 107 | 108 | 110 | 111 | 112 | 113 | 70 | 71 | 71 | 72 | 73 | 73 | 74 |
| | 99th | 114 | 114 | 116 | 117 | 118 | 120 | 120 | 78 | 78 | 79 | 79 | 80 | 81 | 81 |
| 6 | 50th | 91 | 92 | 93 | 94 | 96 | 97 | 98 | 54 | 54 | 55 | 56 | 56 | 57 | 58 |
| 1050 | 90th | 104 | 105 | 106 | 108 | 109 | 110 | 111 | 68 | 68 | 69 | 70 | 70 | 71 | 72 |
| | 95th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 72 | 72 | 73 | 74 | 74 | 75 | 76 |
| | 99th | 115 | 116 | 117 | 119 | 120 | 121 | 122 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| 7 | 50th | 93 | 93 | 95 | 96 | 97 | 99 | 99 | 55 | 56 | 56 | 57 | 58 | 58 | 59 |
| | 90th | 106 | 107 | 108 | 109 | 111 | 112 | 113 | 69 | 70 | 70 | 71 | 72 | 72 | 73 |
| | 95th | 110 | 111 | 112 | 113 | 115 | 116 | 116 | 73 | 74 | 74 | 75 | 76 | 76 | 77 |
| | 99th | 117 | 118 | 119 | 120 | 122 | 123 | 124 | 81 | 81 | 82 | 82 | 83 | 84 | 84 |
| 8 | 50th | 95 | 95 | 96 | 98 | 99 | 100 | 101 | 57 | 57 | 57 | 58 | 59 | 60 | 60 |
| | 90th | 108 | 109 | 110 | 111 | 113 | 114 | 114 | 71 | 71 | 71 | 72 | 73 | 74 | 74 |
| | 95th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 99th | 119 | 120 | 121 | 122 | 123 | 125 | 125 | 82 | 82 | 83 | 83 | 84 | 85 | 86 |
| 9 | 50th | 96 | 97 | 98 | 100 | 101 | 102 | 103 | 58 | 58 | 58 | 59 | 60 | 61 | 61 |
| | 90th | 110 | 110 | 112 | 113 | 114 | 116 | 116 | 72 | 72 | 72 | 73 | 74 | 75 | 75 |
| | 95th | 114 | 114 | 115 | 117 | 118 | 119 | 120 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| | 99th | 121 | 121 | 123 | 124 | 125 | 127 | 127 | 83 | 83 | 84 | 84 | 85 | 86 | 87 |
| 10 | 50th | 98 | 99 | 100 | 102 | 103 | 104 | 105 | 59 | 59 | 59 | 60 | 61 | 62 | 62 |
| | 90th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 73 | 73 | 73 | 74 | 75 | 76 | 76 |
| | 95th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 99th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 84 | 84 | 85 | 86 | 86 | 87 | 88 |

EudraCT number 2015-002876-25


## Blood Pressure Levels for Girls by Age and Height Percentile (Continued)

| | BP | | | Systo | lic BP ( | mmHg) | | | | | Diasto | lic BP | (mmHg) | ) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | | + | Perce | ntile of | Height | <b>→</b> | | 300 | + | Perce | ntile of | Height | <b>→</b> | |
| (Year) | 4 | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 11 | 50th | 100 | 101 | 102 | 103 | 105 | 106 | 107 | 60 | 60 | 60 | 61 | 62 | 63 | 63 |
| | 90th | 114 | 114 | 116 | 117 | 118 | 119 | 120 | 74 | 74 | 74 | 75 | 76 | 77 | 77 |
| | 95th | 118 | 118 | 119 | 121 | 122 | 123 | 124 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 125 | 125 | 126 | 128 | 129 | 130 | 131 | 85 | 85 | 86 | 87 | 87 | 88 | 89 |
| 12 | 50th | 102 | 103 | 104 | 105 | 107 | 108 | 109 | 61 | 61 | 61 | 62 | 63 | 64 | 64 |
| | 90th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 119 | 120 | 121 | 123 | 124 | 125 | 126 | 79 | 79 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 127 | 127 | 128 | 130 | 131 | 132 | 133 | 86 | 86 | 87 | 88 | 88 | 89 | 90 |
| 13 | 50th | 104 | 105 | 106 | 107 | 109 | 110 | 110 | 62 | 62 | 62 | 63 | 64 | 65 | 65 |
| | 90th | 117 | 118 | 119 | 121 | 122 | 123 | 124 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| | 95th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 129 | 130 | 132 | 133 | 134 | 135 | 87 | 87 | 88 | 89 | 89 | 90 | 91 |
| 14 | 50th | 106 | 106 | 107 | 109 | 110 | 111 | 112 | 63 | 63 | 63 | 64 | 65 | 66 | 66 |
| | 90th | 119 | 120 | 121 | 122 | 124 | 125 | 125 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 95th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 81 | 81 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 130 | 131 | 132 | 133 | 135 | 136 | 136 | 88 | 88 | 89 | 90 | 90 | 91 | 92 |
| 15 | 50th | 107 | 108 | 109 | 110 | 111 | 113 | 113 | 64 | 64 | 64 | 65 | 66 | 67 | 67 |
| | 90th | 120 | 121 | 122 | 123 | 125 | 126 | 127 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 95th | 124 | 125 | 126 | 127 | 129 | 130 | 131 | 82 | 82 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 131 | 132 | 133 | 134 | 136 | 137 | 138 | 89 | 89 | 90 | 91 | 91 | 92 | 93 |
| 16 | 50th | 108 | 108 | 110 | 111 | 112 | 114 | 114 | 64 | 64 | 65 | 66 | 66 | 67 | 68 |
| | 90th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 78 | 78 | 79 | 80 | 81 | 81 | 82 |
| | 95th | 125 | 126 | 127 | 128 | 130 | 131 | 132 | 82 | 82 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 132 | 133 | 134 | 135 | 137 | 138 | 139 | 90 | 90 | 90 | 91 | 92 | 93 | 93 |
| 17 | 50th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 64 | 65 | 65 | 66 | 67 | 67 | 68 |
| | 90th | 122 | 122 | 123 | 125 | 126 | 127 | 128 | 78 | 79 | 79 | 80 | 81 | 81 | 82 |
| | 95th | 125 | 126 | 127 | 129 | 130 | 131 | 132 | 82 | 83 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 133 | 133 | 134 | 136 | 137 | 138 | 139 | 90 | 90 | 91 | 91 | 92 | 93 | 93 |

BP, blood pressure

For research purposes, the standard deviations in Appendix Table B–1 allow one to compute BP Z-scores and percentiles for girls with height percentiles given in Table 4 (i.e., the 5th,10th, 25th, 50th, 75th, 90th, and 95th percentiles). These height percentiles must be converted to height Z-scores given by (5% = -1.645; 10% = -1.28; 25% = -0.68; 50% = 0; 75% = 0.68; 90% = 1.28%; 95% = 1.645) and then computed according to the methodology in steps 2–4 described in Appendix B. For children with height percentiles other than these, follow steps 1–4 as described in Appendix B.

<sup>\*</sup> The 90th percentile is 1.28 SD, 95th percentile is 1.645 SD, and the 99th percentile is 2.326 SD over the mean.

EudraCT number 2015-002876-25


## 13 ATTACHMENT 1: SUBSTANTIAL AMENDMENT 1

## I. The purpose of this amendment is:

## **Substantial Changes**

## 1. Add Mirabegron Oral Suspension as a Formulation of the Study Drug

## **DESCRIPTION OF CHANGE:**

Mirabegron oral suspension (8 mg/mL) is added to the protocol as a second study drug formulation.

#### RATIONALE:

As part of the pediatric mirabegron development program, a suspension formulation of the study drug has been developed. This is to ensure availability of an appropriate formulation for smaller children or children who have difficulties with swallowing tablets. This formulation is now available to be included into the study.

## 2. Update of Inclusion Criterion 3

## DESCRIPTION OF CHANGE:

The lower weight range for inclusion of subjects in the study is updated to  $\geq 11$  kg.

## **RATIONALE:**

Due to the addition of mirabegron oral suspension to the protocol, subjects below 35 kg can now be included. Based on the dose prediction performed, the minimum body weight for inclusion of subjects in the study is updated to 11 kg.

## 3. Update of the Age Range for the Study Population

## **DESCRIPTION OF CHANGE:**

The age range for the study population to enter the study is updated to male and female children from 3 to less than 18 years of age.

## RATIONALE:

This study is targeted to fulfill both the EMA and FDA requirements related to the conduct of pediatric trials. A "Written Request" received from the FDA includes a stipulation to decrease the lower limit of the age range from 5 to 3 years of age. Therefore, in order to ensure that the current study meets the needs of both the FDA and the EMA, the age range is adjusted.

Lowering the age range from 5 to 3 years is possible because dose predictions in this study cover doses from a body weight of 11 kg onwards. The cut-off of 11 kg body weight is considered appropriate for the age range of 3 to less than 18 years old.

EudraCT number 2015-002876-25


## 4. Add Extra Self Blood Pressure Measurements

## **DESCRIPTION OF CHANGE:**

Extra Self Blood Pressure Measurements (SBPM) are included at week 1 and 2 after the start of dosing and after a dose escalation.

## RATIONALE:

The EMA and FDA requested additional blood pressure measurements to be performed. This change implements additional SBPM done around 1 and 2 weeks after start of mirabegron (PED25) treatment and after up-titration from PED25 to PED50 (if not already covered by the scheduled SBPM). Triplicate home measurements will be taken in the morning and in the evening.

## **Non-Substantial Changes**

## 1. Remove IND Number on Cover Page

The IND number on the cover page of the protocol is removed.

## RATIONALE:

The study is not conducted under IND. The IND reference number was cited on the cover page of the protocol in error.

## 2. Update Available Clinical Data

## **DESCRIPTION OF CHANGE:**

Preliminary data of ongoing studies 178-CL-203 and 178-CL-208 are included in the protocol. Data from completed study 178-CL-202 are moved to the Investigator's Brochure.

## RATIONALE:

After the finalization of the protocol new data from mirabegron studies within the pediatric program has become available. This preliminary data has now been included in the introduction of the protocol to support dosing in children/adolescents with a body weight < 35 kg. Since the protocol was finalized, the final clinical study report for Study 178-CL-202 has become available and so this information has been removed from the protocol and has been incorporated in the Investigator's Brochure.

## 3. Update Mirabegron Approval Information

#### DESCRIPTION OF CHANGE

The number of countries that Mirabegron has been approved in is updated.

#### RATIONALE:

EudraCT number 2015-002876-25


The pediatric Investigator's Brochure has been updated and this change makes the two documents consistent.

## 4. Remove SMIP Measurement as a Dose Titration Criteria

#### DESCRIPTION OF CHANGE:

The Self Measurement of Intravesical Pressure (SMIP) is removed from the dose titration criteria.

## RATIONALE:

The SMIP was intended to be included as a safety parameter to assess the intravesical pressure in an at-home situation. In the FDA Advice Letter the Sponsor was asked to exclude the results of SMIP as a basis for dose titration in this study.

## 5. Correct Exploratory Efficacy Endpoints

## DESCRIPTION OF CHANGE:

For the e-Diary, the maximum confirmed daytime dry period is removed as an exploratory endpoint and for the endpoints on total catheterized volume an explanation is included on how catheterizations are assigned to a certain period of the day.

## RATIONALE:

The maximum confirmed daytime dry period and the maximum confirmed dry daytime period/7 days were included to take into account the intervals between the catheterizations. It was deleted to reduce the number of exploratory parameters.

To ensure a correct assignment of the catheterization times to daytime and/or night-time, a clarification is included to explain that the first morning catheterization after waking up is regarded as part of the 'night', whilst the last evening catheterization before sleep time is part of the 'day'.

## 6. Include Missing Variable for Bladder Diary

#### DESCRIPTION OF CHANGE:

The number of leakages between CICs is included in the sections on collected Patient Reported Outcome data in the protocol.

## RATIONALE:

The number of leakages between CICs is used in the calculation of secondary and exploratory endpoints. The collection of this variable is included in the eDiary and its' submitted documentation, but was not correctly specified as a collected variable in the protocol.

EudraCT number 2015-002876-25


## 7. Include Preferred Method for Clinic Vital Signs Measurements

## **DESCRIPTION OF CHANGE:**

Auscultation is included in the protocol as the preferred method for measuring vital signs in the clinic.

#### RATIONALE:

The Fourth Report on the Diagnosis, Evaluation, and Treatment of High Blood Pressure in Children and Adolescents, which is used as the basis for the blood pressure percentiles used in this study states that "The BP tables are bases on auscultatory measurements, therefore the preferred measurement is auscultation" †.

This method has been included in the protocol as the preferred method for measuring vital signs.

† The Fourth Report on the Diagnosis, Evaluation, and Treatment of High Blood Pressure in Children and Adolescents. U.S. Department of Health and Human Services, National Institutes of Health National Heart, Lung, and Blood Institute. NIH Publication No. 05-5267 Originally printed September 1996 (96-3790) Revised May 2005

## 8. Add Conversion Factor for Urine Weight-to-Volume

## **DESCRIPTION OF CHANGE:**

A gram-to-milliliter conversion factor is included in the protocol to calculate urine volume based on the subject's reported urine weight in the eDiary.

## RATIONALE:

The protocol did not include the conversion factor to calculate the urine volume based on the urine weight that is reported by the subject in the eDiary.

## 9. Add eGFR Parameters

## **DESCRIPTION OF CHANGE:**

Two additional eGFR parameters are included for reporting in the Clinical Study Report. For subjects from 3 to 12 years of age, the modified Schwartz formula (2009) is added and for subjects from 12 to 18 years of age, the Cockcroft-Gault equation.

#### RATIONALE:

The calculation of eGFR according to both the modified Schwartz formula and the Cockcroft-Gault Equation will be summarized in line with a request form the FDA. No additional assessment or increase in collected blood volume is required. Both parameters will be derived based on already collected biochemistry results.

EudraCT number 2015-002876-25


## 10. Amend Text for Start of Adverse Event Collection

## **DESCRIPTION OF CHANGE:**

The text on the start of adverse event collection is updated to avoid any misunderstanding.

## RATIONALE:

The current text in the protocol was ambiguous, possibly leading to confusion on when the collection of AEs start. The sentence has been re-worded to provide clarity.

## 11. Correct Text for Safety Reporting

## **DESCRIPTION OF CHANGE:**

The text related to the safety reporting timeline between the CRO and the Sponsor is updated from 24 hours, to 1 working day.

#### RATIONALE:

In line with ICH-GCP E6, chapter 5.2, Astellas has outsourced the safety reporting process for sites to the CRO

. The ultimate responsibility for safety reporting will remain with the Sponsor, as will be the responsibility for adhering to the reporting timelines according to section 5.1.5 of the EU guideline "Detailed guidance on the collection, verification and presentation of adverse event/reaction reports arising from clinical trials on medicinal products for human use" (CT3). Instead of a reporting timeline of 1 working day between receipt of the SAE worksheet at the CRO and forwarding of this worksheet to the Sponsor, the protocol listed a 24 hour reporting timeline. This has been corrected.

For the Sponsor's reporting obligations, the clock starts at the time the CRO has first knowledge of the minimum criteria for expedited reporting. This correction will not affect the regulatory reporting timelines.

## 12. Add SAE Reporting Procedure after End of Treatment

## **DESCRIPTION OF CHANGE:**

Timelines for SAE reporting after End of Study are included in the protocol.

## RATIONALE:

The protocol did not mention the cut-off timelines for reporting of new SAEs occurring after the End of Study visit. This timeline is 28 days and the information has now been included into the protocol.

## 13. Amend Text for Pharmacokinetic Sampling Times

## DESCRIPTION OF CHANGE:

The preferred timing of pharmacokinetic sampling is added to the protocol.

#### RATIONALE:

To allow for an early assessment of the dose-response relationship by the Data Safety

EudraCT number 2015-002876-25


Monitoring Board (DSMB), it is preferred the pharmacokinetic sampling takes place as early in the study as possible.

## 14. Addition of Subgroup Analyses

## **DESCRIPTION OF CHANGE:**

Subgroup analyses for selected safety parameters are added to the statistical section of the protocol.

## RATIONALE:

Subgroup analyses related to formulation (tablet or suspension) and dosing regimen (PED25 or PED50) for selected safety parameters have been added to further characterize the safety profile.

## 15. Administrative-type Changes

## DESCRIPTION OF CHANGE:

Various edits related to consistency, formatting and numbering are made throughout the protocol.

#### RATIONALE:

To provide clarification to the protocol and to ensure complete understanding of the study procedures.

#### II. Amendment Summary of Changes: Substantial

# Cover Page, 2 Investigator's Signature and IV Synopsis, Title of Study and Study Population

## WAS:

An Open-label, Baseline-controlled, Multicenter, Phase 3 Dose-titration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents From 5 to Less Than 18 Years of Age With Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)

## IS AMENDED TO:

An Open-label, Baseline-controlled, Multicenter, Phase 3 Dose-titration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents From 5 3 to Less Than 18 Years of Age \(\frac{\text{W}}{\text{w}}\)ith Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)

# IV Synopsis, Number of Subjects to be Enrolled/Randomized and 2 Study Objectives(s), Design, and Endpoints

2.2.1 Study Design

EudraCT number 2015-002876-25


#### WAS:

At least 44 evaluable subjects (estimate 63 enrolled), with at least 10 subjects from each age group (children aged 5 to less than 12 years of age; adolescents aged 12 to less than 18 years of age) are planned. A subject is considered being evaluable if the subject has a nonmissing maximum cystometric capacity (MCC) measurement at baseline and at a postbaseline visit.

## IS AMENDED TO:

At least 44 evaluable subjects (estimate 63 enrolled), with at least 10 subjects from each age group (children aged 5 3 to less than 12 years of age; adolescents aged 12 to less than 18 years of age) are planned. A subject is considered being evaluable if the subject has a valid (as by the central reviewer's assessment) nonmissing maximum cystometric capacity (MCC) measurement at baseline and at a postbaseline visit.

# IV Synopsis, Inclusion/Exclusion Criteria, 2 Study Objectives(s), Design, and Endpoints, 3 Study Population and 8 Operational and Administrative Considerations

2.2.1 Study Design, 3.1 Selection of Study Population, 3.2 Inclusion Criteria and 8.2.3.1 Subject Information and Consent

## WAS:

2. Subject is male or female from 5 to less than 18 years of age.

#### IS AMENDED TO:

2. Subject is male or female from 5 3 to less than 18 years of age.

# IV Synopsis, Inclusion/Exclusion Criteria and 3 Inclusion/Exclusion Criteria

3.2 Inclusion Criteria

## WAS:

3. Subject has a body weight of  $\geq$  35 kg.

## IS AMENDED TO:

3. Subject has a body weight of  $\geq 3511$  kg.

## IV Synopsis, Investigational Product(s)

## WAS:

## **Investigational Product(s):**

Mirabegron tablets, strengths 25 mg and 50 mg

#### Dose(s):

The initial dose will be PED25. The dose may be up-titrated to PED50 according to the dose-titration criteria.

#### **Mode of Administration:**

Study drug will be taken orally, once a day in the morning around the same time of day and around time of food intake (i.e., within 1 hour before or after breakfast). Tablet to be taken with a sip of water (tablet should be taken as a whole and should not be chewed, divided or

EudraCT number 2015-002876-25


#### crushed).

On visit days where a pharmacokinetic sample is planned in the clinic, completion of breakfast and study drug dosing should occur in the clinic.

## IS AMENDED TO:

## **Investigational Product(s):**

Mirabegron prolonged-release tablets, strengths 25 mg and 50 mg

Mirabegron oral suspension, strength 8 mg/mL

#### Dose(s):

The initial dose will be PED25. The dose may be up titrated to PED50 according to the dose titration criteria.

## **Selection of the formulation:**

Subjects with a body weight < 35 kg: mirabegron oral suspension.

Subjects with a body weight  $\geq$  35 kg: mirabegron tablets.

## **Selection of the dose:**

Doses are calculated weight-based. The bodyweight at visit 3/baseline determines the weight range for the starting dose (PED25) and the up-titration dose (PED50) to be used in the table below:

Weight-based Doses for Tablets or Suspension

| PED | Weight Range | Suspension Volume † | <b>Tablet Dose</b> |
|-------|---------------|---------------------|--------------------|
| | 11 - < 22 kg | 3 mL | - |
| PED25 | 22 - < 35 kg | 4 mL | - |
| | ≥35 kg | 6 mL | 25 mg |
| | 11 - < 22 kg | 6 mL | - |
| 50 | 22 - < 35 kg | 8 mL | - |
| | ≥35 kg | 11 mL | 50 mg |

PED25: Pediatric equivalent dose 25 mg; PED50: Pediatric equivalent dose 50 mg † Suspension strength: 8 mg/mL

## **Further dosing information:**

- For subjects with a body weight  $\geq$  35 kg who do not want to or are unable to take tablets, the oral suspension can be supplied.
- At visit 8/week 24 subjects on mirabegron oral suspension may switch to tablets if the body weight turns to be  $\geq$  35 kg.
- Subjects receiving mirabegron tablets can switch to mirabegron oral suspension (and vice versa) for acceptability reasons after Sponsor's prior approval and on a case-by-case basis.

#### **Mode of Administration:**

Study drug will be taken orally, once a day in the morning around the same time of day and around time of food intake (i.e., within 1 hour before or after breakfast).

**Mirabegron** Ttablets to will be taken with a sip of water (tablet should be taken as a whole and should not be chewed, divided or crushed).

Mirabegron oral suspension will be administered via an oral syringe with a sip of water afterwards.

EudraCT number 2015-002876-25


On visit days where a pharmacokinetic sample is planned in the clinic, completion of breakfast and study drug dosing should occur in the clinic.

# IV Synopsis, Endpoints for Evaluation and 2 Study Objectives(s), Design, and Endpoints

2.3.2.3 Patient- or Clinician-reported Questionnaire Endpoints

#### WAS:

## Based on questionnaires:

• Acceptability questionnaire at visit 8/week 24 and visit 10/week 52 (EOT/EOS)

## IS AMENDED TO:

## Based on questionnaires:

• Acceptability questionnaire at **visit 5/week 4,** visit 8/week 24 and visit 10/week 52 (EOT/EOS)

# IV Synopsis, Endpoints for Evaluation, safety, Assessments, 2 Study Objective(s), Design, and Endpoints and 5 Treatments and Evaluation

2.3.3 Safety Endpoints and 5.4.1.2 Self-measurement of Vital Signs

#### WAS:

• Change from baseline in vital signs (SBPM): systolic blood pressure, diastolic blood pressure, pulse rate at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS)

#### IS AMENDED TO:

• Change from baseline in vital signs (self blood pressure measurement [SBPM]): systolic blood pressure, diastolic blood pressure, pulse rate at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) and on 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50 (visit 4/week 2, visit 5/week 4 or visit 6/week 8), if not already covered by the scheduled visit 4/week 2 and/or visit 5/week 4 SBPM.

#### 1 Introduction

1.4 Risk-Benefit Assessment

#### WAS:

Mirabegron has a favorable risk-benefit profile in adults in the indication OAB. In the pediatric phase 1 study executed thus far, mirabegron has an acceptable safety profile and was well tolerated.

#### IS AMENDED TO:

Mirabegron tablets has have a favorable risk-benefit profile in adults in the indication OAB. Mirabegron oral suspension has been shown to be safe and well tolerated in 2 phase 1

EudraCT number 2015-002876-25


**studies in healthy adult subjects (Studies 178-CL-201 and 178-CL-208).** In the pediatric phase 1 studyies executed thus far, mirabegron **tablets and mirabegron oral suspension** hasd an acceptable safety profile and wasere well tolerated.

#### 1 Introduction

## 1.4 Risk-Benefit Assessment

## WAS:

Regarding the formulation to be administered: the tablets are the same as used in adults. All excipients are pharmaceutical materials and are considered safe for the intended pediatric population.

## IS AMENDED TO:

Regarding the formulations to be administered: the tablets are the same as used in adults. for both the tablet and the suspension formulation, Aall excipients are pharmaceutical grade materials and are considered safe for the intended pediatric population.

## 2 Study Design and Dose Rationale

#### 2.2.2 Dose Rationale

## WAS:

The approved posology in adults for the treatment of OAB is either once daily 25 or 50 mg prolonged-release tablets. In children, the dosing strategy is based on extrapolation of efficacious doses in adults. Based on data obtained from adult and pediatric subjects following tablet and oral suspension dosing, a popPK model of steady state exposures will be used to predict the pediatric doses equivalent to 25 and 50 mg mirabegron administered once daily in adults. The target exposures for these pediatric equivalent doses (PED25 and PED50) are 69 ng·h/mL and 188 ng·h/mL, respectively. The popPK model indicates that pediatric subjects with a body weight of 35 kg or above can safely be dosed with the available tablets.

For pediatric subjects with a weight too low for dosing with tablets, or who cannot swallow the tablets, an oral suspension is under development. All subjects will start with the PED25 dose. Based on the criteria as described in [Section 5.1.2], the dose will be up-titrated to PED50 or will remain at PED25.

## IS AMENDED TO:

The approved posology in adults for the treatment of OAB is either once daily 25 or 50 mg prolonged release tablets. In children, the dosing strategy is based on extrapolation of efficacious doses in adults. Based on data obtained from adult and pediatric subjects following tablet and oral suspension dosing, a popPK model of steady state exposures will be used to predict the pediatric doses equivalent to 25 and 50 mg mirabegron administered once daily in adults. The target exposures for these pediatric equivalent doses (PED25 and PED50) are 69 ng h/mL and 188 ng h/mL, respectively. The popPK model indicates that pediatric subjects with a body weight of 35 kg or above can safely be dosed with the available tablets.

**Sponsor: APEB**EudraCT number 2015-002876-25


For pediatric subjects with a weight too low for dosing with tablets, or who cannot swallow the tablets, an oral suspension is under development. All subjects will start with the PED25 dose. Based on the criteria as described in [Section 5.1.2], the dose will be up titrated to PED50 or will remain at PED25.

The target exposures of 69 and 188 ng·h/mL for pediatric equivalent dose 25 mg (PED25) and pediatric equivalent dose 50 mg (PED50) were derived from the adult phase 3 program and are the mean steady state  $AUC_{tau}$  values following 25 and 50 mg prolonged-release tablets once daily in adults.

A population pharmacokinetic model was used to predict the PED for subjects in the 178-CL-206A study. In brief, this popPK model was developed on adult phase 3 data, and allometric (weight-based) scaling was added to all clearance and volume terms to allow for scaling of the pharmacokinetics to pediatric subjects. The model was validated on pediatric data in Study 178-CL-202 (single ascending-dose study) and was shown to appropriately predict the pharmacokinetics of mirabegron in pediatric subjects.

Simulations were then performed to determine a body weight at which subjects would have steady state exposures comparable to those in adults when dosed with 25 or 50 mg daily; this weight was determined to be  $\geq$  35 kg. Based on prior experience obtained in an ongoing Astellas study in another program in patients with NDO (Study 905-CL-047; IND 58135), the average age at which children reach a body weight of 35 kg is approximately 11 years. The dosing recommendation based on this modeling is in line with the literature [Momper et al, 2013] in which a meta-analysis of compounds submitted to the FDA with a similar indication in adults and adolescents showed that in almost all cases, the adolescents required the same dose as the adults.

Therefore, subjects with a body weight of  $\geq$  35 kg can be dosed with mirabegron tablets. Subjects with a body weight < 35 kg cannot be dosed with the 25 and 50 mg tablets because that would result in higher than target exposures. Subjects with a body weight < 35 kg will therefore be dosed with mirabegron oral suspension.

Mirabegron oral suspension (8 mg/mL) has been developed for use in the pediatric population. The population pharmacokinetic model referred to above includes a formulation factor to account for the different (lower) relative bioavailability of the oral suspension compared to the tablet. This factor has been used in simulations to predict the suspension doses and weight categories that would have a reasonable variance around the target exposures.

For dosing with oral suspension, the weight range to be covered is from 11 kg (the approximate body weight of a 3-year-old child, according to the NHANES database [McDowell et al, 2008]) to 35 kg (above which pediatric subjects could be dosed with the tablet formulation). Subjects with a body weight < 11 kg will not be included in the study. Suspension dosing for body weights  $\ge$  35 kg was also determined for cases in which a pediatric subject in that weight category does not want or would be unable to swallow a tablet. The simulation resulted in the 3 body weight categories that can be found in the dosing schedule (see [Section 5.1.1]).

EudraCT number 2015-002876-25


## 4 Treatment(s)

## 4.1.1 Test Drug

#### WAS:

For detailed information on mirabegron tablets, please refer to the Investigational Medicinal Product Dossier (IMPD) or IND.

Mirabegron is supplied as tablets containing 25 mg or 50 mg of active ingredient.

## IS AMENDED TO:

Mirabegron oral suspension has been developed as an appropriate formulation for weight based dosing in smaller children.

For detailed information on mirabegron **prolonged-release** tablets and **mirabegron granules for oral suspension**, please refer to the **applicable** Investigational Medicinal Product Dossier (IMPD)-or IND.

Mirabegron **tablets are** is supplied as **prolonged-release** tablets containing 25 mg or 50 mg of active ingredient.

For the oral suspension, mirabegron prolonged-release granules are supplied and will be reconstituted with water to prepare an oral suspension of 8 mg/mL. Detailed information on the preparation of the mirabegron oral suspension will be provided to the subject and subject's parent(s)/caregiver(s) in local language. Due to shelf-life limitations, an additional dispensing visit is foreseen at visit 9/week 36 for subjects receiving mirabegron oral suspension. This dispensing visit does not need to be accompanied by the subject.

## **5 Treatments and Evaluation**

5.1.1 Dose/Dose Regimen and Administration Period

## WAS:

Each tablet is to be taken with a sip of water. The tablet should be taken as a whole and should not be chewed, divided or crushed.

#### IS AMENDED TO:

Each Mirabegron tablets is to will be taken with a sip of water. The tablet should be taken as a whole and should not be chewed, divided or crushed.

Mirabegron prolonged-release granules will be reconstituted with water to prepare a mirabegron oral suspension of 8 mg/mL. Administration will be via an oral syringe with a sip of water afterwards. Detailed information on the preparation of the suspension will be provided to the subject and subject's parent(s)/caregiver(s) in local language. For subjects receiving mirabegron oral suspension, an additional (optional) dispensing visit is scheduled at visit 9/week 36.

## **Selection of the formulation:**

Subjects with a body weight < 35 kg: mirabegron oral suspension.

Subjects with a body weight  $\geq$  35 kg: mirabegron tablets.

## **Selection of the dose:**

Doses are calculated weight-based. The bodyweight at visit 3/baseline determines the

**Sponsor: APEB** EudraCT number 2015-002876-25


weight range for the starting dose (PED25) and the up-titration dose (PED50) to be used [Table 4].

Table 4 Weight-based doses for tablets or suspension

| | Weight Range | Suspension Volume † | Tablet Dose |
|-------|--------------|---------------------|-------------|
| | 11 - < 22 kg | 3 mL | - |
| PED25 | 22 - < 35 kg | 4 mL | - |
| | ≥ 35 kg | 6 mL | 25 mg |
| | 11 - < 22 kg | 6 mL | - |
| PED50 | 22 - < 35 kg | 8 mL | - |
| | ≥ 35 kg | 11 mL | 50 mg |

PED25: Pediatric equivalent dose 25 mg; PED50: Pediatric equivalent dose 50 mg † Suspension strength: 8 mg/mL

## **Further dosing information:**

- For subjects with a body weight  $\geq$  35 kg who do not want to or are unable to take tablets, the oral suspension can be supplied.
- At visit 8/week 24 subjects on mirabegron oral suspension may switch to tablets if the body weight turns to be  $\geq$  35 kg.
- Subjects receiving mirabegron tablets can switch to mirabegron oral suspension (and vice versa) for acceptability reasons after Sponsor's prior approval and on a case-by-case basis.

#### **5 Treatments and Evaluation**

## 5.3.3 Questionnaires

## WAS:

- The PIN-Q [Appendix 12.4] will be administered on one weekend day preceding visit 3/baseline, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The PGI-S [Appendix 12.5] will be administered on one weekend day preceding visit 3/baseline, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The Acceptability Questionnaire [Appendix 12.6] will be administered on one weekend day preceding visit 8/week 24 and at visit 10/week 52 (EOT/EOS).
- The CGI-C [Appendix 12.7] will be administered at visit 8/week 24 and at visit 10/week 52 (EOT/EOS).

## IS AMENDED TO:

- The PIN-Q [Appendix 12.4] will be administered completed on one weekend day preceding visit 3/baseline, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The PGI-S [Appendix 12.5] will be administered completed on one weekend day preceding visit 3/baseline, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The Acceptability Questionnaire [Appendix 12.6] will be administered completed on one weekend day preceding visit 5/week 4, visit 8/week 24 and at visit 10/week 52 (EOT/EOS). For each formulation a separate questionnaire is available [Appendix 12.6 and Appendix 12.7].

**Sponsor: APEB** EudraCT number 2015-002876-25


11 References

ADDED:

• The CGI-C [Appendix **12.–78**] will be administered completed at visit 8/week 24 and at visit 10/week 52 (EOT/EOS).

McDowell MA, Fryar CD, Ogden CL, Flegal KM. Anthropometric reference data for children

| | and adults: United States, 2003–2006. Natl Health Stat Report. 2008;22(10):1-48. | | | |
|---|---|---|---|---|
| Momper JD, Mulu | | | | |
| | | | | lments Act of 2007. |
| JAMA Pedia | tr. 2013;167(10):92 | 6-932. doi:10.1001/ | jamapediatrics.201 | 3.465. |
| 12 Appendices | | | | |
| ADDED: | | | | |
| 12.7 Acceptability Questionnaire for Oral Suspension | | | | |
| Questions | | | | |
| 3. How was the <u>TASTE</u> of the study drug? | | | | |
| 0 | 1 | 2 | 3 | 4 |
| (••) (••) (••) (••) (••) | | | | |
| ( | | | | |
| Really bad Bad Not bad, not Good Really good | | | | |
| Really bad | Bud | good | dood | really good |
| 4. How was t | he <u>SMELL</u> of tl | ne study drug? | | |
| 0 | 1 | 2 | 3 | |
| l | 1 | 2 | 3 | 4 |
| (••) (••) (••) (••) | | | | |
| Really bad | Bad | Not bad, not | Good | Really Good |
| | | good | | |
| 5. How was i | 5. How was it to <u>TAKE</u> the study drug? | | | |

EudraCT number 2015-002876-25


| 0 Really difficult | 1<br>Difficult | 2 Not difficult, not easy | 3<br>Easy | 4 Really easy |
|---|---|---|---|---|
| | A DDEDADE | | | |
| 6. How was I | t to <u>PREPARE</u> | the study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| Really difficult | Difficult | Not difficult,<br>not easy | Easy | Really easy |

# III. Amendment Summary of Changes: Non-Substantial

| Cover Page |
|------------|
| DELETED: |
| IND 69,416 |

## IV. Synopsis

Study Design Overview

# WAS:

If a symptomatic UTI is present at baseline, all baseline assessments are allowed to be postponed for a maximum of 7 days until the UTI is successfully treated.

## IS AMENDED TO:

If a symptomatic UTI is present at baseline, all baseline assessments are allowed to should be postponed for a maximum of 7 days until the UTI is successfully treated (clinical recovery). The 7-day baseline e-diary does not have to be repeated if at least the 2-day

EudraCT number 2015-002876-25


weekend e-diary and 1 day of the weekday e-diary were completed while the subject did not suffer from a symptomatic UTI.

## IV. Synopsis

Study Design Overview

## ADDED:

The 7-day e-diary does not have to be repeated if at least the 2-day weekend e-diary and 1 day of the weekday e-diary were completed while the subject did not suffer from a symptomatic UTI.

If a subject suffers from a symptomatic UTI in the week prior to any other study visit, these visits do not need to be postponed and the 7-day e-diary does not have to be repeated.

# IV Synopsis, Study Design Overview and 2 Study Objective(s), Design, and Endpoints 2.2.1.1 Pretreatment Period

#### WAS:

Subjects will enter the efficacy treatment period if they meet the eligibility criteria and satisfactorily complete the pretreatment period (ability to complete bladder diary, catheterized volumes, self-measurement of intravesical pressures [SMIP], questionnaires and self blood pressure measurement [SBPM]).

#### IS AMENDED TO:

Subjects will enter the efficacy treatment period if they meet the eligibility criteria and satisfactorily complete the pretreatment period (ability to complete bladder diary, catheterized volumes, self measurement of intravesical pressures [SMIP], and questionnaires).

## IV Synopsis, Dose Titration and 5 Treatments and Evaluation

5.1.2 Increase or Reduction in Dose of the Study Drug(s)

## WAS:

1. The investigator considers the subject to be effectively treated with PED25, based on urodynamics, e-diary and SMIP (if available);

#### IS AMENDED TO:

1. The investigator considers the subject to be effectively treated with PED25, based on urodynamics, and the e-diary-and SMIP (if available);

# IV. Synopsis, Exploratory Efficacy and 2 Study Objective(s), Design, and Endpoints

2.3.5.1 Exploratory Efficacy Endpoints

WAS:

EudraCT number 2015-002876-25


#### Based on e-diary:

Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) in:

- Mean grade of leakage
- Total catheterized volume per 24 h
- Maximum confirmed daytime dry period/24 h
- Maximum confirmed daytime dry period/7 days
- Change from baseline in SMIP-derived bladder compliance
- Number of CICs/day
- Responder in respect to leakage (complete, partial, no response)

#### IS AMENDED TO:

## Based on e-diary:

Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) in:

- Mean grade of leakage
- Total catheterized volume per 24 hday
- Maximum confirmed daytime dry period/24 h
- Maximum confirmed daytime dry period/7 days
- Change from baseline in SMIP-derived bladder compliance
- Number of CICs/day
- Responder in respect to leakage (complete, partial, no response)

## IV Synopsis, Assessments and 5 Treatments and Evaluation

5.3.1 Urodynamic Assessments

#### WAS:

Additional urodynamic assessments can be performed at visit 10/week 52 (EOT/EOS), or at any other time point when deemed necessary by the investigator (e.g., confirmatory urodynamic assessments at visit 7/week 12 if up-titration or down-titration was done at visit 6/week 8, or when the SMIP was not performed).

## IS AMENDED TO:

Additional urodynamic assessments can be performed at visit 10/week 52 (EOT/EOS), or at any other time point when deemed necessary by the investigator (e.g., confirmatory urodynamic assessments at visit 7/week 12 if up titration or down titration was done at visit 6/week 8, or when the SMIP was not performed).

# IV. Synopsis, Patient Reported Outcome Data and 8 Operational and Administrative Considerations

8.1.1.1 Electronic Patient Reported Outcomes

## WAS:

- Bladder diary:
  - o Each day for 7 days: time of CICs
  - o Each day for 7 days: presence of leakage between CICs
  - o Each day for 7 days: sleep time and wake-up time

02 Nov 2016 Astellas 

ISN/Protocol 178-CL-206A

**Sponsor: APEB**EudraCT number 2015-002876-25


- o On the 2 weekend days: catheterized volume
- o On the 2 weekend days: SMIP (if applicable)
- o On the 2 weekend days: grade of leakage between CICs
- o On the 2 weekend days (visit 3/baseline and visit 8/week 24): weight of diaper/pad
- SBPM (blood pressure and pulse rate):
  - o On the 2 weekend days: triplicate measurements in the morning and evening
- Questionnaires: on 1 weekend day at selected visits
  - o PIN-Q
  - o PGI-S
  - Acceptability
- Confirmation of study drug intake: daily

## IS AMENDED TO:

- Bladder diary:
  - o Each day for 7 days: time of CICs
  - o Each day for 7 days: presence of leakage between CICs
  - o Each day for 7 days: sleep time and wake-up time
  - o On the 2 weekend days: catheterized volume
  - o On the 2 weekend days: SMIP (if applicable)
  - o On the 2 weekend days: grade and number of leakages between CICs
  - On the 2 weekend days (visit 3/baseline and visit 8/week 24): weight of diaper/pad
- SBPM (blood pressure and pulse rate):
  - o On the 2 weekend days: triplicate measurements in the morning and evening
  - On 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM.
- Questionnaires: on 1 weekend day at selected visits
  - o PIN-Q
  - o PGI-S
  - o Acceptability
- Confirmation of study drug intake: daily

The Investigator must guide the subject and subject's parent(s)/caregiver(s) to ensure that on the evening before and during the two weekend days of collection of catheterized volume and SMIP (if applicable), the subject's fluid intake should be regulated to an appropriate level taking e.g. age, sex and subject's condition into account. The intake must remain as consistent as possible on these volume collecting days throughout the entire study.

## IV. Synopsis, Statistical Methods

#### WAS:

## Sample size justification:

In order to allow the detection of a statistically significant change from baseline in MCC in the overall NDO with CIC study population with 90% power, 44 evaluable subjects for the assessment of the endpoint need to be enrolled, i.e., subjects with a nonmissing MCC measurement at baseline and at a postbaseline visit. The power calculation is based upon a paired t-test with a 2-sided significance level of 0.05, a real change from baseline of at least 52 mL and a SD of not larger than 103 mL. Assuming 30% of enrolled subjects will not be

EudraCT number 2015-002876-25


evaluable, a total of approximately 63 subjects may need to be enrolled.

Four analysis populations will be defined: the safety analysis set (SAF), full analysis set (FAS), per protocol set (PPS), and pharmacokinetic analysis set (PKAS) for pharmacokinetic population analysis.

#### IS AMENDED TO:

## Sample size justification:

In order to allow the detection of a statistically significant change from baseline in MCC in the overall NDO with CIC study population with 90% power, 44 evaluable subjects for the assessment of the endpoint need to be enrolled, i.e., subjects with a **valid** (as by the central reviewer's assessment) nonmissing MCC measurement at baseline and at a postbaseline visit. The power calculation is based upon a paired t-test with a 2-sided significance level of 0.05, an real expected change from baseline of at least 52 mL and a SD of not larger than 103 mL. Assuming 30% of enrolled subjects will not be evaluable, a total of approximately 63 subjects may need to be enrolled.

Four analysis populations will be defined: the safety analysis set (SAF), full analysis set (FAS), per protocol set (PPS), and pharmacokinetics analysis set (PKAS) for pharmacokinetic population analysis.

## V Flowchart and Schedule of Assessments

Table 1: Schedule of Assessments

See next page.

Sponsor: APGD - CONFIDENTIAL -

| WAG | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| WAS: | | | | | | | | | | |
| | Visit 1 | Visit 2 /TC 1 | Visit 3 | Visit 4<br>/TC 2 <sup>†</sup> | Visit 5 | Visit 6<br>/TC 3 <sup>†</sup> | Visit 7 | Visit 8 | Visit 9<br>/TC 4 <sup>†</sup> | Visit 10<br>/EOS <sup>‡</sup> |
| Assessments | Screening | Start of<br>Washout ††† | Baseline | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | Week 36 | Week 52 |
| | Day -28 to<br>Day -15 | Day -15 to<br>Day -8 | Day -1 | Day 14<br>(±3 days) | Day 28<br>(±3 days) | Day 56<br>(±7 days) | Day 84<br>(±7 days) | Day 168<br>(±7 days) | Day 252<br>(±14 days) | Day 364<br>(±14 days) |
| Signing informed consent form | X | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | X | | | | | | | |
| Demographics | X | | | | | | | | | |
| Height & weight | X | | X | | | | | X | | X |
| Medical history (including NDO) | X | | | | | | | | | |
| Current NDO medications | X | X | | | | | | | | |
| Vital signs (triplicate) and body temperature (ear) § | x | | X | | X | | X | X | | X |
| Physical examination | X | | | | | | | | | X |
| 12-lead ECG (triplicate) ¶ | X | | X | | X | | X | X | | X |
| Hematology/Biochemistry/eGFR | X | | (X) †† | | (X) †† | | X | | | X |
| Urinalysis | X | | X | | X | | X | X | | X |
| Pregnancy test ‡‡ | X | | X | | X | | X | X | | X |
| Pharmacokinetics §§ | | | | | (X) | (X) | (X) | (X) | (X) | (X) |
| Upper urinary tract ultrasound | | | X | | | | | | | X |
| Urodynamic assessments 11 | | | X | | X | | | X | | |
| Dose-titration assessment | | | | X | X | X | | | | |
| Dispense study drug ††† | | | X | | X | | X | X | | |
| Bladder diary, SMIP and collection of catheterized volume 1111 | | X | X | X | X | Х | X | X | X | Х |
| SBPM (triplicate) §§§ | | X | X | X | X | X | X | X | X | X |
| PIN-Q, PGI-S | | | X | | | | | X | | X |
| CGI-C | | | | | | | | X | | X |
| Acceptability questionnaire | | | | | | | | X | | X |
| Adverse events and previous and | _ | | | | | | | | | _ |
| concomitant medication | • | | | | | | | | | • |

ECG: Electrocardiogram; EOS: end of study; CGI-C: Clinician Global Impression of Change scale; DSMB: Data and Safety Monitoring Board; NDO: neurogenic detrusor overactivity; PGI-S: Patient Global Impression of Severity Scale; PIN-Q: Pediatric Incontinence Questionnaire; SBPM: self blood pressure measurement; SMIP: self-measurement of intravesical pressure; TC: telephone contact.

See Footnotes on next page

- † For the visits where a TC is indicated there is no need for the subject to visit the clinic, provided that the e-diary data is reviewed by the investigator prior to the TC and discussed and confirmed with the subject or parent(s)/caregiver(s) during the TC.
- \$\frac{1}{2}\$ Subjects who withdraw early from the study after having received study drug should complete the EOS visit. If the final dose is reached before the last possibility for uptitration at 8 weeks, the fixed-dose treatment period will be extended to keep the entire treatment period 364 days as a minimum. The maximum is 378 days in order to allow for visit windows.
- § Triplicate vital signs with an interval of approximately 2 minutes in the sitting position (when possible, otherwise supine, but always in the same position). Preferably the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Clinic measurements will be used to assess eligibility. Single measurements for body temperature must be performed with an ear thermometer.
- Triplicate 12-lead ECG with an interval of about 30 seconds to 5 minutes in the supine position (when possible, but always in the same position). Subject should have been calm and without distress for at least 5 minutes.
- †† Additional hematology/biochemistry taken at baseline only if an AE related to hematology/biochemistry parameters occurred between visit 1/screening and visit 3/baseline. The first group of subjects (minimum of 5, maximum of 10) who reach study visit 5/week 4 will have an additional blood draw for a DSMB-mandated interim safety check at this visit. For sampling, preferably the left arm should be used. Blood sampling should occur after vital signs and ECG measurements.
- Pregnancy test in female subjects of childbearing potential in serum (if blood is drawn) or urine (at other visits).
- §§ If the subject reached steady state of her/his optimal dose, a total of 4 pharmacokinetic samples will be collected, divided over 2 sampling days. Sampling day 1: 1 trough sample; Sampling day 2: 1 trough and 2 postdose samples between 2 h and 5 h postdose, with at least 1 hour in between the samples. These 2 sampling days do not have to be in a specific order and can be selected from the given options. Dosing on a sampling day with postdose samples must occur within 1 hour after completion of breakfast [Section 5.3.4]. On days where a pharmacokinetic visit is planned in the clinic, breakfast and dosing should occur in the clinic. Blood sampling should occur after vital signs and ECG measurements.
- Additional urodynamic assessments may be performed if deemed necessary by the investigator (e.g., if SMIP is not performed at visit 4/week 2, confirmatory urodynamic assessments at visit 7/week 12 if up-titration or down-titration was done at visit 6/week 8, or an additional urodynamic assessment at visit 10/week 52 [EOT/EOS]).
- ††† Daily study drug administration will begin on Day 1 (the day after visit 3/baseline).
- ‡‡‡ After a successful screening visit, all subjects start with the completion of a 2-day weekend e-diary visit to get acquainted with the e-diary and the assessments.

  Completion of this diary should start in the weekend prior to visit 2. Completion of subsequent bladder diaries should start approximately 7 days prior to the indicated visit (or TC). If successful completion of the 2-day weekend e-diary is confirmed at visit 2, subjects from group A start with collection of the 7-day baseline e-diary, followed by the baseline visit. Subjects in group B start with a 14-day washout. In the second week of the washout period, collection of their 7-day baseline e-diary starts, followed by the baseline visit.

§§§ Triplicate SBPM will be performed in the morning and evening during the 2-day weekend e-diary collection period. Measurements to be taken with an interval of approximately 2 minutes in the sitting position (when possible, otherwise supine, but always in the same position). Preferably the right arm should be used. Morning measurements should be taken after waking-up, before breakfast and before study drug intake, evening measurements prior to bedtime. Subject should have been calm and without distress for at least 5 minutes.

02 Nov 2016 Astellas 

Sponsor: APGD - CONFIDENTIAL -

| IS A | MEN | DED | TO: |
|------|-----|-----|-----|
|------|-----|-----|-----|

| | Visit 1 | Visit 2/TC 1 | Visit 3 | Visit 4<br>/TC 2 <sup>†</sup> | Visit 5 | Visit 6<br>/TC 3 <sup>†</sup> | Visit 7 | Visit 8 | Visit 9<br>/TC 4 <sup>†</sup> | Visit 10<br>/EOS <sup>‡</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Screening | Start of<br>Washout ††† | Baseline | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | Week 36 | Week 52 |
| | Day -28 to<br>Day -15 | Day -15 to<br>Day -8 | Day -1 | Day 14 (±+3 days) | Day 28<br>(±+3 days) | Day 56<br>(±7 days) | Day 84<br>(±7 days) | Day 168<br>(±7 days) | Day 252<br>(±14 days) | Day 364<br>(±14 days) |
| Signing informed consent form | X | | | • | | | | • | • | • |
| Inclusion/Exclusion criteria | X | | X | | | | | | | |
| Demographics | X | | | | | | | | | |
| Height & weight | X | | X | | | | | X | | X |
| Medical history (including NDO) | X | | | | | | | | | |
| Current NDO medications | X | X | | | | | | | | |
| Vital signs (triplicate) and body temperature (ear) § | X | | X | | X | | X | Х | | X |
| Physical examination | X | | | | | | | | | X |
| 12-lead ECG (triplicate) | X | | X | | X | | X | X | | X |
| Hematology/Biochemistry/eGFR | X | | (X) †† | | (X) <sup>††</sup> | | X | | | X |
| Urinalysis | X | | X | | X | | X | X | | X |
| Pregnancy test ‡‡ | X | | X | | X | | X | X | | X |
| Pharmacokinetics §§ | | | | | (X) | (X) | (X) | (X) | (X) | (X) |
| Upper urinary tract ultrasound | | | X | | | | | | | X |
| Urodynamic assessments ¶ | | | X | | X | | | X | | |
| Dose-titration assessment | | | | X | X | X | | | | |
| Dispense study drug ††† | | | X | | X | | X | X | (X) | |
| Bladder diary, SMIP and collection of catheterized volume ††‡ | | X | X | X | X | X | X | X | X | X |
| SBPM (triplicate) §§§ | | X | X | X | X | X | X | X | X | X |
| PIN-Q, PGI-S | | | X | | | | | X | | X |
| CGI-C | | | | | | | | X | | X |
| Acceptability questionnaire | | | | | X | | | X | | X |
| Adverse events and previous and | | | | | | | | | | |
| concomitant medication | | | | | | | | | | |

ECG: Electrocardiogram; EOS: end of study; CGI-C: Clinician Global Impression of Change scale; DSMB: Data and Safety Monitoring Board; NDO: neurogenic detrusor overactivity; PGI-S: Patient Global Impression of Severity Scale; PIN-Q: Pediatric Incontinence Questionnaire; SBPM: self blood pressure measurement; SMIP: self-measurement of intravesical pressure; TC: telephone contact.

See Footnotes on next page

- † For the visits where a TC is indicated there is no need for the subject to visit the clinic, provided that the e-diary data is reviewed by the investigator prior to the TC and discussed and confirmed with the subject or **the subject's** parent(s)/caregiver(s) during the TC.
- \$\frac{1}{2}\$ Subjects who withdraw early from the study after having received study drug should complete the EOS visit. If the final dose is reached before the last possibility for uptitration at 8 weeks, the fixed-dose treatment period will be extended to keep the entire treatment period 364 days as a minimum. The maximum is 378 days in order to allow for visit windows.
- § Triplicate vital signs with an interval of approximately 2 minutes in the sitting position (when possible, otherwise supine, but always in the same position). Preferably the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Clinic measurements will be used to assess eligibility. Single measurements for body temperature must be performed with an ear thermometer.
- Triplicate 12-lead ECG with an interval of about 30 seconds to 5 minutes in the supine position (when possible, but always in the same position). Subject should have been calm and without distress for at least 5 minutes.
- †† Additional hematology/biochemistry taken at baseline only if an AE related to hematology/biochemistry parameters occurred between visit 1/screening and visit 3/baseline. The first group of subjects (minimum of 5, maximum of 10) who reach study visit 5/week 4 will have an additional blood draw for a DSMB-mandated interim safety check at this visit. For sampling, preferably the left arm should be used. Blood sampling should occur after vital signs and ECG measurements.
- ‡‡ Pregnancy test in female subjects of childbearing potential in serum (if blood is drawn) or urine (at other visits).
- If the subject reached steady state of her/his optimal dose, a total of 4 pharmacokinetic samples will be collected, divided over 2 sampling days. Sampling day 1: 1 trough sample; Sampling day 2: 1 trough and 2 postdose samples between 2 h and 5 h postdose, with at least 1 hour in between the samples. These 2 sampling days do not have to be in a specific order and can be selected from the given options. **To allow for an early assessment of the dose-response relationship by the DSMB, it is preferred the pharmacokinetic sampling takes place as early in the study as possible.** Dosing on a sampling day with postdose samples must occur within 1 hour after completion of breakfast [Section 5.3.4]. On days where a pharmacokinetic visit is planned in the clinic, breakfast and dosing should occur in the clinic. Blood sampling should occur after vital signs and ECG measurements.
- Additional urodynamic assessments may be performed if deemed necessary by the investigator (e.g., if SMIP is not performed at visit 4/week 2, confirmatory urodynamic assessments at visit 7/week 12 if up titration or down titration was done at visit 6/week 8, or an additional urodynamic assessment at visit 10/week 52 [EOT/EOS]).
- ††† Daily study drug administration will begin on Day 1 (the day after visit 3/baseline). Due to shelf-life limitations, an additional dispensing visit is foreseen at visit 9/week 36 for subjects receiving mirabegron oral suspension. This dispensing visit does not need to be accompanied by the subject.
- ‡‡‡ After a successful screening visit, all subjects start with the completion of a 2-day weekend e-diary visit to get acquainted with the e-diary and the assessments.

  Completion of this diary should start in the weekend prior to visit 2. Completion of subsequent bladder diaries should start approximately 7 days prior to the indicated visit (or TC). If successful completion of the 2-day weekend e-diary is confirmed at visit 2, subjects from group A start with collection of the 7-day baseline e-diary, followed by the baseline visit. Subjects in group B start with a 14-day washout. In the second week of the washout period, collection of their 7-day baseline e-diary starts, followed by the baseline visit.
- §§§ Triplicate SBPM will be performed in the morning and evening during the 2-day weekend e-diary collection period and on 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM. Measurements to be taken with an interval of approximately 2 minutes in the sitting position (when possible, otherwise supine, but always in the same position). Preferably the right arm should be used. Morning measurements should be taken after waking-up, before breakfast and before study drug intake, evening measurements prior to bedtime. Subject should have been calm and without distress for at least 5 minutes.

02 Nov 2016 Astellas 

EudraCT number 2015-002876-25


## 1 Introduction

## 1.2.2 Clinical Data

## WAS:

The global pediatric development program for mirabegron in NDO and OAB currently consists of 8 studies in various stages of completion.

The first available clinical data of mirabegron in children comes from study 178-CL-202: a single ascending dose phase 1 study with mirabegron tablets in pediatric subjects diagnosed with OAB or NDO.

Cohort 1: male and female adolescents (12 to less than 18 years); low dose and fed

Cohort 2: male and female children (5 to less than 12 years); low dose and fed

Cohort 3: male and female adolescents (12 to less than 18 years); high dose and fed

Cohort 4: male and female children (5 to less than 12 years); high dose and fed

Cohort 5: male and female children (5 to less than 12 years); high dose and fasted Fed: within one hour after a light breakfast

Low dose: single oral doses that are predicted to result in an exposure comparable to that in adults when dosed with 25 mg mirabegron tablets once daily at steady-state (69 ng.h/mL). High dose: single oral doses that are predicted to result in an exposure comparable to that in adults when dosed with 50 mg mirabegron tablets once daily at steady-state (188 ng.h/mL). The doses in Study 178-CL-202 were predicted applying an allometric scaling approach of the data obtained in adults under non standardized food conditions.

A dose escalation committee including a pediatric nephrologist and pediatric cardiologist has reviewed the data obtained in these cohorts and concluded that mirabegron exposure was within the predicted target ranges for all cohorts and that mirabegron showed an acceptable safety profile at the doses tested.

5 TEAEs were reported: 'vomiting'(2x), 'fever', 'mean QT interval corrected by Bazett's formula (QTcB) of 452 ms' and 'QTcB prolongation'. The intensity for all TEAEs was mild and only one (QTcB prolongation versus baseline) was judged by the investigator to be possibly related to study drug. No QTc prolongation > 60 ms versus baseline was observed (mean of triplicates).

No clinically significant increases in vital signs have been observed. Increases in pulse rate were observed across all cohorts but these were not considered clinically significant/relevant per investigator's assessment.

The centrally read Holter observations in cohort 4 and 5 showed a trend towards 2 episodes of a mean and median increase in mean hourly heart rate; the first one starting 4 to 6 hours postdose and reaching the highest values at 6 to 8 hours after dosing and the second one starting 10-12h after dosing and continuing until the end of the recording, without a change in circadian rhythm. This was not considered as clinically relevant by the dose escalation committee.

For pediatric subjects an oral suspension is under development.

## IS AMENDED TO:

The global pediatric development program for mirabegron in NDO and OAB currently consists of 8 studies in various stages of completion.

The first available clinical data of mirabegron in children comes from study 178 CL 202: a single ascending dose phase 1 study with mirabegron tablets in pediatric subjects diagnosed with OAB or NDO.

Sponsor: APEB
EudraCT number 2015-002876-25


- Cohort 1: male and female adolescents (12 to less than 18 years); low dose and fed
- Cohort 2: male and female children (5 to less than 12 years); low dose and fed
- Cohort 3: male and female adolescents (12 to less than 18 years); high dose and fed
- Cohort 4: male and female children (5 to less than 12 years); high dose and fed
- Cohort 5: male and female children (5 to less than 12 years); high dose and fasted Fed: within one hour after a light breakfast

Low dose: single oral doses that are predicted to result in an exposure comparable to that i adults when dosed with 25 mg mirabegron tablets once daily at steady state (69 ng.h/mL). High dose: single oral doses that are predicted to result in an exposure comparable to that it adults when dosed with 50 mg mirabegron tablets once daily at steady state (188 ng.h/mL)

The doses in Study 178 CL 202 were predicted applying an allometric scaling approach of the data obtained in adults under non standardized food conditions.

A dose escalation committee including a pediatric nephrologist and pediatric cardiologist has reviewed the data obtained in these cohorts and concluded that mirabegron exposure was within the predicted target ranges for all cohorts and that mirabegron showed an acceptable safety profile at the doses tested.

5 TEAEs were reported: 'vomiting'(2x), 'fever', 'mean QT interval corrected by Bazett's formula (QTcB) of 452 ms' and 'QTcB prolongation'. The intensity for all TEAEs was mild and only one (QTcB prolongation versus baseline) was judged by the investigator to be possibly related to study drug. No QTc prolongation > 60 ms versus baseline was observed (mean of triplicates).

No clinically significant increases in vital signs have been observed. Increases in pulse rate were observed across all cohorts but these were not considered clinically significant/ relevant per investigator's assessment.

The centrally read Holter observations in cohort 4 and 5 showed a trend towards 2 episodes of a mean and median increase in mean hourly heart rate; the first one starting 4 to 6 hours postdose and reaching the highest values at 6 to 8 hours after dosing and the second one starting 10 12h after dosing and continuing until the end of the recording, without a change in circadian rhythm. This was not considered as clinically relevant by the dose escalation committee.

For pediatric subjects an oral suspension is under development.

The main clinical aspects of mirabegron prolonged-release tablets in adults are described in the current locally-available product information for mirabegron. To support the doses and formulations (tablets and oral suspension) selected for this study, the pediatric development program for mirabegron includes 4 phase 1 studies [Table 2].

Table 2 Overview of Current Supporting Mirabegron Studies in the Pediatric Clinical Development Program for NDO and OAB

| Study Number | Study Title | Study Progress |
|---|---|---|
| 178-CL-201 | A phase 1, single dose, 4-period crossover study to assess the bioavailability of mirabegron oral suspension relative to the mirabegron prolonged-release tablet and to assess the effect of food on the pharmacokinetics of mirabegron oral suspension in healthy young male and | Completed |

EudraCT number 2015-002876-25


| | female subjects. | |
|---|---|---|
| 178-CL-202 | A multicentre, open-label, single ascending dose phase 1 study to evaluate the pharmacokinetics, safety and tolerability of mirabegron OCAS tablets in pediatric subjects from 5 to less than 18 years of age with neurogenic detrusor overactivity (NDO) or overactive bladder (OAB). | Completed |
| 178-CL-203 | A multicentre, open-label, single dose, phase 1 study to evaluate the pharmacokinetics, safety and tolerability of mirabegron oral suspension in pediatric subjects from 3 to less than 12 years of age with neurogenic detrusor overactivity (NDO) or overactive bladder (OAB). | Ongoing |
| 178-CL-208 | A phase 1, single dose, 3-period crossover study to assess the bioavailability of an oral suspension of 8 mg/mL mirabegron relative to the oral suspension of 2 mg/mL mirabegron and to assess the effect of food on the pharmacokinetics of the oral suspension of 8 mg/mL mirabegron in healthy male and female adult subjects | Ongoing |

The results of studies 178-CL-201 and 178-CL-202 are reported in the most recent version of the pediatric IB. The data from these studies were used to support the use of tablets in pediatric subjects with a body weight of ≥ 35 kg in this study. For those pediatric subjects that cannot be dosed with tablets because their body weight is 35 kg or less or because they cannot swallow tablets, an oral suspension with a strength of 2 mg/mL was developed. The relative bioavailability was assessed in healthy subjects (178-CL-201) to be 53.44% lower compared to tablets. The results of this study and study 178-CL-202 were used to support the use of the 2 mg/mL in study 178-CL-203.

That study is a single dose phase 1 study with mirabegron oral suspension in pediatric subjects from 3 to less than 12 years of age with NDO and in pediatric subjects from 5 to less than 12 years of age with OAB. This study is currently ongoing with 6 of 9 planned subjects having completed the study. Single doses of mirabegron are administered that are predicted to result in an exposure comparable to that in adults when dosed with 50 mg mirabegron tablets once daily at steady-state (188 ng·h/mL). Subjects received mirabegron oral suspension within 1 hour after a light breakfast. Doses were compensated for the lower bioavailability of suspension versus tablets (see above). This study is ongoing but the preliminary results are provided below. It became apparent that with a strength of 2 mg/mL the volume of the doses the patients have to take every day would be too high (up to 44 mL). To overcome this issue, an oral suspension of 8 mg/mL was developed.

To support the use of this 8 mg/mL mirabegron oral suspension in pediatric subjects, study 178-CL-208 was conducted. The study follows a single dose, three period cross over design in healthy subjects. Subjects received the following three treatments in

ISN/Protocol 178-CL-206A

Sponsor: APEB
EudraCT number 2015-002876-25


random order: 1) 11mL 8 mg/mL oral suspension of mirabegron under fasted conditions, 2) 11mL 8 mg/mL oral suspension of mirabegron under fed conditions and 3) 44 mL 2 mg/mL oral suspension of mirabegron under fasted conditions. This study is ongoing, but a summary of the preliminary results is provided below. Exposure:

The single doses of the 2 mg/mL oral suspension for Study 178-CL-203 were predicted using a population pharmacokinetic (popPK) model developed on pharmacokinetic data obtained in Study 178-CL-201, with food, dose, and formulation effects on the bioavailability, and was validated on data from Study 178-CL-202. The observed exposures were in line with the target exposure of 188 ng·h/mL; the median AUC24 was 207 ng·h/mL (n=6, mean (SD): 226.4 (152.3), range: 39.7-467). These preliminary results suggest that the use of the popPK model is appropriate for dose selection. The model predictions of the PED50 doses at a strength of 2 mg/mL would require large volumes of oral suspension every day (up to 44 mL). Therefore, to reduce the volume, a higher strength oral suspension was developed.

The primary objective of study 178-CL-208 was to assess the relative bioavailability of the 8 mg/mL oral suspension compared to the 2 mg/mL oral suspension under fasted conditions. The results of study 178-CL-208 show that the bioavailability of both strengths is comparable [Table 3].

Table 3

178-CL-208 Draft Results: Relative Bioavailability of the Mirabegron
8 mg/mL Oral Suspension Formulation versus 2 mg/mL Oral suspension
Formulation (Pharmacokinetics Analysis Set)

| Parameter (units) | Geometric LS Mean<br>for 8 mg/mL<br>Suspension Fasted<br>(n=24) | Geometric LS Mean for<br>2 mg/mL Oral Suspension<br>Fasted<br>(n=23) | Geometric LS<br>Mean Ratio<br>(%)† | 90% CI of<br>Ratio (%)† |
|---|---|---|---|---|
| AUC <sub>inf</sub><br>(ng·h/mL) | 253 | 251 | 100.6 | (90.9, 111.3) |
| AUC <sub>last</sub><br>(ng·h/mL) | 234 | 232 | 100.9 | (90.6, 112.4) |
| C <sub>max</sub><br>(ng/mL) | 12.1 | 11.3 | 106.7 | (84.2, 135.2) |

CI: confidence interval; LS: least squares.

The analysis was performed on log-transformed pharmacokinetic parameters using a linear mixed model with treatment and investigational period as fixed effects and accounting for the longitudinal nature of the data by subject using a REPEATED statement. The covariance matrix is structured by period.

† The geometric LS mean ratios (and associated 90% CIs) were obtained by back-transforming (antilogging) the LS means of the treatment differences.

The information obtained in studies 178-CL-203 and 178-CL-208 was taken into account when predicting the doses for this study as outlined in Section 2.2.2 of this protocol. The doses described in Section 2.2.2 suggest tablets for pediatric subjects with a body weight of  $\geq$  35 kg, and the 8 mg/mL oral suspension for children with a body weight between 11 and 35 kg, or for those subjects with a body weight  $\geq$  35 kg who do not want to or are unable to take tablets.

Safety and tolerability:

In study 178-CL-203 the safety and tolerability of the oral suspension when dosed in children was evaluated and it was concluded that it was safe and well tolerated. From the 6 subjects who completed the study (3 with NDO and 3 with OAB) 1

EudraCT number 2015-002876-25


treatment emergent adverse event (TEAE) was reported: pyrexia on day 1 in a NDO subject. The intensity was mild and was judged by the investigator not to be related to study drug. No clinically significant electrocardiogram (ECG) abnormalities have been seen throughout the study, there were no QTcF values > 450 ms and no QTc prolongation > 30 ms versus baseline was observed (mean of triplicates). Increases in vital signs have been observed but these were not considered clinically significant per investigator's assessment.

A 24-hour Holter recording was recorded in all subjects on a reference day and on the dosing day. The main objective of the Holter recording was to evaluate the effect of mirabegron on heart rate in a time-matched manner, taking into account the circadian rhythm. A median increase in 24-hour heart rate of 5.1 bpm has been observed. This was not considered as clinically relevant taken into account the multiple blood draws, the low number of subjects and the absence of a placebo group.

Some changes in laboratory values were observed, but they were not considered as clinically relevant.

For Study 178-CL-208 single doses of 88 mg mirabegron oral suspension to adults were safe and well tolerated. Eleven of 24 subjects reported 22 adverse events (AEs). All except for 2 events (1 headache moderate and 1 dysmenorrhea moderate) were mild. 20 AEs were considered not related; 2 were considered possibly related (dizziness, mild and orthostatic dizziness mild).

## 1 Introduction and 4 Treatment(s)

1.3 Summary of Key Safety Information for Study Drugs and 4.1.1 Test Drug

## WAS:

Mirabegron has been approved in more than 50 countries including the US, Japan and the EU.

#### IS AMENDED TO:

Mirabegron has been approved in more than 50 65 countries including the US, Japan and the EU worldwide.

#### 1 Introduction

1.4 Risk-Benefit Assessment

## WAS:

• Beyond 4 weeks of therapy, repeated home measurements of the intravesical pressure and at least 1 urodynamic investigation allow the investigator to adapt the CIC-regimen or to withdraw the subject if considered necessary. If SMIP evaluations are not done, the investigator can perform additional urodynamic assessments if deemed necessary.

## IS AMENDED TO:

 Beyond 4 weeks of therapy, repeated home measurements of the intravesical pressure and at least 1 urodynamic investigation allow the investigator to adapt the CIC regimen or to withdraw the subject if considered necessary. If SMIP evaluations are not done, the investigator can perform additional urodynamic assessments if deemed necessary.

ISN/Protocol 178-CL-206A

Sponsor: APEB
EudraCT number 2015-002876-25


• Additional urodynamic assessments may be performed at any time in the study study if deemed necessary by the investigator.

## 2 Study Objective(s), Design, and Endpoints

2.3.2.2 Bladder Volume and Leakage Measures

## ADDED:

For this study the first morning catheterization after waking up is regarded as part of the 'night', whilst the last evening catheterization before sleep time is part of the 'day'. The collected urine volume will be weighed by the subject or subject's parent(s)/caregiver(s) and the results will be entered in the e-diary. The conversion factor used for weight-to-volume is 1g = 1mL.

## 2 Study Objective(s), Design, and Endpoints

2.3.3 Safety Endpoints

## WAS:

 Change from baseline in ECG parameters at visit 5/week 4 and visit 10/week 52 (EOT/EOS)

## IS AMENDED TO:

• Change from baseline in ECG parameters at visit 5/week 4, visit 7/week 12, visit 8/week 24, and visit 10/week 52 (EOT/EOS)

# 2 Study Objective(s), Design and, Endpoints

2.3.4 Pharmacokinetics

## WAS:

The following pharmacokinetic parameters will be determined at visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24 and/or visit 9/week 36:

• C<sub>max</sub>, t<sub>max</sub>, AUC<sub>24</sub>, C<sub>trough</sub>, CL/F and V<sub>z</sub>/F

Additional pharmacokinetic parameters as may be calculated based on the model used.

#### IS AMENDED TO:

The following pharmacokinetic parameters will be determined **for each individual** at visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24 and/or visit 9/week 36:

• C<sub>max</sub>, t<sub>max</sub>, AUC<sub>24</sub>, C<sub>trough</sub>, CL/F and V<sub>z</sub>/F

Additional pharmacokinetic parameters as may be calculated based on the model used.

## 3 Study Population

3.3 Exclusion Criteria

ISN/Protocol 178-CL-206A

Sponsor: APEB

EudraCT number 2015-002876-25


## WAS:

1. Subject has a known genitourinary condition (other than NDO) that may cause overactive contractions or incontinence (e.g., bladder extrophy, urinary tract obstruction, urethral diverticulum or fistula) or kidney/bladder stones or another persistent urinary tract pathology that may cause symptoms.

#### IS AMENDED TO:

1. Subject has a known genitourinary condition (other than NDO) that may cause overactive contractions or incontinence (e.g., bladder extrophy, urinary tract obstruction, urethral diverticulum or fistula) or kidney/bladder stones or another persistent **local** urinary tract pathology that may cause **urinary** symptoms.

## 3 Study Population

3.3 Exclusion Criteria

#### ADDED:

For exclusion criterion 9 please refer to Appendix 12.9 and for exclusion criterion 10 please refer to Appendix 12.10, Appendix 12.11, Appendix 12.12 and Appendix 12.13.

## **5 Treatments and Evaluation**

5.3.4 Pharmacokinetics

## WAS:

These 2 days can be selected from the options given in the schedule of assessments (i.e., on visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24 or visit 9/week 36) and do not have to be in a specific (consecutive) order:

## IS AMENDED TO:

These 2 days can be selected from **any of** the options given in the schedule of assessments (i.e., on visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, or visit 9/week 36, or **visit 10/week 52**) and do not have to be in a specific (consecutive) order:

## **5 Treatments and Evaluation**

5.3.4 Pharmacokinetics

## ADDED:

To allow for an early assessment of the dose-response relationship by the DSMB, it is preferred the pharmacokinetic sampling takes place as early in the study as possible.

## **5 Treatments and Evaluations**

5.4.1.1 Clinic Measurement of Vital Signs

## WAS:

The measurements will be per standard clinic practices and should be consistent for all visits.

EudraCT number 2015-002876-25


## IS AMENDED TO:

The preferred method of measurement is via the auscultatory technique. If this method is not available at the site, measurements will be per standard clinic practices. The method for measuring vital signs and should be consistent for all visits.

## **5 Treatments and Evaluation**

5.4.2 Adverse Events

#### WAS:

AEs will be collected from visit 1/screening until visit 10/week 52 (EOT/EOS). See [Section 5.5] for information regarding AE collection and data handling. Collection of AEs will start once the ICF is signed.

#### IS AMENDED TO:

AEs will be collected from visit 1/screening until visit 10/week 52 (EOT/EOS). See [Section 5.5] for information regarding AE collection and data handling. Collection of AEs will start once the ICF is signed.

## **5 Treatments and Evaluation**

5.4.6 Self-measurement of Intravesical Pressure

#### WAS:

SMIP will be performed as part of the bladder diary [Section 5.3.2].

## IS AMENDED TO:

SMIP will be performed as part of the bladder diary [Section 5.3.2]. In case the measuring device is not available/approved for use at the site, the subject or parent(s)/caregiver(s) are not able or willing to perform the SMIP, or there is a technical problem, the SMIP may be omitted.

## **5 Treatments and Evaluation**

5.5.5 Reporting of Serious Adverse Events

## WAS:

In the case of an SAE, the investigator must contact the CRO by telephone or fax/e-mail immediately (within 24 hours of awareness).

The investigator should complete and submit an SAE Worksheet containing all information that is required by the Regulatory Authorities to CRO by fax/e-mail immediately (within 24 hours of awareness). If the faxing/e-mailing of an SAE Worksheet is not possible or is not possible within 24 hours, the local drug safety contact should be informed by phone. Within 24 hours after receipt of the information, the CRO will forward the SAE details to the Sponsor.

## IS AMENDED TO:

In the case of an SAE, the investigator must contact the CRO by telephone or fax/e-mail immediately (within 24 hours 1 working day of awareness).

02 Nov 2016 Astellas 

ISN/Protocol 178-CL-206A

Sponsor: APEB
EudraCT number 2015-002876-25


The investigator should complete and submit an SAE Worksheet containing all information that is required by the Regulatory Authorities to CRO by fax/e-mail immediately (within 24 hours 1 working day of awareness). If the faxing/e-mailing of an SAE Worksheet is not possible or is not possible within 24 hours 1 working day, the local drug safety contact should be informed by phone. Within 24 hours 1 working day during weekdays or within 60 hours during weekends, whatever is shorter, after receipt of the information, the CRO will forward the SAE details to the Sponsor.

SAEs must be reported up to 28 days after the End of Study visit or up to 28 days after early discontinuation of dosing.

## 7 Statistical Methodology

7.1 Sample Size

## WAS:

A study with 44 evaluable subjects who have MCC measurements at treatment week 24 and at baseline would have a 90 percent power to detect a statistical significant change from baseline, if the real change from baseline in the subject population is at least 52 mL and the real SD for change from baseline is  $\leq 103$  mL.

#### IS AMENDED TO:

A study with 44 evaluable subjects who have **valid** (as by the central reviewer's assessment) nonmissing MCC measurements at treatment visit 8/week 24 and at baseline would have a 90 percent power to detect a statistical significant change from baseline, if the real change from baseline in the subject population is at least 52 mL and the real SD for change from baseline is  $\leq 103$  mL.

## 7 Statistical Methodology

7.2.1 Full Analysis Set

## WAS:

The full analysis set (FAS) will consist of all subjects who:

- Took at least 1 dose of study drug, and
- Provided both valid baseline and at least 1 postbaseline value for the primary efficacy endpoint (MCC).

#### IS AMENDED TO:

The full analysis set (FAS) will consist of all subjects who:

- Took at least 1 dose of study drug, and
- Provided both Had a valid (as by the central reviewer's assessment) nonmissing MCC measurement at baseline and at least 1 a post baseline value visit for the primary efficacy endpoint (MCC).

## 7 Statistical Methodology

7.2.4 Pharmacokinetics Analysis Set

EudraCT number 2015-002876-25


## WAS:

Since the actual bioanalytical results from the last treatment group may only become available after the data review meeting, additional data points may be excluded at the time of pharmacokinetic analysis at the discretion of the pharmacokineticist.

## IS AMENDED TO:

Since the actual bioanalytical results from the last treatment group may only become available after the data review meeting, additional data points may be excluded at the time of pharmacokinetic analysis at the discretion of the pharmacokineticist.

## 7 Statistical Methodology

7.4.1.3 Subgroup and Sensitivity Analyses of Primary Endpoint

#### WAS:

For the primary efficacy endpoint, MCC, 95% CI will be calculated for mean change from baseline per age group.

A subgroup analysis of the primary efficacy endpoint by whether NDO medication treatment was received at screening/prior to start of washout for both groups of subjects will be performed if there are sufficient subject numbers (with and without LOCF) on the FAS.

A subgroup analysis of the primary efficacy endpoint of patients with insufficient efficacy under antimuscarinics specifically intended for NDO treatment (i.e. stopping the medication for lack of efficacy prior to start of treatment) will be performed if there are sufficient subject numbers (with and without LOCF) on the FAS.

The following sensitivity analyses of the primary efficacy endpoint will be performed if there are sufficient subject numbers (without LOCF only) on the FAS:

• Excluding those subjects who had a positive urine culture at visit 3/baseline and/or visit 8/week 24.

## IS AMENDED TO:

For the primary efficacy endpoint, MCC, 95% CI will be calculated for mean change from baseline per age group, **per formulation**, and **per dosing regimen** (with and without LOCF).

Dosing regimen here refers to whether the subjects had been up-titrated to PED50 at least once or maintained at PED25 for safety reasons at least until visit 8/week 24.

A subgroup analysis of the primary efficacy endpoint by whether NDO medication treatment was received at screening/prior to start of washout for both groups of subjects will be performed if there are sufficient subject numbers (with and without LOCF) on the FAS.

A subgroup analysis of the primary efficacy endpoint of patients subjects with insufficient efficacy under antimuscarinics specifically intended for NDO treatment (i.e. stopping the medication for lack of efficacy prior to start of treatment) will be performed if there are sufficient subject numbers (with and without LOCF) on the FAS.

The following sensitivity analyses of the primary efficacy endpoint will be performed if there are sufficient subject numbers (without LOCF only) on the FAS:

EudraCT number 2015-002876-25


• Excluding those subjects who had a positive urine culture at visit 3/baseline and/or visit 8/week 24.

• For any of the subgroups specified, at least 10 subjects by stratum are required.

## 7 Statistical Methodology

7.4.2 Analysis of Secondary Endpoints

#### WAS:

The change from baseline for secondary endpoint based on urodynamic assessments, the subject's e-diary (including bladder diary) and questionnaires will be summarized and analyzed using similar statistical methods as for the primary endpoint, where appropriate.

## IS AMENDED TO:

The change from baseline for secondary endpoint based on urodynamic assessments, the subject's e-diary (including bladder diary) and questionnaires will be summarized and analyzed using similar **primary** statistical methods as for the primary endpoint, where appropriate.

CGI-C and acceptability results will be tabulated per time point of assessment.

## 7 Statistical Methodology

7.5 Analysis of Safety

## WAS:

Safety parameters such as vital signs, height and weight will also be summarized with respect to age- and sex-specific percentiles.

## IS AMENDED TO:

Safety parameters such as vital signs, height and weight will also be summarized with respect to ageheight- and sex-specific percentiles. Height will also be summarized with respect to age- and sex-specific percentiles.

Subgroup presentations regarding age (children and adolescents), formulation (tablets and suspension) and dosing regimen (PED25 and PED50) will be tabulated for the following parameters: AEs, vital signs and ECGs. For any of the subgroups specified, at least 10 subjects by stratum are required.

## 7 Statistical Methodology

7.5.1 Vital Signs

## WAS:

Descriptive statistics will be used to summarize vital sign results and changes from baseline by treatment group and time. Z-scores and percentiles for SBP and DBP will be calculated and summarized based on a comparison with age and sex norms supplied by the Center for Disease Control and Prevention.

EudraCT number 2015-002876-25


#### IS AMENDED TO:

Descriptive statistics will be used to summarize vital sign results and changes from baseline by treatment group and time. **For clinic measurements** Z-scores and percentiles for SBP and DBP will be calculated and summarized based on a comparison with age and **sexheight** norms supplied by the Center for Disease Control and Prevention.

Z-scores and percentiles for pulse rate will be calculated and summarized based on a comparison with age norms based on Fleming [Fleming et al, 2011].

## 7 Statistical Methodology

7.5.2 Adverse Events

## WAS:

AEs will be coded using MedDRA. The number and percentage of AEs, SAEs, AEs leading to discontinuation, and AEs related to study drug will be summarized by system organ class, preferred term and treatment group. The number and percentage of AEs by severity will also be summarized.

## IS AMENDED TO:

AEs will be coded using MedDRA. The number and percentage of AEs, SAEs, AEs leading to discontinuation, and AEs related to study drug will be summarized by system organ class, and preferred term-and treatment group. The number and percentage of AEs by severity will also be summarized.

#### 7 Statistical Methodology

7.5.3 Laboratory Assessments

## WAS:

For quantitative laboratory measurements descriptive statistics will be used to summarize results and change from baseline by treatment group and time point. Shifts relative to normal ranges from baseline to each time point during treatment period in lab tests will also be tabulated.

#### IS AMENDED TO:

For quantitative laboratory measurements descriptive statistics will be used to summarize results and change from baseline by treatment group and time point. Shifts relative to normal ranges from baseline to each time point during treatment period in lab tests will also be tabulated.

## 7 Statistical Methodology

7.5.5 Electrocardiograms

## WAS:

12-lead ECG parameters (QT, QTc, QT interval corrected by Fridericia's formula [QTcF], QTcB, HR, PR, QRS and RR) and their changes from baseline will be summarized with descriptive statistics by visit. The following thresholds will be used to characterize an

ISN/Protocol 178-CL-206A

EudraCT number 2015-002876-25


Sponsor: APEB

individual subject's QTc data: QTc interval > 450 ms for children, and QTc interval > 450 ms and >500 ms for male adolescents and >480 ms and >500 ms for female adolescents. These categories are cumulative in that subjects satisfying criterion for a more extreme category will also be counted in each applicable less extreme category. Similar tables will be provided for QTcF and QTcB as well. A summary of normal, abnormal not clinical significant and abnormal clinical significant findings will be provided.

## IS AMENDED TO:

12-lead ECG parameters (QT, QTe, QT interval corrected by Fridericia's formula [QTcF], QTeB, HR, PR, QRS and RR) and their changes from baseline will be summarized with descriptive statistics by visit. The following thresholds will be used to characterize an individual subject's QTcF data (QTeB and QTeF): QTcF interval > 4540 ms for children, and QTcF interval > 450 ms and >500 ms for male adolescents and >480 ms and >500 ms for female adolescents. These categories are cumulative in that subjects satisfying criterion for a more extreme category will also be counted in each applicable less extreme category. Similar tables will be provided for QTcF and QTcB as well. A summary of normal, abnormal not clinical significant and abnormal clinical significant findings will be provided.

In addition for QTcF, the impact of concomitant medications potentially prolonging QTc will be evaluated.

To perform this analysis, all QTcF post-baseline values will be presented (regardless of time point). If anomalies occur, an additional presentation will be provided using only QTcF values not under the influence of respective concomitant medications. Details on how these will be derived, will be described in the SAP.

## 7 Statistical Analyses

7.5.6 Estimated Glomerular Filtration Rate and Upper Urinary Tract Ultrasound

#### WAS:

For eGFR and upper urinary tract ultrasound, descriptive statistics will be used to summarize results and change from baseline by time point.

#### IS AMENDED TO:

For eGFR and upper urinary tract ultrasound, descriptive statistics will be used to summarize results and change from baseline by time point. The eGFR results will be summarized based upon the Larsson, the modified Schwartz 2009 (for children < 12 years old) and the Cockcroft-Gault equation (for adolescents).

## 7 Statistical Methodology

7.6 Analysis of Pharmacokinetics

## WAS:

Descriptive statistics (N, mean, SD, minimum, median, maximum, coefficient of variation and geometric mean) will be provided for plasma concentration data and derived pharmacokinetic parameters. Further details will be specified in the SAP.

EudraCT number 2015-002876-25


#### IS AMENDED TO:

Descriptive statistics (N, mean, SD, minimum, median, maximum, coefficient of variation and geometric mean) will be provided for plasma concentration data and derived pharmacokinetic parameters. Further details will be specified in the SAP.

# 7 Statistical Methodology 7.6.1 Analysis of Pharmacokinetics Noncompartmental methods will be used to derive the PK parameters using WinNonlin software ( USA). The following plasma PK parameters of mirabegron will be calculated for each individual: C<sub>max</sub>, t<sub>max</sub>, AUC<sub>24</sub>, C<sub>trough</sub>, CL/F and V<sub>z</sub>/F. IS AMENDED TO: Noncompartmental methods will be used to derive the PK parameters using WinNonlin software ( USA). The plasma concentrations will be analyzed with nonlinear mixed effects modeling (population pharmacokinetics) using NONMEM (version 7.3 or higher, USA). The following plasma PK pharmacokinetic parameters of mirabegron will be calculated for each individual subject:

## 8 Operational and Administrative Considerations

 $C_{max}$ ,  $t_{max}$ ,  $AUC_{24}$ ,  $C_{trough}$ , CL/F and  $V_z/F$ .

8.1.1 Data Collection

WAS:

For Screen failures the demographic data, reason for failing, informed consent, inclusion and exclusion criteria and AEs will be collected in the eCRF.

## IS AMENDED TO:

For Screen failures the demographic data, reason for failing, informed consent, inclusion and exclusion criteria and AEs will be collected in the eCRF **and listed**.

#### 11 References

WAS:

U.S. Department of Health and Human Services, National Institutes of Health. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Available from:

https://www.nhlbi.nih.gov/files/docs/resources/heart/hbp\_ped.pdf [Accessed 25 November 2015]

EudraCT number 2015-002876-25


#### IS AMENDED TO:

U.S. Department of Health and Human Services, National Institutes of Health. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. U.S. Department of Health and Human Services, National Institutes of Health National Heart, Lung, and Blood Institute. NIH Publication No. 05-5267 Originally printed September 1996 (96-3790) Revised May 2005. Available from:

https://www.nhlbi.nih.gov/files/docs/resources/heart/hbp\_ped.pdf [Accessed 25 November 2015]

## 11 References

ADDED:

Cockcroft DW, Gault MH (1976). Prediction of creatinine clearance from serum creatinine. Nephron. 16 (1): 31–41. doi:10.1159/000180580. PMID 1244564.

Schwartz GJ, Muñoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, et al. New Equations to Estimate GFR in Children with CKD. J Am Soc Nephrol. 2009;20:629–37.

## 12.3 Laboratory Assessments

**Biochemistry** 

WAS:

Estimated glomerular filtration rate (Larsson)

IS AMENDED TO:

Estimated glomerular filtration rate (Larsson, modified Schwartz and Cockcroft-Gault)


Sponsor: APEB

EudraCT number 2015-002876-25


# 14 SPONSOR'S SIGNATURES